

Biogen MA Inc. 225 Binney Street Cambridge, MA 02142 United States

PROTOCOL NUMBER: 251AD201/NCT03352557

Biogen Idec Research Limited Innovation House 70 Norden Road Maidenhead Berkshire SL6 4AY United Kingdom

PHASE OF DEVELOPMENT: 2

**PROTOCOL TITLE:** Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with Mild Alzheimer's Disease

**EUDRA CT NUMBER:** 2017-002901-37

**IND NUMBER**: 136300

**DATE:** 13 January 2020

Version 4
Final

Supersedes previous Version 3 dated 29 March 2019

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

# SPONSOR SIGNATURE PAGE

Protocol 251AD201 was approved by:

| | 17 - January - 2020 |
|-------|---------------------|
| , PhD | Date |

# **TABLE OF CONTENTS**

| SPONS | OR SIGNATURE PAGE | 2 |
|--------|---------------------------------------------------|----|
| 1. | SYNOPSIS | 9 |
| 2. | LIST OF ABBREVIATIONS | 17 |
| 3. | SPONSOR INFORMATION | 19 |
| 4. | INTRODUCTION | 20 |
| 4.1. | Overview of Alzheimer's Disease | 20 |
| 4.2. | Current Therapies for Alzheimer's Disease | 21 |
| 4.3. | Profile of Previous Experience With BIIB092 | 21 |
| 4.3.1. | Nonclinical Experience | 21 |
| 4.3.2. | Clinical Experience | 21 |
| 4.4. | Study Rationale | 22 |
| 4.5. | Overall Benefits and Risks Assessment | 24 |
| 4.5.1. | Overall Benefit | 24 |
| 4.5.2. | Potential Risks | 24 |
| 4.5.3. | Summary | 25 |
| 5. | SCHEDULE OF ACTIVITIES | 26 |
| 6. | STUDY OBJECTIVES AND ENDPOINTS | 47 |
| 7. | STUDY DESIGN | 51 |
| 7.1. | Study Overview | 51 |
| 7.2. | Study Duration for Participants | 53 |
| | | 55 |
| 7.4. | Study Stopping Rules | 56 |
| 7.5. | End of Study | 56 |
| 8. | SELECTION OF PARTICIPANTS | 57 |
| 8.1. | Inclusion Criteria | 57 |
| 8.2. | Exclusion Criteria | 58 |
| 8.3. | Inclusion Criteria for Long-Term Extension Period | 64 |
| 8.4. | Exclusion Criteria for Long-Term Extension Period | 65 |
| 9. | SCREENING AND RANDOMIZATION | 67 |
| 9.1. | Screening | 67 |
| 9.2. | Randomization | 68 |

| 9.3. | Blinding Procedures | 69 |
|---|---|---|
| 10. | DISCONTINUATION OF STUDY TREATMENT AND WITHDRAWAL OF PARTICIPANTS FROM THE STUDY | 71 |
| 10.1. | Discontinuation of Study Treatment. | 71 |
| 10.2. | Lost to Follow-Up. | 72 |
| 10.3. | Withdrawal of Participants From Study | 72 |
| 11. | STUDY TREATMENT USE | 74 |
| 11.1. | Regimen | 74 |
| 11.1.1. | Placebo-Controlled Period | 74 |
| 11.1.2. | Long-Term Extension Period | 74 |
| 11.2. | Modification of Dose and/or Treatment Schedule | 74 |
| 11.2.1. | Dose Suspension | 75 |
| 11.2.2. | Infusion Interruption | 75 |
| 11.3. | Compliance | 75 |
| 11.4. | Concomitant Therapy and Procedures | 75 |
| 11.4.1. | Concomitant Therapy | 75 |
| 11.4.1.1. | Allowed Concomitant Therapy | 76 |
| 11.4.1.2. | Disallowed Concomitant Therapy | 76 |
| 11.4.2. | Concomitant Procedures | 78 |
| 11.4.3. | Tobacco Use | 78 |
| 11.5. | Continuation of Treatment | 78 |
| 12. | STUDY TREATMENT MANAGEMENT | 79 |
| 12.1. | BIIB092 | 79 |
| 12.1.1. | BIIB092 Preparation | 79 |
| 12.1.2. | BIIB092 Storage | 79 |
| 12.1.3. | BIIB092 Handling and Disposal | 80 |
| 12.1.4. | BIIB092 Accountability | 80 |
| 12.2. | Placebo | 80 |
| 12.3. | Additional Protocol-Designated Products – | 80 |
| 13. | EFFICACY, PHARMACOKINETIC, PHARMACODYNAMIC, IMMUNOGENICITY, AND HEALTH OUTCOMES ASSESSMENTS | |
| 13.1. | Clinical Efficacy Assessments. | |

| 13.2. | Pharmacokinetic Assessments | 82 |
|---|---|---|
| 13.3. | Pharmacodynamic Assessments | 83 |
| | | 83 |
| | | 84 |
| 13.6. | Immunogenicity | 84 |
| 13.7. | Health Outcomes Assessments | 85 |
| 14. | SAFETY ASSESSMENTS | 86 |
| 14.1. | Clinical Safety Assessments | 86 |
| 14.2. | Laboratory Safety Assessments | 86 |
| 15. | SAFETY DEFINITIONS, RECORDING, REPORTING, AND RESPONSIBILITIES | 88 |
| 15.1. | Definitions | 88 |
| 15.1.1. | Adverse Event | 88 |
| 15.1.2. | Serious Adverse Event | 88 |
| 15.1.3. | Prescheduled or Elective Procedures or Routinely Scheduled Treatments | 89 |
| 15.2. | Safety Classifications. | 89 |
| 15.2.1. | Investigator Assessment of Events | 89 |
| 15.2.2. | Relationship of Events to Study Treatment | |
| 15.2.3. | Severity of Events | |
| 15.2.4. | Expectedness of Events | |
| 15.3. | Monitoring and Recording Events | 91 |
| 15.3.1. | Adverse Events | 91 |
| 15.3.2. | Adverse Events of Special Interest | 92 |
| 15.3.3. | Serious Adverse Events | 92 |
| 15.3.4. | Immediate Reporting of Serious Adverse Events | 92 |
| 15.3.4.1. | Deaths | 92 |
| 15.3.5. | Suspected Unexpected Serious Adverse Reactions | 93 |
| 15.4. | Procedures for Handling Special Situations | 93 |
| 15.4.1. | Pregnancy | 93 |
| 15.4.2. | Overdose | 93 |
| 15.4.3. | Medical Emergency | 93 |
| 15.4.3.1. | Unblinding for Medical Emergency | 94 |

| 15.5. | Contraception Requirements | 94 |
|---|---|---|
| 15.6. | Safety Responsibilities | 95 |
| 15.6.1. | The Investigator | 95 |
| 15.6.2. | Biogen | 96 |
| 16. | STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE | 97 |
| 16.1. | General Considerations | 97 |
| 16.2. | Demography and Baseline Disease Characteristics | 97 |
| 16.3. | Safety | 97 |
| 16.3.1. | Analysis Population | 97 |
| 16.3.2. | Methods of Analysis | 97 |
| 16.3.2.1. | Adverse Events | 97 |
| 16.3.2.2. | Clinical Laboratory Results | 98 |
| 16.3.2.3. | Vital Signs | 98 |
| 16.3.2.4. | Electrocardiograms | 98 |
| 16.3.2.5. | Physical and Neurological Examinations | 98 |
| 16.3.2.6. | Columbia - Suicide Severity Rating Scale | 98 |
| 16.4. | Efficacy | 98 |
| 16.4.1. | Analysis Population | 98 |
| 16.4.2. | Methods of Analysis | 99 |
| 16.4.2.1. | Analysis of Primary Efficacy Endpoint (Clinical Dementia Rating Scale – Sum of Boxes) | 99 |
| 16.4.2.2. | Analysis of Exploratory Clinical Endpoints | 99 |
| 16.4.3. | Analysis for the Long-Term Extension Period | 100 |
| 16.5. | Pharmacokinetics | 100 |
| 16.5.1. | Analysis Population | 100 |
| 16.5.2. | Methods of Analysis | 100 |
| 16.6. | Pharmacodynamics | 101 |
| 16.6.1. | Analysis Population | 101 |
| 16.6.2. | Methods of Analysis for Tau Positron Emission Tomography Results | 101 |
| 16.6.3. | Methods of Analysis for Other Pharmacodynamic Parameters | 101 |
| 16.7. | Health Outcomes | 102 |
| 16.7.1. | Analysis Population | 102 |

| 16.7.2. | Methods of Analysis | 102 |
|---|---|---|
| 16.8. | Immunogenicity | 102 |
| 16.8.1. | Analysis Population | 102 |
| 16.8.2. | Methods of Analysis | 102 |
| 16.9. | Interim Analyses | 102 |
| 16.10. | Sample Size Considerations | 103 |
| 17. | ETHICAL REQUIREMENTS | 105 |
| 17.1. | Declaration of Helsinki | 105 |
| 17.2. | Ethics Committee | 105 |
| 17.3. | Participant Information and Consent | 106 |
| 17.4. | Participant Data Protection | 107 |
| 17.5. | Compensation for Injury | 108 |
| 17.6. | Conflict of Interest | 108 |
| 17.7. | Registration of Study and Disclosure of Study Results | 108 |
| 18. | ADMINISTRATIVE PROCEDURES | 109 |
| 18.1. | Study Site Initiation | 109 |
| 18.2. | Quality Control and Quality Assurance | 109 |
| 18.3. | Monitoring of the Study | 109 |
| 18.4. | Study Funding | 110 |
| 18.5. | Publications | 110 |
| 19. | FURTHER REQUIREMENTS AND GENERAL INFORMATION | 111 |
| 19.1. | External Contract Organizations | 111 |
| 19.1.1. | Contract Research Organization | 111 |
| 19.1.2. | Interactive Response Technology | 111 |
| 19.1.3. | Electronic Data Capture | 111 |
| 19.1.4. | Central Laboratories for Laboratory Assessments | 111 |
| 19.1.5. | Central Facility for Other Assessments | 111 |
| 19.1.6. | Neurocognitive Assessments | 112 |
| 19.2. | Study Committees | 112 |
| 19.3. | Changes to Final Study Protocol | 112 |
| 19.4. | Ethics Committee Notification of Study Completion or Termination | 112 |
| 19.5. | Retention of Study Data | 113 |

### 1. SYNOPSIS

Protocol Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study

to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with

Mild Alzheimer's Disease

Protocol Number: 251AD201

Version Number: 4

Name of Study Treatment: BIIB092 (formerly known as BMS 986168, IPN007)

Study Phase: 2

Study Indication: Mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or

mild AD

Study Rationale: BIIB092 is a humanized immunoglobulin G4 monoclonal antibody that

has been shown to bind tau at the amino terminus. Although tau is primarily an intracellular protein, a portion of tau is secreted by

neurons as N-terminal tau fragments.

BIIB092 has been shown to lower cerebrospinal fluid (CSF) concentrations of N-terminal tau in nonclinical studies, a single-ascending-dose study in healthy participants, and a multiple-ascending-dose study in participants with progressive supranuclear palsy. Based upon the close links between tau pathology, neurodegeneration, and clinical features consistent with AD, coupled with the evidence that tau pathology can spread via neuronal release

and uptake of pathological tau species, examination of BIIB092 in the clinical AD setting is strongly supported as a potential

disease-modifying therapy. This study will assess the safety and efficacy of BIIB092 in participants with MCI due to AD or with mild AD and help to inform on dose selection in this patient population.

Study Objectives and Endpoints:

### **Placebo-Controlled Period**

The primary objective of the study for the placebo-controlled period is to evaluate the safety and tolerability of BIIB092 in participants with MCI due to AD or with mild AD.

The primary safety endpoints that relate to this objective are the incidence of adverse events (AEs) and serious AEs (SAEs) during the


The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

placebo-controlled period.

Secondary objectives and endpoints are as follows:

- To evaluate the efficacy of multiple doses of BIIB092 in slowing cognitive and functional impairment in participants with MCI due to AD or with mild AD as measured by the change from Baseline over time at Week 78 on the Clinical Dementia Rating Scale (CDR) - Sum of Boxes (CDR-SB). This is the primary efficacy objective, with the primary efficacy endpoint.
- To evaluate the immunogenicity of BIIB092 after multiple doses in participants with MCI due to AD or with mild AD as measured by the incidence of anti-BIIB092 antibodies in serum over time up to Week 90.

Exploratory objectives and endpoints are as follows:

- To assess the effect of BIIB092 on the clinical progression of AD as measured by changes from Baseline over time up to Week 78 on the Mini-Mental State Examination (MMSE), International Shopping List Test Immediate Recall (ISLT), Category Fluency and Letter Fluency tests from the Delis-Kaplan Executive Function System (DKEFS), Digit Symbol Substitution Test (DSST), Trail Making Test Part A (Trails A), Everyday Cognition (eCog), Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL), Functional Activities Questionnaire (FAQ), Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog 13 [13 item]), and Neuropsychiatric Inventory-10 (NPI-10).
- To assess the effect of BIIB092 on changes in caregiver burden and participant quality of life as measured by changes from Baseline over time up to Week 68 on the Zarit Burden Interview (ZBI) and Quality of Life for Alzheimer's Disease (QoL-AD).
- To assess the effect of BIIB092 on resource utilization as measured by the Resource Utilization in Dementia-Lite (RUD-Lite) Version results over time up to Week 68.
- To assess BIIB092 pharmacokinetics (PK) in serum (trough serum BIIB092 concentrations and end-of-infusion serum BIIB092 concentrations) from the samples collected at the

visits indicated in the Schedule of Activities in participants with MCI due to AD or with mild AD.



 To assess the effect of BIIB092 on biomarkers in blood as measured by changes from Baseline over time up to Week 76 on blood levels of disease-related biomarkers, including but not limited to, tau and other markers of neurodegenerative disease.



 To assess the effect of BIIB092 on brain structure as measured by changes from Baseline over time up to Week 78 on magnetic resonance imaging (MRI) morphometric measures, including volume and cortical thickness of certain brain areas.

### **Long-Term Extension Period**

The primary objective for the long-term extension (LTE) period is to evaluate the long-term safety and tolerability of BIIB092 in participants with MCI due to AD or with mild AD.

The primary safety endpoint that relates to this objective is the


The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

incidence of AEs and SAEs over the placebo-controlled period and LTE period of the study.

Exploratory objectives and endpoints are as follows:

- To further evaluate the immunogenicity of BIIB092 after multiple doses in participants with MCI due to AD or with mild AD as measured by the incidence of anti-BIIB092 antibodies in serum over time up to Week 238.
- To further assess the effect of BIIB092 on disease progression as measured by fluid and radiological biomarkers, as well as additional clinical and health outcomes as measured by the following:
  - Changes over the placebo-controlled period and LTE period on the CDR-SB, MMSE, ISLT, Category Fluency and Letter Fluency tests from the DKEFS, DSST, Trails A, eCog, ADCS-ADL, FAQ, ADAS-Cog-13 (13-item), and NPI-10
  - Changes over the placebo-controlled period and LTE period on the ZBI, QoL-AD, and RUD-Lite



- Changes over the placebo-controlled period and LTE period on MRI brain morphometric measures
- To assess BIIB092 PK in serum (trough serum BIIB092 concentrations)

  from

from the samples collected at the visits indicated in the Schedule of Activities in participants with MCI due to AD or with mild AD.

Study Design:

This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group study consisting of a double-blind, placebo-controlled period and an LTE period.





Study Location: Approximately 100 study sites globally are planned.

Number of Planned Participants: Approximately 528 participants were planned to be randomized. Due to fast recruitment, the study was over-enrolled and 654 participants have been randomized.

Study Population:

This study will be conducted in participants aged 50 to 80 years, inclusive, with MCI due to AD or mild AD according to National Institute on Aging-Alzheimer's Association criteria.

Participants must also perform at 1 standard deviation below the age-adjusted normative mean on either the ISLT or the International Shopping List Test Delayed Recall and have a CDR global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD, an MMSE score of 22 to 30 (inclusive), and a CDR Memory Box score of >0.5.

Detailed eligibility criteria are described in Section 8.

**Treatment Groups:** 

During the placebo-controlled period, randomized participants will receive 1 of the following study treatments by intravenous (IV) infusion, starting on Study Day 1:

- low-dose BIIB092 125 mg once every 4 weeks or 375 mg once every 12 weeks (88 participants planned in total, 44 per regimen)
- medium-dose BIIB092 600 mg once every 4 weeks (88 participants planned)
- high-dose BIIB092 2000 mg once every 4 weeks (176 participants planned)
- placebo (176 participants planned)


The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

During the dose-blinded LTE period, participants will receive BIIB092 by IV once every 4 weeks beginning at Week 80. Participants who were randomized to receive BIIB092 during the placebo-controlled period will continue to receive BIIB092 at the dose they were randomly assigned. Participants randomized to receive placebo during the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period.

Duration of Treatment and Follow-up:

The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. For participants who complete both the placebo-controlled period and the LTE period, the total study duration will be approximately 247 weeks.

### **Placebo-Controlled Period**

Participation in the placebo-controlled period will be approximately 99 weeks, which includes the Screening Period of approximately 9 weeks, the 76-week Treatment Period, and the End-of-Study (EOS) Visit at Week 78, and for participants not entering the LTE period, a Follow-up Safety Visit at Week 90, or approximately 14 weeks after the last dose of study treatment. It is recommended that all the screening procedures be completed within 65 days; however, the overall Screening Period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate

Participants will have

approximately 25 outpatient clinic visits:

- Participant eligibility will be determined at up to 3 visits during the Screening Period (Screening Visits 1, 2, and 3).
- On Study Day 1, eligible participants will be randomized, have scheduled assessments per the Schedule of Activities, and receive the first infusion of randomized study treatment.
- Participants will return to the clinic at 4-week intervals during the Treatment Period for infusions of study treatment and study assessments (Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76). The last dose of study treatment will be administered at Week 76 (End-of-Treatment Visit).
- For a participant who completes the Treatment Period at Week 76, there will be an EOS Visit at Week 78 for final

study assessments of the placebo-controlled period. A Follow-up Safety Visit will occur at Week 90 (14 weeks after the last dose of study treatment is administered), unless the participant elects to enter an extension study following the Week 78 Visit.

- Participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures. These participants should be encouraged to attend at least the Week 24, Week 52, and Week 78 visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely will also be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment.
- Participants who withdraw from the study prematurely are to return to the study site for an Early Termination (ET) Visit and assessments and for the Follow-up Safety Visit 14 weeks after administration of the final infusion of study treatment.

### **Long-Term Extension Period**

Participants who meet the LTE inclusion and exclusion criteria will be eligible to enter the dose-blinded LTE period, which includes the LTE Screening Period of approximately 4 weeks starting at Week 76, the 144-week Treatment Period starting at Week 80, the EOS Visit at Week 226, and the Follow-up Visit at Week 238.

Participants will have approximately 39 outpatient clinic visits during the LTE period:

- Participant eligibility will be determined at Week 76 or Week 78 of the placebo-controlled period and confirmed at Week 80 of the LTE period.
- At the Week 80 Visit, eligible participants will have scheduled assessments per the Schedule of Activities and receive the first infusion of BIIB092 during the LTE period.

All participants receiving placebo in the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period.

- Participants will return to the clinic at 4-week intervals during the Treatment Period for infusions of study treatment and study assessments.
- The last dose of study treatment will be administered at Week 224 (End-of-Treatment Visit). The EOS Visit will occur at Week 226 and the Follow-up Visit at Week 238.
  - Participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures. These participants should be encouraged to attend at least the Week 80, 104, 116, 128, 152, 156, 176, 196, 200, 224, and 226 Visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely will also be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment.
  - Participants who withdraw from the study prematurely are to return to the study site for an Early Termination
     Visit and assessments and for the Follow-up Safety Visit
     14 weeks after receiving the last dose of study treatment.

# 2. LIST OF ABBREVIATIONS

| Αβ | amyloid beta |
|-------------|-------------------------------------------------------------|
| AD | Alzheimer's disease |
| ADAS-Cog 13 | Alzheimer's Disease Assessment Scale – Cognitive (13 item) |
| ADCS-ADL | Alzheimer's Disease Cooperative Study – Activities of Daily |
| | Living |
| ADNI | Alzheimer's Disease Neuroimaging Initiative |
| AE | adverse event |
| ALT | alanine aminotransferase |
| anti-HBc | hepatitis B core antibody |
| anti-HBs | hepatitis B surface antibody |
| AST | aspartate aminotransferase |
| BUN | blood urea nitrogen |
| CBC | complete blood count |
| CDR | Clinical Dementia Rating Scale |
| CDR-SB | Clinical Dementia Rating Scale – Sum of Boxes |
| CI | confidence interval |
| CRF | case report form |
| CRO | contract research organization |
| , | |
| C-SSRS | Columbia – Suicide Severity Rating Scale |
| DBP | diastolic blood pressure |
| DHA | Directions for Handling and Administration |
| DKEFS | Delis-Kaplan Executive Function System |
| DMC | Data Monitoring Committee |
| DSST | Digit Symbol Substitution Test |
| ECG | electrocardiogram |
| eCog | Everyday Cognition |
| Emax | maximum response |
| EOS | end of study |
| ET | early termination |
| FAQ | Functional Activities Questionnaire |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |

| Ĭα | immunoglobulin |
|-----------|-------------------------------------------------------|
| Ig<br>INR | international normalized ratio |
| IRT | |
| | interactive response technology |
| ISLR | International Shopping List Test Delayed Recall |
| ISLT | International Shopping List Test Immediate Recall |
| ITT | intent-to-treat |
| IV | intravenous |
| LS | least squares |
| LTE | long-term extension |
| MAD | multiple-ascending-dose |
| MAO | monoamine oxidase |
| MCI | mild cognitive impairment |
| MCP – MOD | multiple comparison procedure – modelling |
| MMRM | mixed model with repeated measures |
| MMSE | Mini-Mental State Examination |
| MRI | magnetic resonance imaging |
| NFT | neurofibrillary tangle |
| NIA-AA | National Institute on Aging – Alzheimer's Association |
| NPI-10 | Neuropsychiatric Inventory – 10 |
| PD | pharmacodynamic(s) |
| PET | positron emission tomography |
| PK | pharmacokinetic(s) |
| PSP | progressive supranuclear palsy |
| QoL-AD | Quality of Life for Alzheimer's Disease |
| RUD-Lite | Resource Utilization in Dementia-Lite Version |
| SAD | single-ascending-dose |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SUSAR | suspected unexpected serious adverse reaction |
| Trails A | Trail Making Test, Part A |
| ULN | upper limit of normal |
| UTI | urinary tract infection |
| UV | unscheduled visit |
| ZBI | Zarit Burden Interview |
| 201 | Land Danger Hiller (10 ) |

### 3. SPONSOR INFORMATION

Biogen MA Inc. 225 Binney Street Cambridge, MA 02142 United States Biogen Idec Research Limited Innovation House 70 Norden Road Maidenhead, Berkshire SL6 4AY United Kingdom Biogen Japan Ltd. Nihonbashi 1-chome Mitsui Building 14F 4-1 Nihonbashi 1-chome Chuo-ku, Tokyo 103-0027 Japan

Biogen Australia PTY Ltd. Suite 1, Level 3 123 Epping Road North Ryde, NSW 2113 Australia

For urgent medical issues in which the study Medical Director should be contacted, please see the Study Reference Guide's Official Study Contact List for complete contact information.

Biogen may transfer any or all of its study-related responsibilities to a contract research organization (CRO) and other third parties; however, Biogen retains overall accountability for these activities.

### 4. INTRODUCTION

### 4.1. Overview of Alzheimer's Disease

Alzheimer's disease (AD) is a progressive neurodegenerative disorder clinically characterized by cognitive impairment, behavioral disturbances, psychiatric symptoms, and disability in activities of daily living. These clinical manifestations constitute the syndrome dementia. AD International estimates that the number of people living with dementia worldwide will increase from (the current estimate of) 46.8 million to 131.5 million by 2050 [Alzheimer's Disease International 2015]. As the most common cause of dementia, AD accounts for 60% to 80% of dementia cases [Alzheimer's Association 2015].

The main neuropathological hallmarks of AD are extracellular senile (neuritic) plaques containing aggregated  $\beta$ -amyloid (A $\beta$ ) peptides and intraneuronal neurofibrillary tangles (NFTs) composed of abnormal hyperphosphorylated tau protein.

The amyloid hypothesis of AD etiology postulates that misfolded Aβ peptide is a causative factor, which is strongly supported by human genetics [Hardy and Selkoe 2002]. While the evidence for Aβ as the initiator of the pathophysiological cascade leading to AD dementia is strong, the link between Aβ pathology and neurodegeneration in AD and the subsequent clinical progression, both temporally and anatomically, is relatively weak [Musiek and Holtzman 2015; Serrano-Pozo 2011]. Amyloid plaques are present in patients with AD 10 to 15 years before onset of AD symptoms and overt neuronal loss, and they reach a plateau around clinical onset [Jack 2013].

A much stronger correlation has been demonstrated between tau pathology (in the form of NFTs of the aggregated, misfolded microtubule-associated protein tau) and neuronal loss and cognitive decline. In AD, atrophy as seen on magnetic resonance imaging (MRI) and hypometabolism as seen with fluorodeoxyglucose (FDG) positron emission tomography (PET), correlate highly with postmortem histochemical analysis of synaptic and neuron loss and, importantly, tau burden [Jack 2013; Serrano-Pozo 2011]. Imaging data obtained using novel PET tau radioligands alone or in combination with functional and structural imaging methods (e.g., FDG PET or structural MRI) as well as cognitive testing demonstrated stronger correlations between tau PET signal and neurodegeneration, hypometabolism, and cognitive deficits, than for amyloid PET signal [Johnson 2016; Pontecorvo 2017]. While these are early findings, and a better understanding of the existing tau PET imaging agents as well as longitudinal studies are needed, the recent findings lend further support to the close link between tau pathology, neurodegeneration and AD symptoms.

There are currently no approved therapies that modify the course of AD. However, due to the central role of tau in neurodegeneration and its close correlation with cognitive decline in AD, modification of tau pathology has potential for the treatment of AD.

# 4.2. Current Therapies for Alzheimer's Disease

No new therapies for AD have been approved in more than a decade. Currently approved therapies (and their approval dates) include the central cholinesterase inhibitors (donepezil [Aricept®; 2004], rivastigmine [Exelon®; 2000], and galantamine [Reminyl®; 2001]) and the N-methyl-D-aspartate antagonist memantine (Ebixa®; Namenda®; 2003). These medications provide only symptomatic benefit and do not attenuate the course of the disease [Birks 2006; McShane 2006].

# 4.3. Profile of Previous Experience With BIIB092

Please see the BIIB092 Investigator's Brochure for detailed information on relevant nonclinical and clinical studies.

### 4.3.1. Nonclinical Experience

In nonclinical pharmacology studies, BIIB092 was shown to recognize a linear, nonphosphorylated, amino terminal epitope (including amino acid residues 15-24 of full-length human tau) of the microtubule-associated protein tau. BIIB092 exhibited high affinity for human and cynomolgus monkey tau, with binding affinities of 7.10<sup>-10</sup> M and 6.35<sup>-10</sup> M, respectively. The primary site of action of BIIB092 is believed to be the interstitial space between neurons where it binds tau, thereby reducing eTau-mediated spread of tau pathology, and this proposed site of action is supported by nonclinical studies.

Pharmacokinetic (PK) and pharmacodynamic (PD) analysis of serum and cerebrospinal fluid (CSF) BIIB092 concentrations from 3 experiments in cynomolgus monkeys (intravenous [IV] injection/infusion doses of 0.5 to 60 mg/kg) showed that CSF N-terminal tau levels were reduced in a dose-dependent manner. The duration of reduction of CSF N-terminal tau was also dose-dependent. Higher doses were associated with longer reductions of N-terminal tau in CSF. For example, the reduction of N-terminal tau in CSF (25% to 50%) persisted for more than 58 days at doses ≥20 mg/kg.

The nonclinical toxicology studies conducted to date have demonstrated an acceptable safety profile for BIIB092 to support continued use in clinical studies.

### 4.3.2. Clinical Experience

The present study is the first study of BIIB092 in AD. Previous clinical studies have been conducted to support development of BIIB092 for the treatment of patients with progressive supranuclear palsy (PSP).

BIIB092 has been evaluated in 4 completed or ongoing clinical studies (Studies CN002001, CN002003, 251PP201 [CN002004], and 251PP301 [CN002012]):

 Study CN002001, the first-in-human study of BIIB092, was a Phase 1, randomized, double-blind, placebo-controlled, single-ascending-dose (SAD) study in healthy participants to characterize the safety, tolerability, PK, PD, and immunogenicity of

single doses of BIIB092 ranging from 21 mg to 4200 mg. Single doses of BIIB092 were safe and well tolerated at all dose levels tested. The extent and duration of suppression of CSF N-terminal tau increased with increasing dose. Following single doses of BIIB092, the mean suppression of CSF N-terminal tau on Study Day 29 ranged from 65% to 96% at doses ranging from 70 mg to 4200 mg. Greater than 80% suppression of CSF N-terminal tau was achieved with single doses of BIIB092  $\geq$ 210 mg. The suppression of N-terminal tau following dosing with BIIB092 persisted over the course of the 12-week study.

- Study CN002003 was a Phase 1b, randomized, double-blind, placebo-controlled multiple-ascending-dose (MAD) study to characterize the safety, tolerability, PK, PD, and immunogenicity of BIIB092 doses of 150 mg, 700 mg, and 2100 mg administered every 4 weeks in participants with PSP. All 3 doses were safe and well tolerated, based on results from the dose-escalation phase of the study. Treatment with multiple monthly doses of BIIB092 decreased CSF N-terminal tau by mean values of approximately 90%, 93%, and 96% on Study Day 29 and 91%, 95%, and 97% on Study Day 85 at doses of 150, 700, and 2100 mg, respectively.
- Study 251PP201 is an ongoing Phase 1b open-label extension study to evaluate the long-term safety and tolerability of multiple doses of BIIB092 in participants with PSP who participated in CN002003.
- Study 251PP301 is an ongoing Phase 2b randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of intravenously administered BIIB092 2000 mg versus placebo (2:1 randomization ratio) in participants with PSP.

# 4.4. Study Rationale

BIIB092 is a humanized immunoglobulin (Ig) G4 monoclonal antibody that has been shown to bind tau at the amino terminus. Although tau is primarily an intracellular protein, a portion of tau is secreted by neurons as N-terminal tau fragments.

BIIB092 has been shown to lower CSF concentrations of N-terminal tau in nonclinical studies, a SAD study in healthy participants (Study CN002001), and a MAD study in participants with PSP (Study CN002003). AD is defined by 2 neuropathologic hallmarks: extracellular neuritic plaques containing Aβ peptide and intraneuronal NFTs composed of hyperphosphorylated tau protein. Based upon the close links between tau pathology, neurodegeneration, and clinical features consistent with AD, coupled with the evidence that tau pathology can spread via neuronal release and uptake of pathological tau species, examination of BIIB092 in the clinical AD setting is strongly supported as a potential disease-modifying therapy. This study will assess the safety and efficacy of BIIB092 in participants with mild cognitive impairment (MCI) due to AD or with mild AD, selected by proof of brain amyloid burden. This study will also help to inform on dose selection in this patient population.

### Rationale for BIIB092 dose selection

The present study is primarily designed to assess the safety and tolerability of IV BIIB092 at doses of 125, 600, and 2000 mg administered once every 4 weeks or 375 mg administered once every 12 weeks versus placebo in participants with MCI due to AD or with mild AD. As a secondary objective, the study will evaluate the efficacy of BIIB092 in slowing cognitive and functional impairment in the study participants, as measured by changes from Baseline in the Clinical Dementia Rating Scale (CDR) - Sum of Boxes (CDR-SB), the primary efficacy endpoint.



### Rationale for use of placebo

Placebo is included as a randomized treatment in this study to avoid bias in the evaluation of BIIB092, including the reporting of adverse events (AEs) to address the primary objective. Concomitant therapy specifications for the study will protect participant safety by allowing the continuation of medications for chronic conditions as long as dosage has been stable for 4 weeks prior to the first Screening Visit and the use of therapies for AD if the participant was on a stable dose for at least 8 weeks prior to Screening Visit 1 and is expected to stay on a stable dose while in the study. (See Section 11.4.1 for details on concomitant therapy use.)

### 4.5. Overall Benefits and Risks Assessment

### 4.5.1. Overall Benefit

BIIB092 has the potential to slow or stop the spread of tau pathology observed in neurodegenerative diseases such as PSP, AD, and other tauopathies.

In participants with PSP, BIIB092 has been evaluated in 2 completed clinical studies (Studies CN002001 and CN002003) and is currently being evaluated in the ongoing Studies 251PP201 and 251PP301. The first-in-human study of BIIB092 (Study CN002001) was designed as a randomized, double-blind, placebo-controlled, SAD study in healthy participants to characterize the safety, tolerability, PK, PD, and immunogenicity of single doses of BIIB092, ranging from 21 to 4200 mg. Study CN002003, a Phase 1b study, was designed as a randomized, double-blind, placebo-controlled MAD study to characterize the safety, tolerability, PK, PD, and immunogenicity of multiple doses of BIIB092, ranging from 150 to 2100 mg, in participants with PSP. In both of these completed studies, BIIB092 was found to be well tolerated at the doses tested in both healthy participants and participants with PSP. The ongoing Phase 1b study, Study 251PP201, is designed as an open-label extension study to evaluate the long-term safety and tolerability of multiple doses of BIIB092 in participants with PSP who participated in Study CN002003. Several interim analyses of the data being collected in this study have been performed to date. Study 251PP301 is an ongoing Phase 2b study designed as a randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of IV-administered BIIB092 in participants with PSP.

In participants with AD, this study (Study 251AD201) will evaluate the safety and efficacy of BIIB092.

Based on the PK and PD data from Studies CN002001 and CN002003, the mean concentrations of BIIB092 in CSF increased in a generally dose-proportional manner. A robust and persistent lowering of unbound N-terminal tau was observed following administration of single and multiple doses of BIIB092 in healthy participants and in participants with PSP, consistent with the observations in cynomolgus monkeys.

### 4.5.2. Potential Risks

The nonclinical studies conducted to date have demonstrated an acceptable safety profile for BIIB092 to support continued use in clinical studies.

As of 25 November 2018, an estimated 486 healthy participants or participants with PSP or AD have been exposed to BIIB092 in clinical studies. The following summary of the safety profile of BIIB092 is based on safety data from the completed Studies CN002001 and CN002003 and the ongoing Study 251PP201. In the SAD study in healthy participants, there were no safety findings of note, and development continued in patients with PSP. In participants with PSP, to date, the most commonly reported AEs were fall, urinary tract infection (UTI), contusion, and headache. Most AEs have been reported as mild or moderate in intensity. Serious AEs (SAEs) have generally been consistent with disease (UTI, respiratory arrest, aspiration pneumonia, and progressive PSP) or are not unexpected in the patient population enrolled in the trials

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

(cholecystitis, cancer, fractures, and anemia). There have been 3 deaths, all of which were likely related to underlying disease (respiratory arrest, aspiration pneumonia, and progressive disease). None of the SAEs or deaths were considered related to BIIB092 by Investigators. No safety concerns have been identified from laboratory, vital signs, or electrocardiogram (ECG) assessments. Nonserious infusion reactions have been observed and are an identified risk of BIIB092.

BIIB092 is a humanized IgG4 monoclonal antibody. While a low risk of immunogenicity is suggested by preclinical studies, the risk of immunogenicity in humans is unknown. Immunogenicity is an AE of special interest that is under monitoring in all ongoing studies. No safety data regarding this topic have emerged that would change the safety profile of BIIB092.

In general, BIIB092 has been well tolerated in the clinical study participants. There are no important identified or potential risks in the program. The safety profile is acceptable to continue development.

#### 4.5.3. **Summary**

Currently available treatments for AD offer modest symptomatic relief, but none has the potential to modify the underlying disease pathology or course of the disease. In addition, no medications have been approved for the treatment of PSP. Therefore, there is a significant unmet need for the development of effective disease-modifying therapies in both PSP and AD.

Based on the PK and PD data from Studies CN002001 and CN002003, the mean concentrations of BIIB092 in CSF increased in a generally dose-proportional manner. A robust and persistent lowering of unbound N-terminal tau was observed following administration of single and multiple doses of BIIB092 in healthy participants and in participants with PSP, consistent with the observations in cynomolgus monkeys.

Based on the safety data from the completed Studies CN002001 and CN002003 and the data from an interim analysis of the ongoing Study 251PP201, BIIB092 was generally well tolerated and demonstrated an acceptable safety profile for continued development.

The overall analysis of potential benefits (based on the robust and persistent lowering of unbound N-terminal tau in healthy participants and in participants with PSP, consistent with cynomolgus monkeys) and risks (available safety data indicating that BIIB092 is generally well tolerated) supports the continued development of BIIB092 in both PSP and AD.

# 5. SCHEDULE OF ACTIVITIES

The schedule of study activities is presented in Table 1, Table 2, Table 3, and Table 4.

Table 1: Schedule of Activities During the Placebo-Controlled Period and the LTE Screening Period

| | S<br>Perio | Baselin<br>creenir<br>od <sup>1, 2</sup> w<br>ays <sup>3</sup> of<br>1 | ig<br>ithin | | | | | | | | | I | Placebo | o-Cont | rolled l | Period <sup>4</sup> | I | | | | | | | | UV for<br>Change in<br>AD<br>Medication | FUV <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>7</sup> | | 90 |
| Study Day | S1 | S2 | S38 | 1 | 29<br>±7 | 57<br>±<br>7 | 85<br>±7 | 11<br>3<br>±7 | 14<br>1<br>±7 | 169<br>±7 | 19<br>7<br>±7 | 22<br>5<br>±7 | 25<br>3<br>±7 | 28<br>1<br>±7 | 30<br>9<br>±7 | 337<br>±7 | 36<br>5<br>±7 | 39<br>3<br>±7 | 42<br>1<br>±7 | 44<br>9<br>±7 | 47<br>7<br>±7 | 50<br>5<br>±7 | 533<br>±7 | 547<br>±7 | | 631<br>±7 |
| Study day<br>infusion <sup>4, 9</sup> | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Initial screening<br>consent<br>(optional) <sup>10</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Full informed consent <sup>11</sup> | X | | | | | | | | | | | | | | | | | | | | | | X <sup>12</sup> | X <sup>12</sup> | | |
| Randomization | | | | X | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility criteria | X | X | X | X | | | | | | | | | | | | | | | | | | | X <sup>13</sup> | X <sup>13</sup> | | |
| NIA-AA<br>criteria review | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history | X | X | X | X | | | | | | | | | | | | | | | | | | | | | | |
| Body weight | X | | | X | X | X | X | | | X | | | | X | | | X | | | X | | | X | X | | X |
| Height | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy<br>test <sup>14</sup> | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Follicle-<br>stimulating<br>hormone <sup>15</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Alcohol/drug<br>screen | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| HbA1c | X | | | | | | | | | | | | | | | | | | | | | | | | | |

| | Se<br>Perio | Baselin<br>creenin<br>od <sup>1, 2</sup> w<br>ays <sup>3</sup> of<br>1 | ıg<br>ithin | | | | | | | | | ] | Placebo | -Cont | olled l | Period <sup>4</sup> | ı | | | | | | | | UV for<br>Change in<br>AD<br>Medication | FUV <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>7</sup> | | 90 |
| Study Day | S1 | S2 | S3 <sup>8</sup> | 1 | 29<br>±7 | 57<br>±<br>7 | 85<br>±7 | 11<br>3<br>±7 | 14<br>1<br>±7 | 169<br>±7 | 19<br>7<br>±7 | 22<br>5<br>±7 | 25<br>3<br>±7 | 28<br>1<br>±7 | 30<br>9<br>±7 | 337<br>±7 | 36<br>5<br>±7 | 39<br>3<br>±7 | 42<br>1<br>±7 | 44<br>9<br>±7 | 47<br>7<br>±7 | 50<br>5<br>±7 | 533<br>±7 | 547<br>±7 | | 631<br>±7 |
| HIV <sup>16</sup> /hepatitis tests | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | | X |
| Neurological examination | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | | X |
| 12-lead paper<br>ECG <sup>18</sup> | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | | X |
| Vital signs <sup>19</sup> | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Hematology/<br>clinical<br>chemistry/<br>urinalysis | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | | X |
| Blood sample<br>for anti-<br>BIIB092 Ab <sup>4</sup> | | | | X | X | | | | | X | | | | | | X | | | | | | | X | | | X |
| Blood sample<br>for BIIB092<br>concentration | | | | X | X <sup>20</sup> | X | X <sup>20</sup> | X | X | $X^{20}$ | X | | | | | X <sup>20</sup> | | | X | | | | $X^{20}$ | | | X |

| | S<br>Peri | Baselin<br>creenin<br>od <sup>1, 2</sup> w<br>lays <sup>3</sup> of<br>1 | ng<br>ithin | | | | | | | | | ] | Placebo | o-Cont | rolled 1 | Period <sup>4</sup> | ı | | | | | | | | UV for<br>Change in<br>AD<br>Medication | FUV <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>7</sup> | | 90 |
| Study Day | S1 | S2 | S38 | 1 | 29<br>±7 | 57<br>±<br>7 | 85<br>±7 | 11<br>3<br>±7 | 14<br>1<br>±7 | 169<br>±7 | 19<br>7<br>±7 | 22<br>5<br>±7 | 25<br>3<br>±7 | 28<br>1<br>±7 | 30<br>9<br>±7 | 337<br>±7 | 36<br>5<br>±7 | 39<br>3<br>±7 | 42<br>1<br>±7 | 44<br>9<br>±7 | 47<br>7<br>±7 | 50<br>5<br>±7 | 533<br>±7 | 547<br>±7 | | 631<br>±7 |
| Blood sample<br>for plasma and<br>serum<br>biomarkers <sup>4</sup> | | | | X | | | | X | | | | | | | | X | | | X | | | | X | | | |
| Brain MRI <sup>22</sup> | | X | | | | | | | | | X | | | | | | X | | | | | | | $X^{23}$ | | |
| CDR <sup>28</sup> | X | | | | | | | | | X | | | | | | | X | | | | | | | X | X | |
| NPI-10 | | | X | | | | | | | X | | | | | | | X | | | | | | | X | | |
| ISLR | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| ISLT | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | X | |
| DKEFS<br>Category<br>Fluency and<br>Letter Fluency<br>tests | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | | |
| DSST | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | | |

| | S<br>Peri | Baselin<br>creening<br>od <sup>1, 2</sup> w<br>lays <sup>3</sup> of | ng<br>⁄ithin | | | | | | | | | ] | Placebo | o-Cont | rolled 1 | Period | 4 | | | | | | | | UV for<br>Change in<br>AD<br>Medication | FUV <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>7</sup> | | 90 |
| Study Day | S1 | S2 | S38 | 1 | 29<br>±7 | 57<br>±<br>7 | 85<br>±7 | 11<br>3<br>±7 | 14<br>1<br>±7 | 169<br>±7 | 19<br>7<br>±7 | 22<br>5<br>±7 | 25<br>3<br>±7 | 28<br>1<br>±7 | 30<br>9<br>±7 | 337<br>±7 | 36<br>5<br>±7 | 39<br>3<br>±7 | 42<br>1<br>±7 | 44<br>9<br>±7 | 47<br>7<br>±7 | 50<br>5<br>±7 | 533<br>±7 | 547<br>±7 | | 631<br>±7 |
| Trails A | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | | |
| eCog (39-item version) | | | X | | | | | | | | X | | | | | | | X | | | | | | X | | |
| ADAS-Cog<br>13 <sup>29</sup> | | X | X | | | | | | | X | | | | | | | X | | | | | | | X | X | |
| FAQ | | | X | | | | | | | X | | | | | | | X | | | | | | | X | X | |
| ADCS-ADL | | | X | | | | | | | X | | | | | | | X | | | | | | | X | X | |
| C-SSRS <sup>29</sup> | | X | X | | | | | | | X | | | | | | | X | | | | | | | X | | |
| MMSE | X | | | | | | X | | | X | | | | X | | | X | | | | X | | | X | X | |
| RUD-Lite | | | X | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | | |
| ZBI | | | X | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | | |
| QoL-AD | | | X | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | | |
| AE reporting | | | | | • | | | | | | Monito | or and r | ecord c | ontinu | ously b | eginnir | ng on S | tudy Da | y 1 at | the star | t of do | sing | | | | |
| SAE reporting | | | | | | | | | | | | Mor | nitor an | d recor | d conti | nuousl | y throu | ghout tl | ne stud | y | | | | | | |
| Concomitant<br>therapy and<br>procedures<br>reporting | | | | Monitor and record continuously throughout the study Monitor and record continuously throughout the study | | | | | | | | | | | | | | | | | | | | | | |

| | Serie<br>Perie | Baselin<br>creenin<br>od <sup>1, 2</sup> w<br>ays <sup>3</sup> of<br>1 | ng<br>vithin | | | | | | | | | | | | | UV for<br>Change in<br>AD<br>Medication | FUV <sup>6</sup> | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>7</sup> | 90 |
| Study Day | S1 | S2 | S38 | 1 | 29<br>±7 | 57<br>±<br>7 | 85<br>±7 | 11<br>3<br>±7 | 14<br>1<br>±7 | 169<br>±7 | 19<br>7<br>±7 | 22<br>5<br>±7 | 25<br>3<br>±7 | 28<br>1<br>±7 | 30<br>9<br>±7 | 337<br>±7 | 36<br>5<br>±7 | 39<br>3<br>±7 | 42<br>1<br>±7 | 44<br>9<br>±7 | 47<br>7<br>±7 | 50<br>5<br>±7 | 533<br>±7 | <b>547</b> ±7 | 631<br>±7 |
| Tobacco use<br>status <sup>31</sup> | | | | Monitor and record continuously throughout the study | | | | | | | | | | | | | | | | | | | | | |

| Cooperative Study – Activities of Daily Living; AE = adverse event; Cacle; Cooperative Study – Activities of Daily Living; AE = adverse event; Cacle; |
|---|
| Function System; DSST = Digit Symbol Substitution Test; ECG = electrocardiogram; eCog = Everyday Cognition; EOS = end of study; EOT = end of treatment; ET = early termination; FAQ = Functional Activities Questionnaire; FUV = Follow-up Visit; HbA1c = glycosylated hemoglobin; HIV = human mmunodeficiency virus; ISLR = International Shopping List Test Delayed Recall; ISLT = International Shopping List Test mmediate Recall; LTE = long-term extension; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; IAA-AA = National Institute on Aging-Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory 10; PK = pharmacokinetic; QoL-AD = Quality of Life in Alzheimer's Disease; RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; DV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| ET = early termination; FAQ = Functional Activities Questionnaire; FUV = Follow-up Visit; HbA1c = glycosylated hemoglobin; HIV = human mmunodeficiency virus; ; ISLR = International Shopping List Test Delayed Recall; ISLT = International Shopping List Test mmediate Recall; ; LTE = long-term extension; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; NIA-AA = National Institute on Aging-Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory 10; ; QoL-AD = Quality of Life in Alzheimer's Disease; ; RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; JV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| immunodeficiency virus; ; ISLR = International Shopping List Test Delayed Recall; ISLT = International Shopping List Test mediate Recall; ; LTE = long-term extension; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; NIA-AA = National Institute on Aging-Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory 10; ; QoL-AD = Quality of Life in Alzheimer's Disease; ; RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; JV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| mmediate Recall; ; LTE = long-term extension; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; NIA-AA = National Institute on Aging-Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory 10; ; QoL-AD = Quality of Life in Alzheimer's Disease; ; QUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; JV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| NIA-AA = National Institute on Aging-Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory 10; (CV) |
| CK = pharmacokinetic; ; QoL-AD = Quality of Life in Alzheimer's Disease; ; QuD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; UV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; JV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| JV = unscheduled visit; ZBI = Zarit Burden Interview The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1 S3). However |
| <u></u> |
| TIME IN THE STATE OF THE STATE |
| additional screening visits may be needed for some procedures, e.g., MRI In addition, it may sometimes be necessary for participants to return for |
| repeat assessments (e.g., if the MRI scan does not pass the quality control process). Brain MRI (S2) will only be performed after the participant has met the |
| eligibility criteria and has acceptable laboratory tests from Visit S1. |

The clinical assessments performed during Visit S1 are to be administered in the order specified: 1) MMSE; 2) neuropsychological tests in the following order: ISLT, DSST, Trails A, Category Fluency and Letter Fluency tests from the DKEFS, ISLR; 3) CDR. Note that the Visit S1 results from CDR, ISLT/ISLR, and MMSE will be used to determine participant eligibility; Visit S3 ISLT assessments will provide baseline measures. At Visit S3, the clinical assessments will be administered as follows: 1) neuropsychological tests in the following order: ISLT, DSST, Trails A, Category Fluency and Letter Fluency tests from the DKEFS; 2) ADAS-Cog 13; 3) QoL-AD.

It is recommended that all the screening procedures be completed within 65 days; however, the overall Screening Period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate (

). The following screening assessments should be repeated if the Screening Period is >65 days: confirmation of eligibility criteria,

Protocol 251AD201 Version 4

abbreviated medical history, and physical examination. In addition, some cognitive and /or safety assessments may require repeating depending on the duration of the screening window extension, in discussion with the Medical Monitor.

<sup>4</sup> All assessments and blood collection during dosing days will be performed prior to infusion, unless otherwise specified. Doses should be administered at least 21 days apart.

- <sup>5</sup> Participants should have a UV prior to the initiation of, change in dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition. See Section 11.4.1.2 for details.
- <sup>6</sup> Participants who complete the Treatment Period and do not enter an extension study are to return to the study site for a Follow-up Safety Visit at Week 90. Participants who discontinue study treatment and withdraw from the study early are to have a Follow-up Safety Visit 14 weeks after the final dose. Participants who discontinue study treatment prematurely are to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Section 10.1 and Section 10.3 for details.
- All participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures. These participants should be encouraged to attend at least the Week 24. Week 52, and Week 78 visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely will also be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Section 10.1 for details. Participants who withdraw from the study prematurely are to return to the study site for an ET Visit and ET assessments. If the withdrawn participant has discontinued treatment within 3 months of the previous primary efficacy assessment (CDR) and no significant changes in cognitive status are suspected by the Investigator, the clinical efficacy assessments specified in the ET visit are not required; the study site should notify the Sponsor in such cases. An MRI scan should be performed if withdrawal occurs ≥6 months after the previous MRI. Blood for biomarker analysis should be collected if the participant withdraws ≥4 weeks after the previous sample was collected.

See Section 10.3 for details.

Visit S3 all clinical assessments must be scheduled within 7 days before Study Day 1 or performed at Study Day 1 before randomization, The overall Screening Period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate

All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

<sup>10</sup>Participants and the participants' partners/informants or their legally authorized representatives, in countries where applicable laws allow, may sign this optional form for an initial screening which allows administration of the CDR, MMSE, ISLT/ISLR, DKEFS Category Fluency and Letter Fluency tests, DSST, and Trails A to determine eligibility based on cognitive assessments. The order of assessments is as specified in footnote 2.

<sup>11</sup>All participants and the participants' partners/informants or their legally authorized representatives, in countries where applicable laws allow, must sign this full informed consent, including those who have previously signed the optional initial screening consent and have met the eligibility criteria based on cognitive assessments.

Protocol 251AD201

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

<sup>12</sup>All participants and the participants' partners/informants or their legally authorized representatives, in countries where applicable laws allow must reconsent by signing this full informed consent before participating in the general during the LTE period.

Version 4

<sup>13</sup>Only for participants entering the LTE period.

<sup>14</sup>Pregnancy testing is required for women of childbearing potential only; for these participants, a serum pregnancy test is to be performed at Screening and EOS (or ET) Visits, and a urine pregnancy test is to be performed at every dosing visit.

<sup>15</sup>Women who report postmenopausal status at Visit S1 must have a follicle-stimulating hormone test at that visit to confirm that they are not of childbearing potential.

16 To be performed based upon Investigator assessment of HIV risk factors. The requirement for testing during Screening may be omitted if it is not permitted by local regulations.



<sup>18</sup>Triplicate 12-lead (paper) ECGs will be obtained at each specified timepoint. ECGs are to be performed in triplicate, with each ECG performed about 1 minut apart and before blood draws on appropriate days. In addition, triplicate ECGs will also be performed 1 hour after the end of infusion on Study Day 1 only. Each ECG must be performed after the participant has been resting (supine) for 10 minutes. ECGs will be read by a central reading facility. Clinical significance of potential ECG abnormalities will be determined by the Investigator.

<sup>19</sup>Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate and will be measured with the participant supine and after the participant has been resting for at least 10 minutes. In addition, blood pressure and heart rate will be measured after the participant has been standing for ≥2 minutes at the following timepoints: preinfusion and 1 hour (±15 minutes) after the end of infusion on Days 1, 29, 57, and 85. Three separate SBP/DBP readings at least 15 minutes apart will be made at the Screening Visit to determine eligibility. Single vital sign readings will be obtained at other timepoints.

<sup>20</sup>Two samples must be obtained: 1 sample taken before infusion and 1 sample taken at ≤15 minutes after the end of infusion.

<sup>21</sup>The results are not required for randomization.

<sup>22</sup>Brain MRI may include, but will not be limited to, the following sequences: 3D T1 weighted, fluid attenuated inversion recovery, T2\* weighted, diffusion weighted imaging, and proton density/T2 weighted MRI. For further details on MRI sequences, please see the procedural manual for MRI. To occur after cognitive testing has concluded for the Screening Period. After randomization, the visit date for this MRI can vary by ±10 days from the specified visit day.

<sup>23</sup>Sites should schedule the Week 78 MRI within 10 days prior to the Week 78 visit where possible to allow for MRI results to be available before participants enter the LTE at Week 80.



<sup>&</sup>lt;sup>28</sup>It is recommended that postbaseline CDR assessments be conducted at the same time of day at which the baseline assessment was performed to avoid diurnal variation. The rater who conducts the CDR for a participant/informant cannot complete any other rating scales for that same participant/partner or be the study site coordinator and will be blinded to all other study-related data.

<sup>&</sup>lt;sup>29</sup>During the Screening Period, ADAS-Cog 13 and C-SSRS are scheduled at Visit S2; however, they may be performed at Visit S1, if more convenient per site and participant's availability. If ADAS-Cog 13 and C-SSRS assessments are performed at Visit S1, all other clinical assessments should be performed before ADAS-Cog 13, followed by C-SSRS.

<sup>&</sup>lt;sup>31</sup>Participants' tobacco use status will be assessed while collecting information on concomitant therapies.

Table 2: Schedule of Activities for Week 80 Through Week 128 of the Long-Term Extension Period

| | Long-Term Extension Period | | | | | | | | | | | UV for Change in AD Medication <sup>1</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 80 | 84 | 88 | 92 | 96 | 100 | 104 | 108 | 112 | 116 | 120 | 124 | 128 | |
| Study Days (±7 days) | 561 | 589 | 617 | 645 | 673 | 701 | 729 | 757 | 785 | 813 | 841 | 869 | 897 | |
| Study day infusion <sup>2, 3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Eligibility criteria | X | | | | | | | | | | | | | |
| Pregnancy test <sup>4</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Physical examination | | | | X | | | X | | | | | | X | |
| Body weight | | | | X | | | X | | | | | | X | |
| Neurological examination | | | | X | | | X | | | | | | X | |
| 12-lead paper ECG <sup>6</sup> | | | | | | | X | | | | | | X | |
| Vital signs <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Hematology/clinical chemistry/ urinalysis | | | | | | X | | | | | | X | | |
| Blood sample for anti-<br>BIIB092 Ab | X | | | | | | X | | | X | | | | |
| Blood sample for<br>BIIB092 concentration | X | | | | | | X | | | X | | | | |
| Blood sample for plasma and serum biomarker | | | | | | | | | | X | | | | |
| Brain MRI <sup>8</sup> | | | | | | | X | | | | | | | |
| CDR <sup>12</sup> | | | | | | | X | | | | | | X | X |

| | Long-Term Extension Period | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 80 | 84 | 88 | 92 | 96 | 100 | 104 | 108 | 112 | 116 | 120 | 124 | 128 | |
| Study Days (±7 days) | 561 | 589 | 617 | 645 | 673 | 701 | 729 | 757 | 785 | 813 | 841 | 869 | 897 | |
| NPI-10 | | | | | | | X | | | | | | X | |
| ISLT | | | | | | | | X | | | | | | X |
| DKEFS Category<br>Fluency and Letter<br>Fluency tests | | | | | | | | X | | | | | | |
| DSST | | | | | | | | X | | | | | | |
| Trails A | | | | | | | | X | | | | | | |
| eCog (39-item version) | | | | | | | | X | | | | | | |
| ADAS-Cog 13 | | | | | | | X | | | | | | X | X |
| FAQ | | | | | | | X | | | | | | X | X |
| ADCS-ADL | | | | | | | X | | | | | | X | X |
| C-SSRS | | | | | | | X | | | | | | X | |
| MMSE | | | | | | | X | | | | | | X | X |
| RUD-Lite | | | | | | | | | | | | X | | |
| ZBI | | | | | | | | | | | | X | | |
| QoL-AD | | | | | | | | | | | | X | | |
| AE reporting | | | | | | Monitor a | and record co | ntinuously th | nroughout the | LTE period | | | | |
| SAE reporting | | Monitor and record continuously throughout the LTE period | | | | | | | | | | | | |
| Concomitant therapy and procedures reporting | | Monitor and record continuously throughout the LTE period | | | | | | | | | | | | |
| Tobacco use status <sup>14</sup> | | | | | | Monitor a | and record co | ntinuously th | nroughout the | LTE period | | | | |
| Ab = antibodies; AD = Cooperative Study - A Columbia-Suicide Sev Substitution Test; ECC Functional Activities | Activitie<br>verity R<br>G = elec | es of Dai<br>ating Sc<br>etrocardi | ly Livin<br>ale; DBI | g; AE = a $P = diasto$ | adverse ev<br>olic blood | vent; CDR<br>pressure; Cognition; | t = Clinica<br>DKEFS =<br>EOS = en | l Dementi<br>Delis-Kap<br>d of study; | a Rating Solan Execut | cale;<br>ive Funct<br>d of treat | ion Syste | em; DSST<br>= early t | ; C-S<br>T = Digit<br>termination | SRS =<br>Symbol |

LTE = long-term extension; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; NPI-10 = Neuropsychiatric Inventory 10; ; PK = pharmacokinetics; QoL-AD = Quality of Life in Alzheimer's Disease; RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; UV = unscheduled visit; ZBI = Zarit Burden Interview.

- 1 Participants should have a UV prior to the initiation of, change in dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition. See Section 11.4.1.2 for details.
- <sup>2</sup> All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.
- <sup>3</sup> All assessments and blood collection during dosing days will be performed prior to infusion, unless otherwise specified. Doses should be administered at least 21 days apart.
- <sup>4</sup> Pregnancy testing is required for women of childbearing potential only; for these participants, a serum pregnancy test is to be performed at EOS [or ET] Visits, and a urine pregnancy test is to be performed at every dosing visit.



- Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate and will be measured with the participant supine and after the participant has been resting for at least 10 minutes. In addition, blood pressure and heart rate will be measured after the participant has been standing for >2 minutes at the following timepoints: preinfusion and 1 hour (±15 minutes) after the end of infusion on Weeks 80, 84, 88, and 92. Single vital sign readings will be obtained at other timepoints.
- <sup>8</sup> Brain MRI may include, but will not be limited to, the following sequences: 3D T1 weighted, fluid attenuated inversion recovery, T2\* weighted, diffusion weighted imaging, and proton density/T2 weighted MRI. For further details on MRI sequences, please see the procedural manual for MRI. During the LTE period, the visit date for the MRI can vary by  $\pm 10$  days from the specified visit day.

12 It is recommended that postbaseline CDR assessments be conducted at the same time of day at which the baseline assessment was performed to avoid diurnal variation. The rater who conducts the CDR for a participant/informant cannot complete any other rating scales for that same participant/partner or be the study site coordinator and will be blinded to all other study-related data.

<sup>14</sup>Participants' tobacco use status will be assessed while collecting information on concomitant therapies.

Table 3: Schedule of Activities for Week 132 Through Week 176 of the Long-Term Extension Period

| | | | | | | Lo | ng-Term Ext | ension Period | | | | | UV for Change in AD Medication <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 132 | 136 | 140 | 144 | 148 | 152 | 156 | 160 | 164 | 168 | 172 | 176 | |
| Study Days (±7 days) | 925 | 953 | 981 | 1009 | 1037 | 1065 | 1093 | 1121 | 1149 | 1177 | 1205 | 1233 | |
| Study day infusion <sup>2, 3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| Pregnancy test <sup>4</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| Physical examination | | | | | | X | | | | | | X | |
| Body weight | | | | | | X | | | | | | X | |
| Neurological examination | | | | | | X | | | | | | X | |
| 12-lead paper ECG <sup>6</sup> | | | | | | X | | | | | | X | |
| Vital signs <sup>7</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| Hematology/clinical chemistry/ urinalysis | | | | | X | | | | | | X | | |
| Blood sample for anti-<br>BIB092 Ab | | | | | | | X | | | | | X | |
| Blood sample for<br>BIIB092 concentration | | | | | | | X | | | | | X | |
| Blood sample for plasma and serum biomarker | | | | | | | X | | | | | | |
| Brain MRI <sup>8</sup> | | | | | | | X | | | | | | |
| CDR <sup>12</sup> | | | | | | X | | | | | | X | X |
| NPI-10 | | | | | | X | | | | | | | |
| ISLT | X | | | | | | X | | | | | | X |
| DKEFS Category | X | | | | | | X | | | | | | |

| | | Long-Term Extension Period | | | | | | | | | UV for Change in<br>AD Medication <sup>1</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 132 | 136 | 140 | 144 | 148 | 152 | 156 | 160 | 164 | 168 | 172 | 176 | |
| Study Days (±7 days) | 925 | 953 | 981 | 1009 | 1037 | 1065 | 1093 | 1121 | 1149 | 1177 | 1205 | 1233 | |
| Fluency and Letter<br>Fluency tests | | | | | | | | | | | | | |
| DSST | X | | | | | | X | | | | | | |
| Trails A | X | | | | | | X | | | | | | |
| eCog (39-item version) | X | | | | | | X | | | | | | |
| ADAS-Cog 13 | | | | | | X | | | | | | X | х |
| FAQ | | | | | | X | | | | | | | х |
| ADCS-ADL | | | | | | X | | | | | | X | X |
| C-SSRS | | | | | | X | | | | | | X | |
| MMSE | | | | | | X | | | | | | Х | Х |
| RUD-Lite | | | | | | | | | | | X | | |
| ZBI | | | | | | | | | | | X | | |
| QoL-AD | | | | | | | | | | | X | | |
| AE reporting | | | | | | Monito | or and record o | continuously th | hroughout the L | TE period | | | |
| SAE reporting | | | | | | Monito | or and record o | continuously th | hroughout the L | TE period | | | |
| Concomitant therapy and procedures reporting | ** * * * | | | | | | | | | | | | |
| Tobacco use status <sup>14</sup> | Tobacco use status <sup>14</sup> Monitor and record continuously throughout the LTE period | | | | | | | | | | | | |
| Ab = antibodies; AD =<br>Cooperative Study – A<br>Suicide Severity Ratin<br>ECG = electrocardiog<br>Questionnaire; | Activitie<br>g Scale<br>ram; eC | s of Dai<br>; DBP =<br>og = Ev | ily Livin<br>diastol<br>eryday | ng; AE =<br>ic blood<br>Cognition; | adverse<br>pressure<br>on; EOS =<br>ISLT = I | event; CD<br>; DKEFS =<br>= end of st<br>nternation | R = Clinica<br>= Delis-Kap<br>udy; EOT =<br>al Shopping | al Dementia<br>plan Execut<br>end of trea<br>List Test I | a Rating Scal<br>tive Function<br>atment; ET =<br>immediate R | le;<br>n System; D<br>= early term<br>ecall; | OSST = Dig<br>nination; FA | ; C-SS<br>it Symbol Su<br>AQ = Function<br>; LTE | SRS = Columbia<br>abstitution Test; |
| extension; $MMSE = N$ | Iini-Me | ntal Sta | te Exam | ination; | MRI = 1 | nagnetic re | esonance in | | I-10 = Neuro | | | | |


; PK = pharmacokinetic;

UV = unscheduled visit; ZBI = Zarit Burden Interview.

RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A;

; QoL-AD = Quality of Life in Alzheimer's Disease;


- 1 Participants should have a UV prior to the initiation of, change in dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition. See Section 11.4.1.2 for details.
- <sup>2</sup> All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.
- <sup>3</sup> All assessments and blood collection during dosing days will be performed prior to infusion, unless otherwise specified. Doses should be administered at least 21 days apart.
- <sup>4</sup> Pregnancy testing is required for women of childbearing potential only; for these participants, a serum pregnancy test is to be performed at EOS (or ET) Visits, and a urine pregnancy test is to be performed at every dosing visit.



- Triplicate 12-lead (paper) ECGs will be obtained at each specified timepoint. ECGs are to be performed in triplicate, with each ECG performed about 1 minute apart and before blood draws on appropriate days. Each ECG must be performed after the participant has been resting (supine) for 10 minutes. ECGs will be read by a central reading facility. Clinical significance of potential ECG abnormalities will be determined by the Investigator.
- <sup>7</sup> Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate and will be measured with the participant supine and after the participant has been resting for at least 10 minutes. Single vital sign readings will be obtained.
- <sup>8</sup> Brain MRI may include, but will not be limited to, the following sequences: 3D T1 weighted, fluid attenuated inversion recovery, T2\* weighted, diffusion weighted imaging, and proton density/T2 weighted MRI. For further details on MRI sequences, please see the procedural manual for MRI. During the LTE period, the visit date for the MRI can vary by  $\pm 10$  days from the specified visit day.



<sup>12</sup>It is recommended that postbaseline CDR assessments be conducted at the same time of day at which the baseline assessment was performed to avoid diurnal variation. The rater who conducts the CDR for a participant/informant cannot complete any other rating scales for that same participant/partner or be the study site coordinator and will be blinded to all other study-related data.

<sup>&</sup>lt;sup>14</sup>Participants' tobacco use status will be assessed while collecting information on concomitant therapies.

Table 4: Schedule of Activities for Week 180 Through Week 238 or Follow-Up Visit of the Long-Term Extension Period

| | | | | | | ] | Long-Te | rm Exter | sion Peri | iod | | | | | UV for Change<br>in AD<br>Medication <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 180 | 184 | 188 | 192 | 196 | 200 | 204 | 208 | 212 | 216 | 220 | 224/<br>EOT | 226/<br>EOS<br>or ET <sup>2</sup> | 238/FUV (14<br>weeks After<br>Last Dose) <sup>3</sup> | |
| Study Days (±7 days) | 1261 | 1289 | 1317 | 1345 | 1373 | 1401 | 1429 | 1457 | 1485 | 1513 | 1541 | 1569 | 1583 | 1667 | |
| Study day infusion <sup>4, 5</sup> | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Pregnancy test <sup>6</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Physical examination | | | | | | X | | | | | | | X | X | |
| Body weight | | | | | | X | | | | | | | X | X | |
| Neurological examination | | | | | | X | | | | | | | X | X | |
| 12-lead paper ECG <sup>8</sup> | | | | | | X | | | | | | | X | X | |
| Vital signs <sup>9</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Hematology/clinical chemistry/ urinalysis | | | | | X | | | | | | X | | X | X | |
| Blood sample for anti-BIIB092 Ab | | | | | X | | | | | | | X | | X | |
| Blood sample for BIIB092 concentration | | | | | X | | | | | | | X | | X | |
| Blood sample for plasma and serum biomarker | | | | | X | | | | | | | X | | | |
| Brain MRI <sup>10</sup> | | | | | | | | | | | | | X | | |
| CDR <sup>14</sup> | | | | | | X | | | | | | | X | | X |
| NPI-10 | | | | | | X | | | | | | | X | | |
| ISLT | | | | | | | X | | | | | | X | | X |
| DKEFS Category Fluency and Letter<br>Fluency tests | | | | | | | X | | | | | | X | | |

| | Long-Term Extension Period | | | | | | | | | | | | | | UV for Change<br>in AD<br>Medication <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 180 | 184 | 188 | 192 | 196 | 200 | 204 | 208 | 212 | 216 | 220 | 224/<br>EOT | 226/<br>EOS<br>or ET <sup>2</sup> | 238/FUV (14<br>weeks After<br>Last Dose) <sup>3</sup> | |
| Study Days (±7 days) | 1261 | 1289 | 1317 | 1345 | 1373 | 1401 | 1429 | 1457 | 1485 | 1513 | 1541 | 1569 | 1583 | 1667 | |
| DSST | | | | | | | X | | | | | | X | | |
| Trails A | | | | | | | X | | | | | | X | | |
| eCog (39-item version) | | | | | | | X | | | | | | X | | |
| ADAS-Cog 13 | | | | | | X | | | | | | | X | | X |
| FAQ | | | | | | X | | | | | | | X | | X |
| ADCS-ADL | | | | | | X | | | | | | | X | | X |
| C-SSRS | | | | | | X | | | | | | | X | | |
| MMSE | | | | | | X | | | | | | | X | | X |
| RUD-Lite | | | | | | | | | | | | | X | | |
| ZBI | | | | | | | | | | | | | X | | |
| QoL-AD | | | | | | | | | | | | | X | | |
| AE reporting | | | | | | Mon | itor and r | ecord cor | ntinuously | through | out the L | TE period | | | |
| SAE reporting | | | | | | Mon | itor and r | ecord cor | ntinuously | / through | out the L | TE period | | | |
| Concomitant therapy and procedures reporting | | Monitor and record continuously throughout the LTE period Monitor and record continuously throughout the LTE period | | | | | | | | | | | | | |
| Tobacco use status <sup>16</sup> | | Monitor and record continuously throughout the LTE period | | | | | | | | | | | | | |

Ab = antibodies; AD = Alzheimer's disease; ADAS-Cog 13 = Alzheimer's Disease Assessment Scale-Cognitive (13 item); ADCS-ADL = Alzheimer's Disease Cooperative Study – Activities of Daily Living; AE = adverse event; CDR = Clinical Dementia Rating Scale; C-SSRS = Columbia-Suicide Severity Rating Scale; DBP = diastolic blood pressure; DKEFS = Delis-Kaplan Executive Function System; DSST = Digit Symbol Substitution Test; ECG = electrocardiogram; eCog = Everyday Cognition; EOS = End of Study; EOT = End of Treatment; ET = early termination; FAQ = Functional Activities Questionnaire; FUV = Follow-up Visit; State =

; QoL-AD = Quality of Life in Alzheimer's Disease; RUD-Lite = Resource Utilization in Dementia-Lite Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; UV = unscheduled visit; ZBI = Zarit Burden Interview.


- 1 Participants should have a UV prior to the initiation of, change in dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition. See Section 11.4.1.2 for details.
- <sup>2</sup> All participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures. These participants should be encouraged to attend at least the Week 80, 104, 116, 128, 152, 156, 176, 196, 200, 224, and 226/EOS Visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely will also be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Section 10.1 for details. Participants who withdraw from the study prematurely are to return to the study site for an ET Visit and ET assessments. If the withdrawn participant has discontinued treatment within 3 months of the previous primary efficacy assessment (CDR) and no significant changes in cognitive status are suspected by the Investigator, the clinical efficacy assessments specified in the ET Visit are not required; the study site should notify the Sponsor in such cases. An MRI scan should be performed if withdrawal occurs ≥6 months after the previous MRI. Blood for biomarker analysis should be collected if the participant withdraws ≥4 weeks after the previous sample was collected.

ee Section 10.3 for details.

- Participants who discontinue study treatment and withdraw from the study early are to have a Follow-up Safety Visit (FUV) 14 weeks after the final dose. Participants who discontinue study treatment prematurely are to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Section 10.1 and Section 10.3 for details.
- <sup>4</sup> All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.
- <sup>5</sup> All assessments and blood collection during dosing days will be performed prior to infusion, unless otherwise specified. Doses should be administered at least
- <sup>6</sup> Pregnancy testing is required for women of childbearing potential only; for these participants, a serum pregnancy test is to be performed at EOS (or ET) Visits, and a urine pregnancy test is to be performed at every dosing visit.

Triplicate 12-lead (paper) ECGs will be obtained at each specified timepoint. ECGs are to be performed in triplicate, with each ECG performed about 1 minute apart and before blood draws on appropriate days. Each ECG must be performed after the participant has been resting (supine) for 10 minutes. ECGs will be read by a central reading facility. Clinical significance of potential ECG abnormalities will be determined by the Investigator.

<sup>9</sup> Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate and will be measured with the participant supine and after the participant has been resting for at least 10 minutes. Single vital sign readings will be obtained.


<sup>&</sup>lt;sup>10</sup>Brain MRI may include, but will not be limited to, the following sequences: 3D T1 weighted, fluid attenuated inversion recovery, T2\* weighted, diffusion weighted imaging, and proton density/T2 weighted MRI. For further details on MRI sequences, please see the procedural manual for MRI. During the LTE period, the visit date for the MRI can vary by ±10 days from the specified visit day.

<sup>&</sup>lt;sup>14</sup>It is recommended that postbaseline CDR assessments be conducted at the same time of day at which the baseline assessment was performed to avoid diurnal variation. The rater who conducts the CDR for a participant/informant cannot complete any other rating scales for that same participant/partner or be the study site coordinator and will be blinded to all other study-related data.

<sup>&</sup>lt;sup>16</sup>Participants' tobacco use status will be assessed while collecting information on concomitant therapies.

## 6. STUDY OBJECTIVES AND ENDPOINTS

| Placebo-Controlled Period Objectives and Endpoints | |
|---|---|
| Primary Objective | Primary Endpoint |
| To evaluate the safety and tolerability of BIIB092 in participants with MCI due to AD or with mild AD | Incidence of AEs and SAEs during the placebo-controlled period |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of multiple doses of BIIB092 in slowing cognitive and functional impairment in participants with MCI due to AD or with mild AD. This is the primary efficacy objective | Change from Baseline over time at Week 78 on the CDR-SB. This is the primary efficacy endpoint |
| To evaluate the immunogenicity of BIIB092 after multiple doses in participants with MCI due to AD or with mild AD | Incidence of anti-BIIB092 antibodies in serum over time up to Week 90 |
| Exploratory Objectives | Exploratory Endpoints |
| To assess the effect of BIIB092 on the clinical progression of AD | Changes from Baseline over time up to Week 78 on the Mini-Mental State Examination (MMSE), International Shopping List Test Immediate Recall (ISLT), Category Fluency and Letter Fluency tests from the Delis-Kaplan Executive Function System (DKEFS), Digit Symbol Substitution Test (DSST), Trail Making Test, Part A (Trails A), Everyday Cognition (eCog), Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL), Functional Activities Questionnaire (FAQ), Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog 13 [13 item]), and Neuropsychiatric Inventory-10 (NPI-10) |
| To assess the effect of BIIB092 on changes in caregiver burden and participant quality of life | Changes from Baseline over time up to<br>Week 68 on the Zarit Burden Interview (ZBI)<br>and Quality of Life for Alzheimer's Disease<br>(QoL-AD) |


| To assess the effect of BIIB092 on resource utilization | Resource Utilization in Dementia-Lite<br>Version (RUD-Lite) results over time up to<br>Week 68 |
|---|---|
| To assess BIIB092 PK in serum in participants with MCI due to AD or with mild AD | Trough serum BIIB092 concentrations and end-of-infusion serum BIIB092 concentrations from the samples collected at the visits indicated in the Schedule of Activities |
| To assess the effect of BIIB092 on biomarkers in blood | Changes from Baseline over time up to<br>Week 76 on blood levels of disease-related<br>biomarkers, including but not limited to, tau<br>and other markers of neurodegenerative<br>disease |
| To assess the effect of BIIB092 on brain structure | Changes from Baseline over time up to<br>Week 78 on MRI morphometric measures,<br>including volume and cortical thickness of<br>certain brain areas |

| Long-Term Extension Period Objectives and Endpoints | |
|---|---|
| Primary Objective | Primary Endpoint |
| To evaluate the long-term safety and tolerability of BIIB092 in participants with MCI due to AD or with mild AD | Incidence of AEs and SAEs over the placebo-controlled period and long-term extension (LTE) period of the study |
| <b>Exploratory Objectives</b> | Exploratory Endpoints |
| To further evaluate the immunogenicity of BIIB092 after multiple doses in participants with MCI due to AD or with mild AD | Incidence of anti-BIIB092 antibodies in serum over time up to Week 238 |
| To further assess the effect of BIIB092 on disease progression as measured by fluid and radiological biomarkers, as well as additional clinical and health outcomes | Changes over the placebo-controlled period and LTE period on the CDR-SB, MMSE, ISLT, Category Fluency and Letter Fluency tests from the DKEFS, DSST, Trails A, eCog, ADCS-ADL, FAQ, ADAS-Cog 13 (13-item), and NPI-10 |
| | Changes over the placebo-controlled<br>period and LTE period on the ZBI,<br>QoL-AD, and RUD-Lite |
| | Changes over the placebo- <u>controlled</u> period and LTE period on MRI brain morphometric measures |
| To assess BIIB092 PK in serum in participants with MCI due to AD or with mild AD | Trough serum BIIB092 concentrations<br>from serum samples collected at the<br>visits indicated in the Schedule of<br>Activities |
| | • |

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

This clinical study will collect samples that, under separate optional consent, may be used for future scientific and genetic research. Specific objectives related to this future research have not been determined.

### 7. STUDY DESIGN

See Figure 1 for a schematic of the study design.

## 7.1. Study Overview

This is a Phase 2, randomized, double-blind, placebo-controlled study of BIIB092 in participants aged 50 to 80 years inclusive, with MCI due to AD or mild AD according to National Institute on Aging-Alzheimer's Association criteria (NIA-AA) [McKhann 2011]. Participants must have

a CDR Memory Box score of ≥0.5.

The study will be conducted in a parallel-group design, with 3 BIIB092 dose groups (including 4 BIIB092 doses) and a placebo group. Approximately 528 participants were planned to be randomized across approximately 100 study sites globally. Due to fast recruitment, the study was over-enrolled and 654 participants have been randomized. Participants will be stratified by , region, baseline disease stage (MCI or mild AD), and baseline AD medication use.

The study consists of a double-blind, placebo-controlled period and a dose-blinded LTE period. The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. For participants who complete both the placebo-controlled period and the LTE period, the total study duration will be approximately 247 weeks. The placebo-controlled period comprises a Screening Period of approximately 9 weeks (65 days), a Treatment Period of 76 weeks, and for participants not entering the LTE period, an End-of-Study (EOS) Visit at Week 78 and a Follow-up Safety Visit at Week 90. or approximately 14 weeks after the last dose of study treatment. However, the Screening Period for the placebo-controlled period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate ( ). At the end of the placebo-controlled period, participants who meet the LTE entry criteria may enter the dose-blinded LTE period. The LTE period comprises an LTE Screening Period of approximately 4 weeks starting at Week 76, a 144-week Treatment Period, an EOS Visit at Week 226, and a Follow-up Safety Visit at Week 238, or approximately 14 weeks after the last dose of study treatment.

Randomized participants will receive 1 of the following study treatments by IV infusion every 4 weeks, starting on Study Day 1 during the placebo-controlled period:

• low-dose BIIB092 - 125 mg once every 4 weeks or 375 mg once every 12 weeks and placebo at the other 4-week dosing visits to maintain the treatment blind (88 participants planned in total, 44 per regimen)

- medium-dose BIIB092 600 mg once every 4 weeks (88 participants planned)
- high-dose BIIB092 2000 mg once every 4 weeks (176 participants planned)
- placebo (176 participants planned)

Overall, participants will have a 2:1 chance of being randomized to BIIB092 or to placebo during the placebo-controlled period.

During the LTE period, participants who were randomized to receive BIIB092 during the placebo-controlled period will continue to receive BIIB092 at the dose they were randomly assigned. Participants receiving placebo during the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period. The BIIB092 dose concentration (i.e. low, medium, or high) to which participants are assigned to receive during LTE period may be changed based on emerging data from the BIIB092 clinical development program.

Throughout the study, all participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

Investigators, study staff (except for a designated Pharmacist/Technician), and study participants and their families, caregivers, and legal representatives will be blinded to the participants' randomized treatment assignments and, during the LTE period, the BIIB092 dose.



The schedule of study assessments is presented in Section 5.

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease



 $A\beta$  = amyloid beta; AD = Alzheimer's disease; EOS = End of Study; LTE = long-term extension; MCI = mild cognitive impairment; N = planned number of participants; Q4W = once every 4 weeks; Q12W = once every 12 weeks

Note: Overall, participants will have a 2:1 chance of being randomized to BIIB092 versus placebo during the placebo-controlled period, and all participants will receive BIIB092 during the dose-blinded LTE period. Note: The study comprises a double-blind, placebo-controlled period and an LTE period. The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. The total study duration for participants who complete both the placebo-controlled period and the LTE period will be approximately 247 weeks. The double-blind placebo-controlled period comprises a Screening Period of approximately 9 weeks (65 days), a Treatment Period of 76 weeks, and for participants not entering the LTE period, an EOS Visit at Week 78 and a Follow-up Safety Visit at Week 90, or approximately 14 weeks after the last dose of study treatment. The LTE period comprises an LTE Screening Period of approximately 4 weeks starting at Week 76, a 144-week Treatment Period starting at Week 80, an EOS Visit at Week 226, and a Follow-up Safety Visit at Week 238, or approximately 14 weeks after the last dose of study treatment.

#### 7.2. **Study Duration for Participants**

Figure 1:

**Study Design** 

The study consists of a double-blind, placebo-controlled period and a dose-blinded LTE period. The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. The total study duration for participants who

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

complete both the placebo-controlled period and the LTE period will be approximately 247 weeks.

#### **Placebo-Controlled Period**

Participation in the double-blind, placebo-controlled period will be approximately 99 weeks, which includes the Screening Period of approximately 9 weeks, the 76-week Treatment Period, the EOS Visit at Week 78, and for participants not entering the LTE period, a Follow-up Safety Visit at Week 90, or approximately 14 weeks after the last dose of study treatment (see Table 1). It is recommended that all the screening procedures be completed within 65 days; however, the overall Screening Period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate (

Participants will have approximately 25 outpatient clinic visits:

- Participant eligibility will be determined at up to 3 visits during the Screening Period (Screening Visits 1, 2, and 3).
- On Study Day 1, eligible participants will be randomized, have scheduled assessments per the Schedule of Activities (Table 1), and receive the first infusion of randomized study treatment.
- Participants will return to the clinic at 4-week intervals during the Treatment Period for infusions of study treatment and study assessments (Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, and 76). The last dose of study treatment will be administered at Week 76 (End-of-Treatment Visit).
- For a participant who completes the Treatment Period at Week 76, there will be an EOS Visit at Week 78 for final study assessments of the placebo-controlled period. A Follow-up Safety Visit will occur at Week 90 (14 weeks after the last dose of study treatment is administered), unless the participant elects to enter an extension study following the Week 78 Visit. Final visit scheduling and procedures are described in Section 10.1 for participants who discontinue study treatment prematurely but remain in the study and in Section 10.3 for participants who withdraw from the study.

All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

#### **Long-Term Extension Period**

Participants who meet the LTE inclusion and exclusion criteria will be eligible to enter the dose-blinded LTE period, which includes the LTE Screening Period of approximately 4 weeks starting at Week 76, the 144-week Treatment Period starting at Week 80, the EOS Visit at Week 226, and the Follow-up Visit at Week 238 (see Table 1, Table 2, Table 3, and Table 4).

Participants will have approximately 39 outpatient clinic visits during the LTE period:

- Participant eligibility will be determined at Week 76 or Week 78 of the placebo-controlled period and confirmed at Week 80 of the LTE period.
- At the Week 80 Visit, eligible participants will have scheduled assessments per the Schedule of Activities (Table 2) and receive the first infusion of BIIB092 during the LTE period. All participants receiving placebo in the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period.
- Participants will return to the clinic at 4-week intervals during the Treatment Period for infusions of study treatment and study assessments (Table 2, Table 3, and Table 4).
- The last dose of study treatment will be administered at Week 224 (End-of-Treatment Visit). The EOS Visit will occur at Week 226 and the Follow-up Visit at Week 238.

All participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

See Section 5 for the details of the activities to be conducted at each visit.




The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease



## 7.4. Study Stopping Rules

Dosing may be terminated by the Sponsor at the recommendation of the independent Data Monitoring Committee (DMC), based exclusively on safety and tolerability data or following futility analysis, or at the discretion of the Sponsor; therefore, there are no study-specific stopping rules defined in this protocol.

Biogen will notify Investigators when the study is to be placed on hold, completed, or terminated.

# 7.5. End of Study

The end of study is last participant, last visit.

#### 8. SELECTION OF PARTICIPANTS

#### 8.1. Inclusion Criteria

To be eligible to participate in this study, candidates must meet the following eligibility criteria at Screening, or at the timepoint specified in the individual eligibility criterion listed:

- Ability of the participant to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations. In countries where applicable laws allow, the participant's informant/study partner and/or legally authorized representative may provide informed consent in lieu of the participant's signature.
- 2. Age 50 to 80 years old, inclusive, at the time of informed consent.
- 3. All women of childbearing potential and all men with female partners of childbearing potential must practice highly effective contraception during the study and for 6 months (24 weeks) after their last dose of study treatment. For further details of contraceptive requirements for this study, see Section 15.5. Female participants should not become pregnant during the study and for 6 months (24 weeks) after their last dose of study treatment. It is recommended that male participants should not father children during their participation in the study and for 6 months (24 weeks) after their last dose of study treatment.
- 4. Must have a gradual and progressive change in memory function over more than 6 months, reported by the participant and/or his/her informant/study partner.
- 5. Must meet all of the clinical criteria for MCI due to AD or mild AD according to the NIA-AA [McKhann 2011], and in addition must have the following at Screening Visit 1:
  - ISLT or ISLR score 1 SD below the age-adjusted normative mean
  - CDR global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD
  - MMSE score of 22 to 30 (inclusive)
  - CDR Memory Box score of ≥0.5
- Apart from a clinical diagnosis of MCI due to AD or mild AD, the participant must be in good health as determined by the Investigator, based on medical history and screening assessments.

7.

8. Body weight ≥43 kg (95 lbs) and ≤120 kg (265 lbs).

9. Must have 1 informant/study partner who, in the Investigator's judgment, has frequent and sufficient contact with the participant (at least 10 hours/week) as to be able to provide accurate information about the participant's cognitive and functional abilities. The study partner must agree to accompany the participant to clinic visits and/or be available by phone at designated times to provide information to the Investigator and study staff about the participant (and to attend in-person clinic visits that require partner input for scale completion) and must agree to monitor the participant's administration of any prescribed medications. A study partner should be available for the duration of the study, and the participation of the same study partner for the duration of the study is encouraged. The study partner must be literate and give informed consent.



## 8.2. Exclusion Criteria

Candidates will be excluded from study entry if any of the following exclusion criteria exist at Screening, or at the timepoint specified in the individual criterion listed:

#### Medical history

- History of, or positive test result at Screening Visit 1 for, human immunodeficiency virus (HIV). HIV testing may be completed based upon Investigator assessment of HIV risk factors. The requirement for testing during Screening may be omitted if it is not permitted by local regulations.
- 2. Current hepatitis C infection (defined as positive hepatitis C virus [HCV] antibody and detectable HCV ribonucleic acid [RNA]). Participants with positive HCV antibody and undetectable HCV RNA are eligible to participate in the study (United States Centers for Disease Control and Prevention).


3. Current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or total hepatitis B core antibody [anti-HBc]). Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as

- negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study.
- 4. Any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment (e.g., current history of substance abuse, uncontrolled vitamin B12 deficiency or abnormal thyroid function, stroke or other cerebrovascular condition, Parkinson's disease, Lewy body dementia, or frontotemporal dementia), or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns.
- 5. History of seizures within 10 years prior to Screening Visit 1 or history of epileptic syndrome (except for history of febrile seizures in childhood).
- 6. History within 5 years prior to Screening Visit 1 of a serious infectious disease affecting the brain (including neurosyphilis, Lyme disease, meningitis, or encephalitis), or severe head trauma, including concussions, that may have resulted in a protracted loss of consciousness.
- 7. Presence of clinically significant and/or unstable psychiatric illness, in the Investigator's opinion (e.g., bipolar affective disorder), within the 6 months prior to Screening Visit 1.
- 8. Any documented prior history of chronic schizophrenia.
- 9. History of long-term major depression or bipolar affective disorder with an active episode in the past 5 years.
- 10. Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening Visit 1.
- 11. Brain MRI performed at Screening Visit 2 (centrally read) that shows evidence of any of the following:
  - Acute or subacute hemorrhage.
  - Prior macrohemorrhage (defined as >1 cm in diameter on T2\* sequence) unless it can be documented that the finding is not due to an underlying structural or vascular abnormality (i.e., finding does not suggest participant is at risk of recurrent hemorrhage).
  - More than 5 microhemorrhages (defined as  $\leq 1$  cm in diameter on T2\* sequence).

- Cortical infarct (including cerebellar infarct) [defined as >1.5 cm in diameter] or any infarct in the hippocampus.
- >2 lacunar infarcts (defined as ≤1.5 cm in diameter).
- Superficial siderosis in >1 zone.
- Superficial siderosis >1 cm<sup>3</sup> in any zone.
- Diffuse white matter disease as defined by a score of 3 on the Age-Related White Matter Changes scale [Wahlund 2001].
- Any finding that, in the opinion of the Investigator, might be a contributing cause of the participant's dementia, might pose a risk to the participant, or might prevent a satisfactory MRI assessment.
- 12. History of bleeding disorder or predisposing conditions, blood clotting, or clinically significant abnormal results on coagulation profile at Screening, as determined by the Investigator.
- 13. Presence of diabetes mellitus that, in the judgment of the Investigator, is not controlled or adequately managed.
- 14. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening Visit 1.
- 15. Clinically significant 12-lead ECG abnormalities, as read by the central reading facility and determined by the Investigator.
- 16. History of severe allergic or anaphylactic reactions.
- 17. Known allergy to BIIB092 or a history of hypersensitivity to any of the inactive ingredients in the drug product (see the Investigator's Brochure for information on the BIIB092 clinical formulation).
- 18. Any major surgery within 12 weeks of Screening Visit 1 or during the Screening Period.
- 19. Uncontrolled hypertension defined as: an average of 3 systolic blood pressure (SBP)/diastolic blood pressure (DBP) readings >165/100 mm Hg at Screening (blood pressure measurements exceeding these limits may be repeated as warranted by the Investigator, but values must be within the specified limits for the participant to be eligible for the study), or persistent SBP/DBP readings >180/100 mm Hg within 12 weeks prior to randomization (Study Day 1) that, in the opinion of the Investigator, are indicative of chronic uncontrolled hypertension.

Version 4

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

- 20. History of premalignant or malignant disease. Exceptions to premalignant disease exclusions may be made after discussion with the Sponsor. The following exceptions may be made for malignant disease exclusions after discussion with the Sponsor:
  - Participants with cancers in remission ≥5 years prior to Screening Visit 1.
  - Participants with a history of excised or treated basal cell or squamous carcinoma of the skin.
  - Participants with localized prostate cancer with treatment cycles that completed at least 6 months prior to Screening Visit 1.
- 21. Indication of impaired liver function as shown by an abnormal liver function profile at Screening (e.g., repeated values of aspartate aminotransferase [AST] and alanine aminotransferase [ALT]  $\ge 2 \times 10^{-5}$  the upper limit of normal [ULN]).
- 22. Indication of impaired renal function at Screening (e.g., repeated values of creatinine and blood urea nitrogen [BUN] ≥1.5 × ULN or estimated glomerular filtration rate <45 mL/minute/1.73 m² and corroborating medical history and physical examination).
- 23. History or evidence of an autoimmune disorder considered clinically significant by the Investigator or requiring long-term use of systemic corticosteroids or other immunosuppressants.
- 24. History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunological, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
- 25. Recent history (within 1 year of Screening Visit 1) of alcohol or substance abuse as determined by the Investigator, a positive urine drug (due to nonprescription drug) or alcohol test at Screening, or use of cannabinoids (prescription or recreational).
- 26. Clinically significant systemic illness or serious infection (e.g., pneumonia, septicemia) within 30 days prior to or during the Screening Period.

#### Medications

- 27. Use of allowed medications for chronic conditions at doses that have not been stable for at least 4 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.
- 28. Use of AD medications (including but not limited to donepezil, rivastigmine, galantamine, tacrine, and memantine) at doses that have not been stable for at least 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.

29. Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participant at higher risk for AEs, or impair the participant's ability to perform cognitive testing or complete study procedures.

## 30. Use of the following medications:

- Long-acting benzodiazepines (e.g., valium), except for sedation prior to MRI scans for those participants requiring sedation and should not be administered within 24 hours prior to cognitive testing.
- Short/medium-acting benzodiazepines (e.g., alprazolam, lorazepam, oxazepam, temazepam) except if used chronically for sleep and on a stable dose for 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1, or used short term on an as-needed basis. May not be taken within 12 hours prior to cognitive testing.
- Sedating antihistamines if taken within 12 hours prior to cognitive testing.
   Nonsedating antihistamines (e.g., fexofenadine, cetirizine) are allowed.
- Anticonvulsants that have significant effects on cognition per the Investigator's opinion and/or anticonvulsants used for treatment of seizures. Anticonvulsants with limited cognitive effects, such as lamotrigine, pregabalin, levetiracetam for treatment of pain, and other non-epilepsy indications are allowed if, in the opinion of the Investigator, they are not producing sedation or contributing to cognitive impairment. The participant must have been on a stable dose for 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.
- Antidepressants that may, in the Investigator's opinion, affect the participant's cognition (e.g., tricyclic antidepressants). Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. Use of antidepressants is allowed if at stable doses for 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.
- High-dose antipsychotics used on a regular basis. Low doses of atypical and typical antipsychotics if used on an as-needed basis or if used at a stable dose for 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1. The definition of "low dose" and "high dose" should be judged by the Investigator, and the Medical Monitor can be consulted if needed.
- Anticholinergics such as benztropine. Anticholinergics for bladder control with limited cognitive effects are permitted but should be avoided if possible.
- Prior use of levodopa or anti-Parkinsonian medications including dopaminergic agents, amantadine, selegiline, benztropine, and monoamine oxidase (MAO) inhibitors prescribed for the treatment of Parkinsonism or Parkinson's disease.

 Use of prescription narcotic medications within 4 weeks prior to Screening Visit 1. After randomization, short-term use of prescription narcotics is allowed for specific situations (e.g., after surgical procedures) and if administered at least 24 hours prior to cognitive testing.

 Use of any drug of abuse, including but not limited to, amphetamine, cannabis, cocaine, opiate, propoxyphene, methadone, methaqualone, phencyclidine, or barbiturates.

When necessary, the Medical Monitor should be contacted with any questions.

- 31. Vaccinations within 10 days prior to randomization (Study Day 1).
- 32. Prior participation in any active or passive immunotherapy study targeting Aβ or tau, unless documentation of receipt of placebo is available.
- 33. Last administration of  $\beta$ -secretase inhibitors and  $\gamma$ -secretase inhibitors in a study within 3 months or 5 half-lives (whichever is longer) prior to Screening unless documentation of receipt of placebo is available.
- 34. Participation in any study involving an investigational treatment targeting tau, unless documentation of receipt of placebo is available.
- 35. Participation within the 12 months prior to Screening Visit 1 in a study of any other agent(s) not included in exclusion criteria 32, 33, and 34 with a purported disease-modifying effect in AD, unless documentation of receipt of placebo is available.



#### Study Procedures

37. Contraindications to having a brain MRI (e.g., MRI-incompatible pacemaker; MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed). If the MRI compatibility of implanted devices is unknown, the participant must be excluded from the study.



40. Has had or plans to have exposure to experimental radiation within 12 months prior to Screening Visit 1 such that regional radiation dosimetry limits would be exceeded by participating in this study.



 Lack of good venous access, such that IV drug delivery or multiple blood draws would be precluded.

#### Other

- 43. Female participants who are pregnant or currently breastfeeding or who plan to become pregnant.
- 44. Participant living in an organized care facility with extensive intervention and/or support of daily living activities (e.g., a nursing home).
- 45. Blood donation (≥1 unit) within 1 month prior to Screening Visit 1.
- 46. Current enrollment or plan to enroll in any other interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered.
- 47. Inability to comply with study requirements.
- 48. Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the participant unsuitable for the study.

## 8.3. Inclusion Criteria for Long-Term Extension Period

To be eligible to participate in the LTE period, participants must meet the following eligibility criteria at Week 76 or 78 and confirmed at Week 80:

 Ability of the participant to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations. In countries where applicable laws allow, the participant's informant/study partner and/or legally authorized representative may provide informed consent in lieu of the participant's signature (same as above in Section 8.1).

- 2. Participant must have completed the placebo-controlled period of the study, including the Week 78 Visit. Participant must have taken at least 14 doses of study treatment and not have missed more than 4 consecutive doses of study treatment. Participants who do not meet these criteria may enter the LTE period only with the Sponsor's approval.
- 3. All women of childbearing potential and all men with female partners of childbearing potential must practice highly effective contraception during the study and for 6 months (24 weeks) after their last dose of study treatment. For further details of contraceptive requirements for this study, see Section 15.5. Female participants should not become pregnant during the study and for 6 months (24 weeks) after their last dose of study treatment. It is recommended that male participants should not father children during their participation in the study and for 6 months (24 weeks) after their last dose of study treatment (same as above in Section 8.1).
- 4. Medically able to undergo the study procedures and to adhere to the visit schedule at the time of study entry into the LTE period, as determined by the Investigator. Apart from a clinical diagnosis of MCI due to AD or mild AD, the participant must be in good health as determined by the Investigator, based on medical history.
- 5. Must have the ability to comply with procedures for protocol-related tests.
- 6. Must have 1 informant/study partner who, in the Investigator's opinion, has frequent and sufficient contact with the participant (at least 10 hours/week) as to be able to provide accurate information about the participant's cognitive and functional abilities. The study partner must agree to accompany the participant to clinic visits and/or be available by phone at designated times to provide information to the Investigator and study staff about the participant (and to attend in-person clinic visits that require partner input for scale completion) and must agree to monitor the participant's administration of any prescribed medications. A study partner should be available for the duration of the study, and the participation of the same study partner for the duration of the study is encouraged. The study partner must be literate and give informed consent (same as above in Section 8.1).

# 8.4. Exclusion Criteria for Long-Term Extension Period

Participants will be excluded from entering the LTE period if any of the following exclusion criteria exist at Week 76 or 78 and confirmed at Week 80:

- 1. Any medical or psychiatric contraindication or clinically significant abnormality that, in the opinion of the Investigator, will substantially increase the risk associated with the participant's participation in and completion of the study.
- 2. Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the participant unsuitable for the study (same as above in Section 8.2).



#### 9. SCREENING AND RANDOMIZATION

#### 9.1. Screening



The necessary order of the screening assessments is provided in Table 1.

During the first screening visit, under a separate (optional) initial consent process, participants can complete the cognitive scales (including the CDR, MMSE, DKEFS Category and Letter Fluency tests, DSST, Trails A, and ISLT/ISLR). This initial cognitive screening is intended to reduce the burden on participants and study sites by avoiding unnecessary testing if participants do not meet key inclusion criteria. If the participant meets inclusion criteria for the CDR, MMSE, and ISLT/ISLR, then the full consent process must be completed prior to the administration of further screening assessments. Participants may also proceed directly to the full consent process, which would allow the administration of all screening assessments.

Participant eligibility for the study will be determined during up to 3 screening visits in the approximately 9-week (65-day) Screening Period preceding randomization during the placebo-controlled period.

It is recommended that all the screening procedures for the placebo-controlled period be completed within 65 days; however, the overall Screening Period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate ( ). The following screening tests should be repeated if the Screening Period is >65 days: confirmation of eligibility criteria, abbreviated medical history, and physical examination. In addition, some cognitive assessments and/or safety assessments may require repeating depending on the duration of the screening window extension, in discussion with the Medical Monitor.

Screen failures are defined as participants who provide informed consent but are not subsequently randomized. If a participant is considered a screen failure, the reasons for exclusion must be documented in the participant's source documents and on the screening log. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAEs.



Participants or their legally authorized representatives, in countries where applicable laws allow, who chose to participate in the LTE period must provide informed consent before any screening tests are performed (see Section 17.3).

Participants who chose to participate in the LTE period can be screened at Week 76 or Week 78 per Table 1, and confirmation of eligibility will be checked at Week 80 per Table 2.

## 9.2. Randomization

Participants will be randomized on Study Day 1 after all screening and baseline assessments have been completed and after the Investigator has verified that the participants are eligible per criteria in Sections 8.1 and 8.2. Participants will be assigned a unique identification number that will be used on study-related documents pertaining to the participant. Any participant identification numbers that are assigned will not be reused even if the participant does not receive treatment. Rescreened participants will be assigned a new number.



Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease



Participants who are participating in the LTE period and who were randomized to receive placebo during the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period. Participants who were randomized to receive BIIB092 during the placebo-controlled period will continue to receive BIIB092 at the dose they were randomly assigned.

See the Study Reference Guide for details on randomization.

## 9.3. Blinding Procedures

This study consists of a randomized, double-blind, placebo-controlled period, followed by a dose-blinded LTE period with all participants receiving BIIB092.

During the double-blind, placebo-controlled period, all study staff who conduct participant assessments will be blinded to the participant treatment assignments. The individuals conducting the rating scale assessments should remain blinded to treatment assignment as well as to participant care management and only have access to the information necessary to carry out their responsibilities. As a placebo match is not provided by the Sponsor for the study (see Section 12.2), unblinded pharmacy staff are required to manage all aspects of study treatment receipt, dispensing, and preparation. To maintain the study blind, it is imperative that participant treatment assignments are not shared with the participants, their families, or any member of the blinded study team, either at the study site or at Biogen or its representatives, except the unblinded pharmacist (or designee), the unblinded pharmacy monitor, and the unblinded CRO or Biogen safety staff. Members of the DMC will also be unblinded.



All participants will receive infusions of study treatment at 4-week intervals during the double-blind placebo-controlled period. Those participants who are randomized to receive BIIB092 once every 12 weeks versus once every 4 weeks will receive placebo at the other 4-week dosing intervals to maintain the treatment blind. See Section 11.1 for details of the treatment regimens.

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

For the LTE period, the dose information must remain restricted. The study staff, the individuals conducting the rating scale assessments, and the Investigator should remain blinded to dose assignment and only have access to the information necessary to carry out their responsibilities. To maintain the study blind, it is imperative that dose information is not shared with the participants, their families, or any member of the blinded study team, either at the study site or at Biogen or its representatives, except the unblinded pharmacist (or designee), the unblinded pharmacy monitor, and the unblinded CRO or Biogen safety staff.

Once the clinical study report has been finalized, if unblinding will not jeopardize the results of ongoing related studies, Biogen will provide the randomization codes to Investigators, who then can inform their participants about the treatment received.

# 10. DISCONTINUATION OF STUDY TREATMENT AND WITHDRAWAL OF PARTICIPANTS FROM THE STUDY

## **10.1.** Discontinuation of Study Treatment

A participant must permanently discontinue study treatment for any of the following reasons:

- The participant becomes pregnant. Study treatment must be discontinued immediately, and the pregnancy must be reported according to the instructions in Section 15.4.1.
- The participant withdraws consent to continue study treatment.
- The participant experiences a medical emergency that necessitates permanent discontinuation of study treatment or unblinding of the participant's treatment assignment.
- The participant experiences an AE or SAE that does not resolve or requires continued treatment that meets exclusionary criteria.
- The participant experiences a severe infusion reaction
- At the discretion of the Investigator for medical reasons.
- At the discretion of the Investigator or the Sponsor for noncompliance with the terms of the protocol.

The primary reason for discontinuation of study treatment must be recorded in the participant's case report form (CRF).

All participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures for the period in which they discontinued treatment (i.e., placebo-controlled or LTE). Participants who discontinue treatment during the placebo-controlled period should be encouraged to attend at least the Week 24, Week 52, and Week 78/EOS Visits and who discontinue treatment during the LTE should be encouraged to attend at least the Week 80, 104, 116, 128, 152, 156, 176, 196, 200, 224, and 226/EOS Visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely, regardless of the treatment period, will be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Table 1, Table 2, Table 3, and Table 4 for the Schedule of Activities.

## 10.2. Lost to Follow-Up

Participants will be considered lost to follow-up if they repeatedly fail to return for scheduled visits and cannot be contacted by the study site.

The following actions must be taken if a participant fails to return to the study site for a required study visit:

- The study site must attempt to contact the participant and reschedule the missed visit
  as soon as possible and counsel the participant on the importance of maintaining the
  assigned visit schedule and ascertain whether the participant wishes to and/or should
  continue in the study.
- In cases in which the participant is deemed lost to follow-up, the Investigator or
  designee must make every effort to regain contact with the participant. These contact
  attempts should be documented in the participant's medical record.
- Should the participant continue to be unreachable, that participant will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

## 10.3. Withdrawal of Participants From Study

Participants must be withdrawn from the study for any one of the following reasons:

- The participant withdraws consent.
- The participant enrolls into another interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered.
- The participant is unwilling or unable to comply with the protocol.

The primary reason for the participant's withdrawal from the study must be recorded in the participant's CRF.

Participants who withdraw from the study prematurely are to return to the study site for an Early Termination (ET) Visit and assessments as indicated in Table 1, after the reason for withdrawal is identified. For such participants, clinical efficacy assessments specified at the ET Visit are not required if the participant discontinues treatment within 3 months of the previous primary efficacy (CDR) assessment and no significant changes in cognitive status are suspected by the Investigator; the study site should notify the Sponsor in such cases. An MRI scan should be performed if withdrawal occurs ≥6 months after the previous MRI. Blood for biomarker analysis should be collected if the participant withdraws ≥4 weeks after the previous sample was collected.
Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

Participants who are withdrawn from the study are also to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment.



#### 11. STUDY TREATMENT USE

# 11.1. Regimen

Follow the Directions for Handling and Administration (DHA).

#### 11.1.1. Placebo-Controlled Period

Randomized, blinded study treatment will be administered by IV infusion at the study site once every 4 weeks, beginning on Study Day 1 and continuing through Week 76, for a total of 20 infusions (see Table 1).

Participants will receive 1 of the following treatment regimens:

- low-dose BIIB092 125 mg once every 4 weeks or 375 mg once every 12 weeks and placebo at the other 4-week dosing visits to maintain the treatment blind
- medium-dose BIIB092 600 mg once every 4 weeks
- high-dose BIIB092 2000 mg once every 4 weeks
- placebo

#### 11.1.2. Long-Term Extension Period

In the LTE period, participants will receive BIIB092 beginning at Week 80 and continuing through Week 224. Participants who were randomized to receive BIIB092 during the placebo-controlled period will continue to receive BIIB092 at the dose they were randomly assigned. Participants randomized to receive placebo during the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) during the LTE period.

#### 11.2. Modification of Dose and/or Treatment Schedule

See Section 11.2.1 (Dose Suspension) and Section 11.2.2 (Infusion Interruption).

Dosing visits are not to be skipped, but may be delayed within the time window specified in the Schedule of Activities (Table 1). Doses should be administered at least 21 days apart, per the regimen of dosing once every 4 weeks. If the dosing interval cannot be met, the dose administration schedule should be assessed by the study Medical Monitor.

Participants should be carefully monitored for infusion reactions during dose administration. If an acute infusion reaction is observed, the participant should be managed per Section 11.2.2 (Infusion Interruption).

#### 11.2.1. Dose Suspension

The independent DMC will review safety data on an ongoing basis to ensure safe and proper treatment of participants. The DMC, based on the nature, frequency, and/or severity of an AE(s), may recommend dose suspension or dose termination. See Section 19.2 for additional information about the independent DMC.

#### 11.2.2. Infusion Interruption

The IV administration infusion time for all treatment groups is 1 to 2 hours at approximately 100 mL/hour. No premedications should be used prior to the start of study treatment infusion unless discussed with the Medical Monitor in advance and written documentation is received from Biogen authorizing the use of the premedication.

- If any mild or moderate infusion-related reaction occurs during an infusion, the infusion may be slowed or interrupted and appropriate treatment per local standards of care may be given, at the discretion of the Investigator (or designee). Based on the clinical response, the Investigator or designee will determine if the infusion may be resumed/continued, in consultation with the Medical Monitor as needed. If the infusion is resumed/continued, the infusion rate should not exceed the original infusion rate (see the DHA for infusion rate information).
- If a severe infusion-related reaction occurs during an infusion, the participant should be permanently discontinued from treatment and appropriate supportive care must be initiated in accordance with local practice.

Criteria for determining the severity of events are described in Section 15.2.3.

Discussion with the Medical Monitor can occur as needed, and it should not delay management of the medical emergency.

See Section 15.3 for reporting of AEs and Section 10 for discontinuation of study treatment.

# 11.3. Compliance

Compliance with treatment dosing is to be monitored and recorded by study site staff.

# 11.4. Concomitant Therapy and Procedures

#### 11.4.1. Concomitant Therapy

A concomitant therapy is any drug or substance administered between Screening Visit 1 and the Follow-up Safety Visit.

The use of concomitant therapies or procedures as defined below must be recorded on the participant's CRF, according to instructions for CRF completion. AEs related to administration of these therapies or procedures must be documented on the appropriate CRF.

The Medical Monitor should be contacted with any questions about allowed or disallowed concomitant therapies.

#### 11.4.1.1. Allowed Concomitant Therapy

- Medications for chronic conditions are allowed during the study as long as the participant has been on a stable dose of the medication(s) for 4 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.
- AD medications (including, but not limited to, donepezil, rivastigmine, galantamine, tacrine, and memantine) are allowed provided that participants are receiving a stable dose for at least 8 weeks prior to Screening Visit 1 and remains stable during the Screening Period up to Study Day 1 and during the study.
- Vaccination with live or attenuated vaccine is allowed during the study. Administration of any vaccine or booster should not occur <10 days prior to any dosing visit and for 10 days after a dosing visit.

#### 11.4.1.2. Disallowed Concomitant Therapy

Any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participant at higher risk for AEs, or impair the participant's ability to perform cognitive testing or complete study procedures are disallowed.

Use of the following medications is disallowed:

- Long-acting benzodiazepines (e.g., valium), except for sedation prior to MRI scans for those participants requiring sedation and should not be administered within 24 hours prior to cognitive testing.
- Short/medium-acting benzodiazepines (e.g., alprazolam, lorazepam, oxazepam, temazepam) except if used chronically for sleep and on a stable dose for 8 weeks prior to Screening Visit 1 and during Screening or used short term on an as-needed basis. May not be taken within 12 hours prior to cognitive testing.
- Sedating antihistamines if taken within 12 hours prior to cognitive testing. Nonsedating antihistamines (e.g., fexofenadine, cetirizine) are allowed.
- Anticonvulsants that have significant effects on cognition per the Investigator's opinion and/or anticonvulsants used for treatment of seizures. Anticonvulsants with limited cognitive effects, such as lamotrigine, pregabalin, levetiracetam for treatment of pain, and other non-epilepsy indications are allowed if, in the opinion of the Investigator, they are not producing sedation or contributing to cognitive impairment. The participant must have been on a stable dose for 8 weeks prior to Screening Visit 1 and during the Screening Period up to Study Day 1.

- Antidepressants that may, in the Investigator's opinion, affect the participant's
  cognition (e.g., tricyclic antidepressants). Mild depression or depressive mood
  arising in the context of AD are not criteria for exclusion. Use of antidepressants is
  allowed if at stable doses for 8 weeks prior to Screening Visit 1 and during the
  Screening Period up to Study Day 1.
- High-dose antipsychotics used on a regular basis. Low doses of atypical and typical
  antipsychotics if used on an as-needed basis or if used at a stable dose for 8 weeks
  prior to Screening Visit 1 and during the Screening Period up to Study Day 1. The
  definition of "low dose" and "high dose" should be judged by the Investigator, and
  the Medical Monitor can be consulted if needed.
- Anticholinergics such as benztropine. Anticholinergics for bladder control with limited cognitive effects are permitted but should be avoided if possible.
- Prior use of levodopa or anti-Parkinsonian medications include dopaminergic agents, amantadine, selegiline, benztropine, and MAO inhibitors prescribed for the treatment of Parkinsonism or Parkinson's disease.
- Use of prescription narcotic medications within 4 weeks prior to Screening Visit 1.
   After randomization, short-term use of prescription narcotics if not for specific situations (e.g., after surgical procedures) and if administered within 24 hours prior to cognitive testing.
- Use of any drug of abuse, including but not limited to, amphetamine, cannabis, cocaine, opiate, propoxyphene, methadone, methaqualone, phencyclidine, or barbiturates.
- Immunosuppressive drugs (including systemic corticosteroids). Local corticosteroids may be permitted at Sponsor discretion.
- Parenteral Ig, blood products, plasma derivatives, plasma exchange, and plasmapheresis.
- Any investigational drug other than BIIB092.



Participants should be instructed to continue the usual medications they were on at enrollment (see allowed concomitant therapy above) and to avoid starting any new medications or herbal preparations during the study period, as these may confound the results of the study. However, medically indicated medication or treatment should not be withheld. Participants should inform the Investigator of any change in medication. The change should be reviewed by the Investigator and, if needed, the Medical Monitor to determine whether the participant's study treatment should be suspended. Medications used to treat AEs would not result in automatic withdrawal. Biogen may be consulted if required.

Participants should have an unscheduled visit (UV) prior to the initiation of, change in dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition (see Table 1, Table 2, Table 3, and Table 4).

#### 11.4.2. Concomitant Procedures

Concomitant procedures are allowed only when deemed necessary by the participant's healthcare provider. A concomitant procedure is any therapeutic intervention (e.g., surgery/biopsy, physical therapy) or diagnostic assessment (e.g., blood gas measurement, bacterial cultures) performed between the time the participant is enrolled in the study and until the participant's final clinic visit (including the Follow-up Safety Visit), unless the participant is being followed for study-related toxicity.

#### 11.4.3. Tobacco Use

Participants' tobacco use status will be monitored continuously throughout the study and should be assessed while collecting information on concomitant therapies.

#### 11.5. Continuation of Treatment

The participant may elect to enter the LTE following the Week 78 Visit. No further provisions are made for access to the study treatment otherwise.

#### 12. STUDY TREATMENT MANAGEMENT

Study treatment will be manufactured, handled, and stored in accordance with applicable Good Manufacturing Practice.

Study site staff should follow the DHA for specific instructions on the handling, preparation, administration, and disposal of the study treatment. The DHA will also describe the masking of the IV bags of study treatment (both BIIB092 and placebo) to maintain the treatment blind. The DHA supersedes all other references (e.g., protocol or Investigator's Brochure).

Study treatment must be dispensed only by a pharmacist or appropriately qualified staff. Study treatment is to be dispensed only to participants enrolled in this study. Once study treatment is prepared for a participant, it can be administered only to that participant. Study treatment vials are for one-time use only; do not use any study treatment remaining in the vial for another participant.

#### 12.1. BIIB092

BIIB092 is a humanized, hinge-stabilized IgG4 monoclonal antibody derived from a mouse IgG1 monoclonal antibody (IPN002). BIIB092 is produced from cell culture using a Chinese hamster ovary cell line.

BIIB092 is supplied as a liquid drug product in glass vials containing an extractable dose as per the DHA.

The contents of the BIIB092 label will be in accordance with all applicable regulatory requirements. BIIB092 should not be used after the expiration date.

#### 12.1.1. BIIB092 Preparation

The individual preparing BIIB092 should carefully review the instructions provided in the DHA.

BIIB092 is to be administered by IV infusion following dilution with 0.9% sodium chloride solution.

If the packaging is damaged, or if there is anything unusual about the appearance or attributes of the vials or study treatment, do not use the study treatment. The vial in question should be saved at the study site and the problem immediately reported to Biogen.

#### **12.1.2.** BIIB092 Storage

Study treatment must be stored in a secure location.

Vials of BIIB092 are to be stored at 2°C to 8°C (36°F to 46°F), in a locked storage container with limited access. BIIB092 should be protected from light and freezing.


The administration of BIIB092 by infusion must be completed within 24 hours of preparation. If not used immediately, the infusion solution may be stored under refrigeration at 2°C to 8°C (36°F to 46°F) for up to 24 hours, and a maximum of 4 hours of the total 24-hour period can be at room temperature with exposure to room light. The maximum 4-hour period under room temperature and room light conditions includes the product administration time.

For the most up-to-date storage requirements, follow the instructions provided in the DHA.

#### 12.1.3. BIIB092 Handling and Disposal

The Investigator must return all used and unused vials of BIIB092 as instructed by Biogen unless approved for onsite destruction.

If any BIIB092 supplies are to be destroyed at the study site, the institution or appropriate study site staff must obtain prior approval from Biogen, by providing, in writing, the destruction policy or details of the method of destruction. After such destruction, Biogen must be notified, in writing, of the details of the study treatment destroyed (e.g., lot or kit numbers, quantities), the date of destruction, and proof of destruction.

#### 12.1.4. BIIB092 Accountability

Accountability for study treatment is the responsibility of the Investigator. The study site must maintain accurate records demonstrating dates and amount of study treatment received, to whom dispensed (participant-by-participant accounting), and accounts of any study treatment accidentally or deliberately destroyed or lost.

Unless otherwise notified, all vials, both used and unused, must be saved for study treatment accountability. By the end of the study, reconciliation must be made between the amount of BIIB092 supplied, dispensed, and subsequently destroyed, lost, or returned to Biogen. A written explanation must be provided for any discrepancies.

#### 12.2. Placebo

The placebo (0.9% sodium chloride solution) will be provided by the study site.






# 13. EFFICACY, PHARMACOKINETIC, PHARMACODYNAMIC, IMMUNOGENICITY, AND HEALTH OUTCOMES ASSESSMENTS

See Section 5 for the timing of all assessments.

#### 13.1. Clinical Efficacy Assessments

The following clinical assessments will be performed to evaluate the efficacy of BIIB092:

- CDR (to derive the primary efficacy endpoint)
- MMSE, ISLT, DKEFS Category Fluency and Letter Fluency tests, DSST, Trails A, eCog, ADCS-ADL, FAQ, ADAS-Cog 13, and NPI-10 (to derive exploratory efficacy endpoints)

Assessments administered to the participant include the CDR, MMSE, ISLT, ISLR (Screening Visit 1 only), DKEFS Category Fluency and Letter Fluency tests, DSST, Trails A, and ADAS-Cog 13. Assessments that require caregiver/informant input include the CDR, eCog, ADCS-ADL, FAQ, and NPI-10.

The clinical assessments must be administered by a trained clinician or rater, preferably by a neuropsychologist, a psychometrician or another qualified person who is experienced in the assessment of participants with cognitive deficits.

It is recommended that postbaseline CDR assessments be conducted at the same time of day at which the baseline assessment was performed to avoid diurnal variation. The rater who conducts the CDR for a participant/informant cannot complete any other rating scales for that same participant/informant or be the study site coordinator.

The rater must be certified before any assessments may be performed. When possible, the same rater should administer a given test across all visits for a given participant. See the Study Reference Guide for specific guidelines required for administration of each test and the order in which the tests should be performed.

#### 13.2. Pharmacokinetic Assessments

BIIB092 concentrations in serum will be determined using validated assays.

Serum PK parameters of BIIB092 to be assessed may include, but will not be limited to, the following:

• Trough concentration

• End-of-infusion concentration



See Section 5 for the timing of assessments. The timing for collection of postdose serum samples will be based on the completion of the BIIB092 infusion.

#### 13.3. Pharmacodynamic Assessments

The PD properties of BIIB092 will be assessed as described below.

- Morphometric measures of certain brain areas, including volume and cortical thickness, will be assessed by MRI in all participants. Details of the MRI scanning protocol will be described in the procedural manual for MRI.
- Concentrations of disease-related biomarkers in blood, including but not limited to, tau and other markers of neurodegenerative disease will be assessed in all participants.



See Section 5 for the timing of assessments.







#### **13.6. Immunogenicity**

A validated immunoassay will be used to assay samples for the presence of, and measure titers of, anti-BIIB092 antibodies in serum. Samples will be collected on Study Day 1 and at Weeks 4,

24, 48, 76, 80, 104, 116, 156, 176, 196, 224, and 238/FUV (see Section 5). All samples will be collected predose.

#### 13.7. Health Outcomes Assessments

The following tests will be performed to assess the effects of BIIB092 on caregiver burden, participant quality of life, and resource utilization:

- ZBI
- QoL-AD
- RUD-Lite

The ZBI, QoL-AD, and RUD-Lite are administered to the caregiver; the QoL-AD is also administered to the participant. The recommended order of administration of these assessments is specified in the Study Reference Guide.

See Section 5 for the timing of assessments.

#### 14. SAFETY ASSESSMENTS

See Section 5 for the timing of all safety assessments.

# 14.1. Clinical Safety Assessments

The following clinical assessments will be performed to evaluate the safety profile of BIIB092:

- Physical examinations, including height and weight measurements.
- Neurological examinations.
- Vital sign measurements: temperature, pulse rate, SBP, DBP, and respiratory rate.
  Measurements will be recorded after the participant has been resting in a supine
  position for 10 minutes. At selected timepoints (see Table 1), blood pressure and
  pulse rate will also be recorded after the participant has been standing for
  > 2 minutes.
- 12-lead (paper) ECGs, to be performed in triplicate at each timepoint with approximately 1 minute between replicates. Each ECG must be performed after the participant has been resting in a supine position for 10 minutes. The ECGs will be read by a central reader; copies of all raw ECG data must be made available to Biogen.
- Laboratory safety assessments (see Section 14.2).
- Columbia Suicide Severity Rating Scale (C-SSRS).
- Concomitant therapy and procedure recording.
- AE and SAE monitoring.

# 14.2. Laboratory Safety Assessments

Samples will be analyzed using Good Laboratory Practice-validated assays.

The following laboratory assessments will be performed to evaluate the safety profile of BIIB092:

 Hematology: red blood cell count, platelet count, hemoglobin level, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, and total white blood cell count with absolute counts and percentages of differential cells (neutrophils, monocytes, lymphocytes, eosinophils, and basophils).

- Clinical chemistry: total protein, albumin, creatinine, BUN, uric acid, bilirubin (total
  and direct), alkaline phosphatase, ALT, AST, lactate dehydrogenase,
  gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride,
  sodium, and potassium.
- Urinalysis: color, specific gravity, pH, protein, glucose, leukocyte esterase, blood ketones (and microscopic examination, if abnormal).
- Serum and urine pregnancy tests for women of childbearing potential only.
- At the first screening visit only: testing for HIV (to be performed based upon Investigator assessment of HIV risk factors; the requirement for testing during Screening may be omitted if it is not permitted by local regulations), glycosylated hemoglobin, HBsAg, anti-HBc, and hepatitis C antibody; alcohol/drug screen; and follicle-stimulating hormone (FSH; postmenopausal women only).



# 15. SAFETY DEFINITIONS, RECORDING, REPORTING, AND RESPONSIBILITIES

Throughout the course of the study, every effort must be made to remain alert to possible AEs. If an AE occurs, the first concern should be for the safety of the participant. If necessary, appropriate medical intervention should be provided.

At the signing of the ICF, each participant or his/her legally authorized representative, in countries where applicable laws allow, and/or main caregiver must be given the names and telephone numbers of study site staff for reporting AEs and medical emergencies.

#### 15.1. Definitions

#### 15.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

Determination of whether an abnormal laboratory value, vital sign result, and/or ECG result meets the definition of an AE will be made by the Investigator. Abnormal results are not considered AEs unless one or more of the following criteria are met:

- The result meets the criteria for an SAE
- The result requires the participant to receive specific corrective therapy
- The result is considered by the Investigator to be clinically significant

#### 15.1.2. Serious Adverse Event

An SAE is any untoward medical occurrence that at any dose:

- Results in death
- In the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity


The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

- Results in a congenital anomaly/birth defect
- Is a medically important event

A medically important event is an AE that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. (Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or convulsions occurring at home that do not require an inpatient hospitalization.)

#### 15.1.3. Prescheduled or Elective Procedures or Routinely Scheduled Treatments

A prescheduled or elective procedure or a routinely scheduled treatment will not be considered an SAE, even if the participant is hospitalized. The study site must document all of the following:

- The prescheduled or elective procedure or routinely scheduled treatment was scheduled (or was on a waiting list to be scheduled) prior to obtaining the participant's consent to participate in the study.
- The condition requiring the prescheduled or elective procedure or routinely scheduled treatment was present before and did not worsen or progress in the opinion of the Investigator between the participant's consent to participate in the study and the time of the procedure or treatment.
- The prescheduled or elective procedure or routinely scheduled treatment is the sole reason for the intervention or hospital admission.
  - If a participant is hospitalized due to local requirements for administration of the study treatment, the hospitalization should not be considered an SAE unless one of the requirements in Section 15.1.2 is met.

# **15.2.** Safety Classifications

# **15.2.1.** Investigator Assessment of Events

All events must be assessed to determine the following:

- If the event meets the criteria for an SAE as defined in Section 15.1.2.
- The relationship of the event to study treatment, as defined in Section 15.2.2.
- The severity of the event as defined in Section 15.2.3.

# 15.2.2. Relationship of Events to Study Treatment,

The following definitions should be considered when evaluating the relationship of AEs and SAEs to the study treatment.





#### 15.2.3. Severity of Events

The following definitions should be considered when evaluating the severity of AEs and SAEs:

| Severity of Event | |
|---|---|
| Mild | Symptoms barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptoms but may be given because of personality of participant. |
| Moderate | Symptoms of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptoms may be needed. |
| Severe | Symptoms cause severe discomfort; symptoms cause incapacitation or significant impact on participant's daily life; severity may cause cessation of treatment with study treatment; treatment for symptoms may be given and/or participant hospitalized. |

#### 15.2.4. Expectedness of Events

Expectedness of all AEs will be determined by Biogen according to the Investigator's Brochure.

# 15.3. Monitoring and Recording Events

#### 15.3.1. Adverse Events

Any AE experienced by the participant between the time of first dose of study treatment and the participant's final clinic visit (including the Follow-up Safety Visit) is to be recorded on the CRF, regardless of the severity of the event or its relationship to study treatment,

At each study visit, the Investigator will assess the participant for AEs and will record any new AEs or updates to previously reported AEs on the CRF.



AEs that are ongoing when the participant completes or discontinues the study will be followed by the Investigator until the event has resolved, stabilized, or returned to baseline status. AE outcome will be recorded on the CRF, as applicable.

#### 15.3.2. Adverse Events of Special Interest

Immunogenicity is an AE of special interest that is under monitoring in all ongoing studies. Participants will also be monitored for possible infusion-associated AEs and/or hypersensitivity reactions during and after completion of the investigational medicinal product infusion.

#### 15.3.3. Serious Adverse Events

Any SAE experienced by the participant between the time of the signing of the ICF and the participant's final clinic visit (including the Follow-up Safety Visit) is to be recorded on an SAE form, regardless of the severity of the event or its relationship to study treatment. SAEs must be reported to Biogen within 24 hours as described in Section 15.3.4. Follow-up information regarding an SAE also must be reported within 24 hours.

Participants will be followed for all SAEs until the final clinic visit (including the Follow-up Safety Visit). Thereafter, the event should be reported to Biogen only if the Investigator considers the SAE to be related to study treatment.

Any SAEs that is ongoing when the participant completes or discontinues the study will be followed by the Investigator until the event has resolved, stabilized, or returned to baseline status.

#### 15.3.4. Immediate Reporting of Serious Adverse Events

In order to adhere to all applicable laws and regulations for reporting an SAE, the study site must formally notify Biogen within 24 hours of the study site staff becoming aware of the SAE. It is the Investigator's responsibility to ensure that the SAE reporting information and procedures are used and followed appropriately.

#### **Reporting Information for SAEs**

A report <u>must be submitted</u> to Biogen regardless of the following:

- Whether or not the participant has undergone study-related procedures
- Whether or not the participant has received study treatment
- The severity of the event
- The relationship of the event to study treatment

To report initial or follow-up information on an SAE, fax a completed SAE form; see the Study Reference Guide's Official Study Contact List for complete contact information.

#### 15.3.4.1. Deaths

Death is an outcome of an event. The event that resulted in death should be recorded on the appropriate CRF. All causes of death must be reported as SAEs within 24 hours of the study site becoming aware of the event. The Investigator should make every effort to obtain and send CONFIDENTIAL

The information contained herein may not be used, disclosed, or published without the written consent of Biogen MA Inc.

death certificates and autopsy reports to Biogen. The term death should be reported as an SAE only if the cause of death is not known and cannot be determined.

#### 15.3.5. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are SAEs that are unexpected and judged by the Investigator or Biogen to be related to the study treatment administered.

Appropriate personnel at Biogen will unblind SUSARs for the purpose of regulatory reporting. Biogen will submit SUSARs (in blinded or unblinded fashion) to regulatory agencies according to local law. Biogen will submit SUSARs to Investigators in a blinded fashion.

# 15.4. Procedures for Handling Special Situations

# 15.4.1. Pregnancy

Participants should not become pregnant during the study and for 6 months (24 weeks) after their last dose of study treatment. If a female participant becomes pregnant, study treatment must be discontinued *immediately*. It is recommended that male participants should not father children during their participation in the study and for 6 months (24 weeks) after their last dose of study treatment.

The Investigator must report a pregnancy occurring in a female participant by faxing the appropriate form to Biogen within 24 hours of the study site staff becoming aware of the pregnancy. See the Study Reference Guide's Official Study Contact List for complete contact information. The Investigator or study site staff must report the outcome of the pregnancy to Biogen. A pregnancy is not considered an AE and should not be recorded on the AE CRF.

Congenital abnormalities and birth defects in the offspring of male or female participants should be reported as an SAE if conception occurred during the study Treatment Period.

#### **15.4.2.** Overdose

An overdose is any dose of study treatment administered to a participant or taken by a participant that exceeds the dose assigned to the participant according to the protocol. Overdoses are not considered AEs and should not be recorded as an AE on the CRF; however, all overdoses must be recorded on an Overdose form and faxed to Biogen within 24 hours of the study site becoming aware of the overdose. An overdose must be reported to Biogen even if the overdose does not result in an AE. If an overdose results in an AE, the AE must be recorded. If an overdose results in an SAE, both the SAE and Overdose forms must be completed and faxed to Biogen. All study treatment related dosing information must be recorded on the dosing CRF.

#### 15.4.3. Medical Emergency

In a medical emergency requiring immediate attention, study site staff will apply appropriate medical intervention, according to current standards of care. The Investigator (or designee)

should contact Biogen 24-hour emergency medical support: 1-973-659-6677. See the Study Reference Guide's Official Study Contact List for complete contact information.

#### **15.4.3.1.** Unblinding for Medical Emergency

In a medical emergency when knowledge of the participant's treatment assignment may influence the participant's clinical care, the Investigator or appropriate designee may access the participant's treatment assignment in the IRT system by accessing the internet or using a phone-based interface. Further information about the IRT unblinding function or 24-hour, 7-day-a-week support contact information is available in the IRT manual for the study.

The Investigator must document the reasons for unblinding in the participant's source documents. The Investigator is strongly advised not to divulge the participant's treatment assignment to any individual not directly involved in managing the medical emergency, or to personnel involved with the analysis and conduct of the study.

The Investigator can contact Biogen or its designee to discuss such situations, but such a discussion should not delay management of the medical emergency. The Investigator should inform Biogen or its designee as soon as possible if unblinding occurs.

# 15.5. Contraception Requirements

All women of childbearing potential and all men must ensure that highly effective contraception is used during the study and for 6 months (24 weeks) after their last dose of study treatment. In addition, participants should not donate sperm or eggs for the duration of the study and for at least 5 times the half-life of BIIB092 or 6 months, whichever is longer, after their last dose of study treatment.

For the purposes of this study, women who do not meet one of the following criteria are considered to be physiologically capable of becoming pregnant and are, therefore, defined as women of childbearing potential:

- Postmenopausal:
  - 12 continuous months of natural (spontaneous) amenorrhea without an alternative medical cause and a serum FSH level >40 mIU/mL at Screening Visit 1.
  - 6 weeks after surgical bilateral oophorectomy with or without hysterectomy.
- Posthysterectomy.
- Female surgical sterilization (e.g., bilateral tubal ligation).

For the purposes of the study, highly effective contraception is defined as use of 2 of the following:

#### For female participants:

- Established use of oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal methods of contraception associated with the inhibition of ovulation.
- Established use of oral, injected, or implanted hormonal methods of contraception.
- Placement of an intrauterine device or intrauterine hormone-releasing system.
- Barrier methods of contraception with use of a spermicide, including condom, nonprescription sponge, or occlusive cap (diaphragm or cervical vault cap) used with spermicidal foam, gel, film, or cream suppository.
- Sex with a male who has undergone surgical sterilization (with the appropriate postvasectomy documentation of the absence of sperm in the ejaculate).

#### For male participants:

- Vasectomy with negative semen analysis at follow-up.
- Condoms with spermicide.
- Sex with a woman who uses the methods described for females if she is of childbearing potential.

For all participants, true abstinence, when this is consistent with the preferred and usual lifestyle of the participant, can be considered an acceptable method of contraception based on the evaluation of the Investigator who should also take into consideration the duration of the clinical study. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not considered acceptable methods of contraception.

Pregnancy reporting is described in Section 15.4.1.

# 15.6. Safety Responsibilities

#### 15.6.1. The Investigator

The Investigator's responsibilities include the following:

| • | Monitor and record all AEs, including SAEs, on the CRF regardless of the severity or |
|---|---|
| | relationship to study treatment, |

• Determine the seriousness, relationship to study treatment, and severity of each event.

- Determine the onset and resolution dates of each event.
- Monitor and record all pregnancies in female participants and follow up on the outcome of all pregnancies.
- Complete an SAE form for each SAE and fax or email it to Biogen within 24 hours of the study site staff becoming aware of the event.
- Pursue SAE follow-up information actively and persistently. Follow-up information
  must be reported to Biogen within 24 hours of the study site staff becoming aware of
  new information.
- Ensure all AE and SAE reports are supported by documentation in the participants' medical records.
- Pursue AE follow-up information, if possible, until the event has resolved or become stable. Record AE follow-up information, including resolution, on the CRF, as applicable.
- Report SAEs to local ethics committees, as required by local law.

# 15.6.2. Biogen

Biogen's responsibilities include the following:

- Before a study site can enroll any participants, the Clinical Monitor is responsible for reviewing with study site staff the definitions of AE and SAE, as well as the instructions for monitoring, recording, and reporting AEs and SAEs.
- Biogen is to notify all appropriate regulatory authorities, central ethics committees, and Investigators of SAEs, as required by local law, within required time frames.

# 16. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

The objectives of the study and the endpoints to be analyzed are listed in Section 6.

#### 16.1. General Considerations

Data will be collected and analyzed separately for the placebo-controlled period and LTE period:

- 1. After the placebo-controlled period is completed, efficacy and safety analyses will be performed.
- 2. Analyses will be performed as needed during the LTE period. Descriptive statistics will be used to evaluate the long-term safety and efficacy data of BIIB092.

Summary statistics will be presented. For continuous endpoints, summary statistics will generally include: number of participants with data, mean, SD, median, and range. For categorical endpoints, this will generally include: number of participants randomized or dosed, number of participants with data, and the percentage of those with data in each category. Data for participants who were randomized to BIIB092 low dose (125 mg once every 4 weeks or 375 mg once every 12 weeks) will be pooled for statistical testing and modeling for efficacy, PD, and health outcome analyses, unless otherwise specified in the placebo-controlled period. All statistical tests will be 2-sided.

Similar analyses will be applied to both the placebo-controlled and LTE periods, except for efficacy analyses, which will be detailed in the statistical analysis plan (SAP).

# 16.2. Demography and Baseline Disease Characteristics

Demographics and baseline data will be summarized by treatment group with summary statistics or with frequency distributions.

# **16.3. Safety**

# 16.3.1. Analysis Population

The population for safety analyses is defined as all participants who were randomized and who received at least 1 dose of study treatment.

#### 16.3.2. Methods of Analysis

#### 16.3.2.1. Adverse Events

All analyses of AEs will be based on the principle of treatment emergence. An AE is considered to be treatment emergent if it has an onset date on or after the date of first dosing, or if it was


present prior to the first dose and subsequently worsened. The incidence of all AEs will be presented by system organ class and preferred term by dose group and for the overall active treatment group. In addition, the incidence of all AEs will be presented by severity, by relationship to study treatment,

#### 16.3.2.2. Clinical Laboratory Results

Clinical laboratory evaluations include hematology, blood chemistry, and urinalysis evaluations. Analyses of clinically significant abnormalities, shifts from baseline to postbaseline relative to the normal range, as well as changes from baseline by visit, will be presented by dose group and for the overall active treatment group.

## **16.3.2.3.** Vital Signs

The analysis of vital signs will focus on clinically relevant abnormalities, which will be defined in more detail in the SAP. The incidence of clinically relevant abnormalities in vital signs will be summarized by dose group and for the overall active treatment group.

#### 16.3.2.4. Electrocardiograms

The analysis of ECG data will focus on clinically relevant abnormalities, which will be defined in more detail in the SAP. ECG changes from baseline may be summarized using descriptive statistics and presented by dose group, overall active treatment group, and visit.

# 16.3.2.5. Physical and Neurological Examinations

Abnormal findings during physical and neurological examinations will be recorded as AEs and will be reflected in the summary of AEs.

#### 16.3.2.6. Columbia - Suicide Severity Rating Scale

C-SSRS data will be summarized using descriptive statistics and presented by dose group and for the overall active treatment group.

# 16.4. Efficacy

#### 16.4.1. Analysis Population

Efficacy analyses will use the intent-to-treat (ITT) population, defined as all participants who were randomized and who received at least 1 dose of study treatment. For each endpoint, additional conditions may apply to the definition of the population for the analysis. Participants will be analyzed in the groups to which they were randomized. Subgroup analysis may be done for selected endpoints (e.g., CDR-SB).

#### 16.4.2. Methods of Analysis

# 16.4.2.1. Analysis of Primary Efficacy Endpoint (Clinical Dementia Rating Scale – Sum of Boxes)

The CDR-SB is the primary efficacy endpoint. The population for the analysis of CDR-SB will be participants in the ITT population who have a baseline and at least 1 postbaseline CDR-SB score.

A mixed model with repeated measures (MMRM) will be used to analyze changes from Baseline in CDR-SB using fixed effects of treatment, time, treatment-by-time interaction, baseline CDR-SB, baseline CDR-SB-by-time interaction, region, disease stage (MCI versus mild AD), and baseline AD medication use. The correlation between repeated measures of the outcomes will be taken into consideration. The least-squares (LS) means, the differences in LS means between each treatment group versus placebo at Weeks 24, 52, and 78, 95% confidence intervals (CIs), and p-values will be presented. Changes from baseline in CDR subscores will be analyzed in a similar model. Additional details will be provided in the SAP.

The multiple comparison procedure modelling (MCP-MOD) method will be used to assess and model dose-response relationships (potential candidate models will include linear, linear-log, quadratic, maximum response [ $E_{max}$ ], and logistic models as specified in Section 16.10) while controlling for multiplicity. The dose-response parameter of interest for MCP-MOD will be the LS means at Week 78 for each dose group from the mixed-effects model. Pairwise comparisons of each BIIB092 dose group versus placebo will also be conducted.

#### 16.4.2.2. Analysis of Exploratory Clinical Endpoints

The clinical endpoints assessing AD progression from Baseline include the results of the MMSE, ISLT, DKEFS, DSST, Trails A, eCog, ADCS-ADL, FAQ, ADAS-Cog 13, and NPI-10.

These clinical endpoints will be analyzed using data from participants in the ITT population who have a baseline and at least 1 postbaseline score for the specific endpoint being analyzed. As these are exploratory endpoints in this study, no additional multiplicity adjustment procedures will be applied to the analyses of these endpoints.

An MMRM approach will be used to analyze changes from baseline using fixed effects of treatment, time, treatment-by-time interaction, baseline score, baseline score-by-time interaction, region, disease stage (MCI versus mild AD), and baseline AD medication use. The correlation between repeated measures of the outcomes will be taken into consideration. The LS means, the differences in LS means between each treatment group versus placebo at Weeks 24, 52, and 78, and the 95% CIs and p-values will be presented.

Exploratory analysis may be performed to develop a composite cognitive score participants with MCI due to AD and/or participants with mild AD.

#### 16.4.3. Analysis for the Long-Term Extension Period

The analysis will include all participants who received at least 1 dose of study treatment in the LTE period.

The endpoints for the LTE period are change from baseline over the placebo-controlled and LTE periods of the study. Analyses will be presented by treatment group in the LTE period using the placebo-controlled period baseline. Details of the analyses will be prespecified in the SAP.

#### 16.5. Pharmacokinetics

#### 16.5.1. Analysis Population

The population for serum PK analyses is defined as all participants in the ITT population who have at least 1 measurable postbaseline BIIB092 concentration in serum.

Participants who receive BIIB092 125 mg once every 4 weeks will be analyzed separately from those who receive 375 mg once every 12 weeks.

#### 16.5.2. Methods of Analysis

Samples for measuring serum concentrations of BIIB092 will be collected as specified in Section 5. BIIB092 concentrations in serum will be summarized using descriptive statistics for the first 20 participants in the PK/PD analysis at Week 12 and at the end of the study, by dose group.

This study will collect only sparse PK samples, thus the serum concentration data will be summarized descriptively by visit and dose group. No noncompartmental or compartmental methods will be used to analyze the PK data for presentation in the clinical study report. Details of the PK analysis will be described in the SAP.

Mean serum concentrations of BIIB092 will be plotted versus time by dose group on both a linear and a logarithmic scale. No dose proportionality assessments will be conducted due to the sparse PK data sampling.

Atypical drug concentrations (e.g., very low or very high) will be excluded from the analysis, if no apparent explanation exists. Concentration observations will also be removed from the data set if corresponding dosing or sampling times are missing or cannot be reconstructed. Concentration values below the limit of quantification will be appropriately handled per the SAP. All deletions of data points will be appropriately documented.

Population PK analysis may be conducted to estimate BIIB092 population PK parameters and to identify potential covariates (e.g., demographics, body weight, and anti-BIIB092 antibodies) on the variability of BIIB092 PK. Results will be presented in a separate report.

# 16.6. Pharmacodynamics

#### 16.6.1. Analysis Population

The PD analysis population is defined as all participants who in the ITT population who have at least 1 post baseline assessment of the specific parameter being analyzed.



## 16.6.3. Methods of Analysis for Other Pharmacodynamic Parameters

MRI scans and blood samples will be collected as specified in Section 5. MRI results analyzed may include, but will not be limited to, MRI morphometric measures including volume and cortical thickness of certain brain areas.

Data for these exploratory potential biomarker candidates related to BIIB092 biological activity or disease progression will be summarized using descriptive statistics and will be presented by dose group.

# 16.7. Health Outcomes

#### 16.7.1. Analysis Population

The ITT population will be used for the analysis of health outcomes data.

#### 16.7.2. Methods of Analysis

The scores for and changes from baseline in the ZBI and QoL-AD, and cumulative resource utilization collected from the RUD-Lite assessments up to Week 72, will be summarized by treatment group.

# 16.8. Immunogenicity

#### 16.8.1. Analysis Population

The population for analyses of anti-BIIB092 antibodies is defined as all participants who were randomized and received at least 1 dose of study treatment and who have at least 1 postdose serum sample evaluated for anti-BIIB092 antibodies.

#### 16.8.2. Methods of Analysis

The incidence of anti-BIIB092 antibodies will be summarized by treatment group over time.

# 16.9. Interim Analyses

Interim analyses may be performed after 50% to 100% of participants have completed the Week 52 visit (or discontinued) for the purpose of future study planning and/or futility analyses. In order to maintain the treatment blind, an independent group external to Biogen that will not be involved in the conduct of the study after unblinding will perform the interim analyses. This independent group will present the unblinded interim analyses to the DMC for review. After the DMC review, a small internal independent team (separate from the study team) may review the unblinded results for the purpose of future study planning under a study integrity charter. No Type I error adjustment will be made. No changes will be made to this study based on the interim analysis results.

After all participants have completed the placebo-controlled period, the Sponsor may perform an unblinded analysis. The Sponsor may perform additional interim analyses thereafter.

# **16.10.** Sample Size Considerations

There was no formal sample size calculation for the primary endpoint of safety.

The planned sample size is 528 participants, randomized in a 1:1:2:2 ratio, with 88 participants assigned to the BIIB092 low-dose group (44 assigned to 125 mg once every 4 weeks and 44 assigned to 375 mg once every 12 weeks), 88 participants assigned to the medium-dose group (600 mg once every 4 weeks), 176 participants assigned to the high-dose group (2000 mg once every 4 weeks), and 176 participants assigned to the placebo group. This sample size provides approximately 80% power to detect a dose-response relationship in the change from baseline in CDR-SB (primary efficacy endpoint) at 18 months (Week 78), assuming a mean change of 1.99 from baseline in CDR-SB at 18 months in the placebo group and a common SD of 2.38, a maximal 40% reduction for the highest BIIB092 dose group compared with the placebo group, and an estimated 20% dropout rate at 18 months (Week 78) in this study. Six different dose-response relationships will be tested at the 2-sided 5% significance level, using the MCP-MOD method to control for multiplicity [Bretz 2005]. Optimal contrasts will be constructed to detect potential dose-response trends under common dose-response curves (e.g., Emax, exponential, logistic, linear in log dose, and quadratic model) which are illustrated with the parameters shown in Figure 2.

The mean and SD of the change from baseline in CDR-SB at 18 months for the placebo group is based on available Alzheimer's Disease Neuroimaging Initiative (ADNI) data from ADNI 1, ADNI 2, and



Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

In the LTE period, the actual sample size, enterprise period, is dependent on the enrollment rate, and thus, sample size calculation is not needed.

Figure 2: Dose-Response Shapes Based on Clinical Dementia Rating Scale – Sum of Boxes Mean Change from Baseline at Week 78



 $ED_{50}$  = median effective dose; Emax = maximum response

Note: This figure was generated using ADDPLAN® DF Version 3.1.8, by Aptiv solutions.

#### 17. ETHICAL REQUIREMENTS

Biogen, a CRO, and the Investigator must comply with all instructions, regulations, and agreements in this protocol and applicable International Council for Harmonisation (ICH) and Good Clinical Practice (GCP) guidelines and conduct the study according to local regulations.

The Investigator is responsible for endorsing all data on completed CRFs electronically, prior to any Interim lock or Database lock.

The Investigator may delegate responsibilities for study-related tasks where appropriate to individuals sufficiently qualified by education, training, and experience, in accordance with applicable ICH and GCP guidelines. The Investigator should maintain a list of the appropriately qualified persons to whom significant study-related duties have been delegated. The Investigator is responsible for supervising those individuals and for implementing procedures to ensure the integrity of the tasks performed and any data generated.

#### 17.1. Declaration of Helsinki

This study will be performed in alignment with the ethical principles outlined in the Declaration of Helsinki.

#### 17.2. Ethics Committee

The Investigator must obtain ethics committee approval of the protocol, ICF, and other required study documents prior to starting the study. Biogen will submit documents on behalf of the study sites worldwide in compliance with local regulations.

If the Investigator makes any changes to the ICF, Biogen must approve the changes before the ICF is submitted to the ethics committee. A copy of the approved ICF must be provided to Biogen. After approval, the ICF must not be altered without the agreement of the relevant ethics committee and Biogen.

It is the responsibility of the Investigators to ensure that all aspects of institutional review are conducted in accordance with current applicable regulations.

Biogen must receive a letter documenting ethics committee approval, which specifically identifies the protocol, protocol number, and ICF, prior to the initiation of the study. Protocol amendments will be participant to the same requirements as the original protocol.

A progress report must be submitted to the ethics committee at required intervals and not less than annually.

At the completion or termination of the study, the study site must submit a close-out letter to the ethics committee and Biogen.


# 17.3. Participant Information and Consent

Prior to performing any study-related activities under this protocol, including screening tests and assessments, written informed consent with the approved ICF must be obtained from the participant or participant's legally authorized representative (e.g., legal guardian), as applicable, in accordance with local practice and regulations.

During the first screening visit, under a separate (optional) initial consent process, participants can complete the cognitive scales. If the participant meets inclusion criteria for the CDR, MMSE, and ISLT/ISLR, then the full consent process must be completed prior to the administration of further screening assessments. Participants may also proceed directly to the full consent process, which would allow the administration of all screening assessments. See Section 9.1 for details of the screening process.

The background of the proposed study, the procedures (including ApoE testing), the benefits and risks of the study, and that study participation is voluntary for the participant must be explained to the participant (or the participant's legally authorized representative, in countries where applicable laws allow). The participant must be given sufficient time to consider whether to participate in the study.

Participants will be informed that their race and ethnicity will be collected during the study (unless the collection is not permitted by applicable law or not approved by the governing ethics committee) and the data will be used during analysis of study results.

Participants will also be informed that audio recordings may be made of some clinical assessments in order to allow for central review for standardization of test administration, where allowable by country and/or local authorities.



Participants or their legally authorized representatives, in countries where applicable laws allows, who chose to participate in the LTE period must provide informed consent before any LTE period screening tests are performed.

participant's informant/study partner must also provide consent.

Copies of the participant's signed and dated ICF(s) (optional initial consent, if applicable, and full consent) and a copy of the signed and dated optional genetic sampling consent form, if applicable, must be given to the participant or the participant's legally authorized representative, in countries where applicable laws allow. The original signed and dated ICFs will be retained with the study records. Local regulations must be complied with in respect to the final disposition of the original (wet signature) and copies of the signed and dated ICFs.

Confirmation of informed consent must also be documented in the participant's medical record.

The participant's study partner/informant must also provide written informed consent to participate in the study and be reconsented to participate in the LTE period. The original forms will be managed and archived in the same manner as the participants' ICFs, as described above.

Participants or their informant/study partner can withdraw consent to participate in the study at any time.

# 17.4. Participant Data Protection

Prior to any testing under this protocol, including screening tests and assessments, candidates must also provide all authorizations required by local law (e.g., Protected Health Information authorization in North America).

During Screening, participants' race and ethnicity will be collected (unless the collection is not permitted by applicable law or not approved by the governing ethics committee). Race and ethnicity data will be used to describe the demographic profile of the study population and to evaluate the balance of demographic characteristics across the randomized treatment groups. These data may also be used in the analysis of the safety and/or PK profile of the study treatment. It is unknown whether the effects of the study treatment are influenced by race or ethnicity.

Audio recordings may be made of some clinical assessments in order to allow for central review for standardization of test administration, where allowable by country and/or local authorities.

Study reports will be used for research purposes only. The participant will not be identified by name in CRFs, study-related forms, study reports, or any related publications. Biogen, its partners and designees, ethics committees, and various government health agencies may inspect the records of this study. Every effort will be made to keep the participant's personal medical data confidential.

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

# 17.5. Compensation for Injury

Biogen maintains appropriate insurance coverage for clinical studies and will follow applicable local compensation laws.

#### 17.6. Conflict of Interest

The Investigators should address any potential conflicts of interest (e.g., financial interest in Biogen) with the participant before the participant makes a decision to participate in the study.

# 17.7. Registration of Study and Disclosure of Study Results

Biogen will register the study and post study results regardless of outcome on a publicly accessible website in accordance with the applicable laws and regulations.
# 18. ADMINISTRATIVE PROCEDURES

# **18.1.** Study Site Initiation

The Investigator must not screen any participants prior to completion of a study initiation visit, conducted by Biogen. This initiation visit will include a detailed review of the protocol and study procedures.

# 18.2. Quality Control and Quality Assurance

Quality control procedures will be implemented at each stage of data handling to ensure that all data are reliable and have been processed correctly. Data anomalies will be communicated to the study sites for clarification and resolution, as appropriate. The Investigator is responsible for endorsing all CRF data prior to any interim or final database lock.

During and/or after completion of the study, quality assurance officers named by Biogen or the regulatory authorities may wish to perform onsite audits or inspections. The Investigator will be expected to cooperate with any audit or inspection and to provide assistance and documentation (including source data) as requested.

# 18.3. Monitoring of the Study

The Investigator must permit study-related monitoring by providing direct access to source data and to the participants' medical histories. Source data must be attributable, legible, contemporaneous, original, accurate, and complete. Changes to source data must be traceable, not obscure the original entry, and be explained if necessary (e.g., with an audit trail). The Investigator should maintain a record of the location(s) of essential documents.

The Clinical Monitors will visit the study sites at regular intervals during the study and after the study has completed, as appropriate. A clinical site monitoring plan will detail who performs the monitoring, how often, and the extent of review. It also will provide the monitoring strategy, with emphasis on participant safety, data integrity, and critical data and processes.

During these visits, CRFs, supporting documentation, and essential documentation related to the study will be reviewed and any discrepancies or omissions will be resolved.

Monitoring visits must be conducted according to the applicable ICH and GCP guidelines to ensure the protection of participant rights and well-being, protocol adherence, quality of data (accurate, complete, and verifiable), study treatment accountability, compliance with regulatory requirements, and continued adequacy of the study site and its facilities.

Phase 2 Study of BIIB092 in Mild Cognitive Impairment due to Alzheimer's Disease and Mild Alzheimer's Disease

# 18.4. Study Funding

Biogen is the Sponsor of the study and is funding the study. All financial details are provided in the separate contracts between the institution, Investigator, and Biogen.

# 18.5. Publications

Details are included in the clinical trial agreement for this study.

Version 4

# 19. FURTHER REQUIREMENTS AND GENERAL INFORMATION

# 19.1. External Contract Organizations

# 19.1.1. Contract Research Organization

A CRO will be responsible for administrative aspects of the study including but not limited to study initiation, monitoring, and data management. Before participants are screened at each study site, the CRO will review study responsibilities with the Investigators and other study site staff, as appropriate.

# 19.1.2. Interactive Response Technology

IRT will be used in this study. Before participants are screened or enrolled, the IRT vendor will provide each study site with the necessary training, a user manual, and access rights to the system.

### 19.1.3. Electronic Data Capture

Participant information will be captured and managed by study sites in source documents with study data variables entered in electronic CRFs by a web-based electronic data capture tool developed and supported by Medidata Rave and configured by a CRO.

All clinician-reported and caregiver-reported outcomes will be captured in an electronic format and managed by Cogstate.

### 19.1.4. Central Laboratories for Laboratory Assessments

A central laboratory has been selected by Biogen to analyze all standard hematology, blood chemistry, and urinalysis samples collected for this study.

The central laboratory will also receive, track and ship all blood samples for specialized , and anti-drug antibody testing

Laboratories performing specialized testing will be identified in regulatory documentation. These laboratories will use appropriately validated or qualified assays to test study samples.

#### 19.1.5. Central Facility for Other Assessments

All ECGs will be read and interpreted by a central reading facility selected by Biogen. Readings from this central facility will prevail over those conducted by the Investigator.



### 19.1.6. Neurocognitive Assessments

Biogen has selected a rater management group to establish rater qualification, study-specific training, and oversight. The study raters are required to complete qualifications steps and required training prior to administering study assessments. The rater management group will oversee the assessments per project-specific plans.

# 19.2. Study Committees

An independent DMC will be established to review safety data on an ongoing basis to ensure safe and proper treatment of participants. The DMC, based on the nature, frequency, and/or severity of an AE(s), may recommend that the study continue without modification or may recommend protocol modification(s), dose suspension, or dose termination.

The DMC charter will provide full guidance on the function and practices to be followed by the DMC.

# 19.3. Changes to Final Study Protocol

All protocol amendments must be submitted to the ethics committee and regulatory authorities if required by local law. Protocol modifications that affect participant safety, the scope of the investigation, or the scientific quality of the study must be approved by the ethics committee before implementation of such modifications to the conduct of the study. If required by local law, such modifications must also be approved by the appropriate regulatory agency prior to implementation.

However, Biogen may, at any time, amend this protocol to eliminate an apparent immediate hazard to a participant. In this case, the appropriate regulatory authorities will be notified subsequent to the modification.

In the event of a protocol modification, the ICF may require similar modifications (see Section 17).

# 19.4. Ethics Committee Notification of Study Completion or Termination

Where required, the regulatory authorities and ethics committees must be notified of completion or termination of this study, and sent a copy of the study synopsis in accordance with necessary timelines.

# 19.5. Retention of Study Data

The minimum retention time for study records will meet the strictest standard applicable to that study site, as dictated by any institutional requirements or local, national, or regional laws or regulations. Prior to proceeding with destruction of records, the Investigator must notify Biogen in writing and receive written authorization from Biogen to destroy study records. In addition, the Investigator must notify Biogen of any changes in the archival arrangements including but not limited to archival at an offsite facility or transfer of ownership if the Investigator leaves the study site.

# 19.6. Study Report Signatory

Biogen will designate 1 of the participating Investigators as a signatory for the study report. This determination will be made by several factors, including, but not limited to, the Investigator's experience and reputation in the studied indication, the Investigator's contribution to the study in terms of design, management, and/or participant enrollment, or by other factors determined to be relevant by Biogen. Biogen will follow all applicable local regulations pertaining to study report signatories.

### 20. REFERENCES

Alzheimer's Association. 2015 Alzheimer's Disease Facts and Figures. Alzheimers Dement. 2015;11(3):332+.

Alzheimer's Disease International. World Alzheimer Report 2015: The Global Impact of Dementia. London: Alzheimer's Disease International (ADI); 2015.

Birks J. Cholinesterase inhibitors for Alzheimer's disease. Cochrane Database Syst Rev. 2006(1):CD005593.

Bretz F, Pinheiro JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies. Biometrics. 2005;61(3):738-48.

Hardy J, Selkoe DJ. The amyloid hypothesis of Alzheimer's disease: progress and problems on the road to therapeutics. Science. 2002;297(5580):353-6. Epub 2002 Jul 20.



McKhann GM, Knopman DS, Chertkow H, et al. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011;7(3):263-9.

McShane R, Areosa Sastre A, Minakaran N. Memantine for dementia. Cochrane Database Syst Rev. 2006(2):1-80.



Musiek ES, Holtzman DM. Three dimensions of the amyloid hypothesis: time, space and 'wingmen'. Nat Neurosci. 2015;18(6):800-6.

Serrano-Pozo A, Frosch MP, Masliah E, et al. Neuropathological alterations in Alzheimer disease. Cold Spring Harb Perspect Med. 2011;1(1):a006189.

Wahlund LO, Barkhof F, Fazekas F, et al. A new rating scale for age-related white matter changes applicable to MRI and CT. Stroke. 2001;32(6):1318-22.


# 21. SIGNED AGREEMENT OF THE STUDY PROTOCOL

I have read the foregoing protocol, "Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with Mild Alzheimer's Disease," and agree to conduct the study according to the protocol and the applicable ICH guidelines and GCP regulations, and to inform all who assist me in the conduct of this study of their responsibilities and obligations.

| Investigator's Signature | Date |
|-----------------------------|------|
| Investigator's Name (Print) | |
| investigator s rume (r mit) | |
| Study Site (Print) | |



Biogen MA Inc. 225 Binney Street Cambridge, MA 02142 United States

Biogen Idec Research Limited Innovation House 70 Norden Road Maidenhead Berkshire SL6 4AY United Kingdom

# **AMENDMENT SUMMARY**

Biogen Protocol 251AD201

Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with Mild Alzheimer's Disease

Version 2

Date: 07 September 2018

EUDRA CT Number: 2017-002901-37

Version 2.0 of the protocol has been prepared for this amendment, which supersedes Version 1.

### PRIMARY REASON FOR AMENDMENT

The primary reason for this amendment to Protocol 251AD201 is to update the list of allowed concomitant medications for subjects enrolled in this study, washout period of Alzheimer's disease (AD) medications, and to add the requirement for stable doses of key concomitant medications prior to and during Screening and for the duration of the study.

New text is shown in **bold** type; deleted text is shown with a strikethrough.

### Section 8.2, Exclusion Criteria

#### Now reads:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at Screening, or at the timepoint specified in the individual criterion listed:

. . . .

- 24.26 Use of allowed medications for chronic conditions at doses that have not been stable for at least 4 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1.5
- 27. or useUse of AD medications (including but not limited to donepezil, rivastigmine, galantamine, tacrine, and memantine) at doses that have not been stable for at least 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1.
- 25.28. Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the subject at higher risk for AEs, or impair the subject's ability to perform cognitive testing or complete study procedures. Such medications include, but are not limited to, the following:

# 29. Use of the following medications:

- Long-acting benzodiazepines (e.g., valium), except for sedation prior to MRI scans for those subjects requiring sedation and should not be administered within 24 hours prior to cognitive testing.
- Short/medium-acting benzodiazepines (e.g., alprazolam, lorazepam, oxazepam, temazepam) except if used on an as needed basischronically for sleep and on a stable dose for 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1, or used short term on an as-needed basis. May not be taken within 12 hours prior to cognitive testing.

- Short/medium acting benzodiazepines (e.g., alprazolam, lorazepam, oxazepam, temazepam) Sedating antihistamines if taken within 12 hours prior to cognitive testing. Nonsedating antihistamines (e.g., fexofenadine, cetirizine) are allowed.
- Sedating antihistamines if used on a regular basis or if taken more than 3 times per week or if taken within 24 hours prior to cognitive testing. Nonsedating antihistamines (e.g., fexofenadine, cetirizine) are allowed.
- Anticonvulsants used for treatment of seizures and anticonvulsants that have significant effects on cognition per the Investigator's opinion and/or anticonvulsants used for treatment of seizures. Anticonvulsants with limited cognitive effects, such as lamotrigine, pregabalin, levetiracetam for treatment of pain, and other non-epilepsy indications are allowed if, in the opinion of the Investigator, they are not producing sedation or contributing to cognitive impairment. The subject must have been on a stable dose for 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1.
- Sedating antidepressants Antidepressants that may, in the Investigator's opinion, affect the subject's cognition (e.g., tricyclic antidepressants). Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. Use of nonsedating antidepressants is allowed if at stable doses for 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1.
- Antipsychotics used on a regular basis. Low, except for low doses of atypical antipsychotics (e.g., risperidone, aripiprazole, or quetiapine) are allowed if used on an as-needed basis or if used at a stable dose for 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1. The definition of "low doses" should be judged by the Investigator, and the Medical Monitor can be consulted if needed

. . .

- 27.31. Prior participation in any active or passive immunotherapy study targeting A $\beta$  or tau, unless documentation of receipt of placebo is available.
- 32. Last administration of  $\beta$ -secretase inhibitors and  $\gamma$ -secretase inhibitors in a study within 3 months or 5 half-lives (whichever is longer) prior to Screening Visit 1unless documentation of receipt of placebo is available.
- 33. Participation in any study involving an investigational treatment targeting tau, unless documentation of receipt of placebo is available.

28.34. Participation within the 12 months prior to Screening Visit 1 in a study of any **other** agent(s) with a purported disease-modifying effect in AD (e.g., β secretase inhibitors, γ secretase inhibitors), unless documentation of receipt of placebo is available.



**Rationale:** Overall, the eligibility criteria regarding medications was updated to better reflect the target population and to extend the requirement for stable doses through Study Day 1. Subjects are expected to continue on the stable doses of concomitant medications throughout the study treatment period.

The modifications in use of benzodiazepines, antihistamines, anticonvulsants, antidepressants, and antipsychotics while on study are not expected to represent any changes in the safety risk for subjects with AD participating in this study.

Benzodiazepines, antihistamines, anticonvulsants, antidepressants, and antipsychotics as well as medications with platelet anti-aggregant or anticoagulant properties are widely used to manage symptoms in the target patient population.

The restrictions in use of psychoactive medications that are currently included together with the Investigator's assessment and avoidance of concomitant medications that may contribute to cognitive impairment and interfere with cognitive assessments are expected to limit variability of data.



The 12-month washout period was changed to a 3 month or 5 half-lives (whichever is longer) washout period from the last administration for  $\beta$ -secretase inhibitors and  $\gamma$ -secretase inhibitors. Based on the current knowledge, these agents are not expected to represent any change to the safety risk or confounding residual efficacy for the subjects participating in this study after this period.

This change also affects Section 11.4.1.1, Allowed Concomitant Therapy, and Section 11.4.1.2, Disallowed Concomitant Therapy.

### SUMMARY OF MAJOR CHANGES TO THE PROTOCOL

Changes to the protocol are presented chronologically. New text is shown in **bold** type; deleted text is shown with a strikethrough.

# Section 3, Synopsis

The Synopsis was revised to reflect changes made throughout the protocol.

# Section 4.5, Overall Benefits and Risks Assessment

Change: Text was added regarding the benefits and risks to subjects participating in this clinical study.

Now reads:

### 4.5 Overall Benefits and Risks Assessment

Due to its eTau-lowering effects, BIIB092 has the therapeutic potential to prevent transmission of tau pathology in neurodegenerative disorders known as tauopathies, which include PSP and AD. The proposed indications under the current program of research are for use in patients with PSP and AD.

To date, 2 clinical studies have been completed with BIIB092. These include the first-in-human study, CN002001 (SAD study in healthy adult subjects) and CN002003 (MAD study in subjects with PSP). In addition to this study, 2 studies are ongoing: Study 251PP201 (formerly referred to as CN002004), an open-label extension study, and Study 251PP301 (formerly referred to as CN002012), a Phase 2b randomized controlled efficacy and safety study in subjects with PSP. Please refer to Section 4.3.2 for more information.

All available clinical benefit and risk information to date has been derived from studies in healthy volunteers or subjects with PSP. PSP is a rare neurodegenerative disease that results in a rapidly progressing, fatal movement disorder that includes cognitive and behavioral abnormalities. There are currently no approved or effective treatments for PSP. Nonclinical models support the anti-eTau mechanism as potentially efficacious in the treatment of PSP.

Binding to eTau, the murine antibody from which BIIB092 is derived, prevented tau transmission in nonclinical studies. Furthermore, the murine antibody from which BIIB092 was derived prevented tau-dependent behavioral and pathologic changes in a mouse model of tauopathy. Finally, BIIB092 reduced free eTau levels in the CSF of cynomolgus monkeys following a single IV administration. For additional details, please refer to Section 4.3.1. By binding eTau, it is expected that BIIB092 will prevent tau

transmission in diseases such as AD and PSP and thereby potentially provide therapeutic benefit.

The nonclinical toxicity profile of BIIB092 was used to determine the starting dose and eligibility criteria and to develop appropriate safety monitoring for BIIB092 studies. Clinical data from the completed first-in-human SAD study in healthy adult subjects (CN002001) demonstrated that single doses of BIIB092 up to 4200 mg in Caucasian subjects and up to 2100 mg in Japanese subjects were generally safe and well tolerated. The completed (MAD) study in subjects with PSP (CN002003) evaluated multiple doses of BIIB092 (150, 700, and 2100 mg) or placebo administered once every 4 weeks for 3 months. The available data suggest that multiple doses of BIIB092 up to 2100 mg are safe and well tolerated in subjects with PSP. Correspondingly, the current ongoing open-label, long-term extension, safety and tolerability study (251PP201) also suggests that multiple doses of BIIB092 up to 2100 mg are safe and well tolerated in subjects with PSP.

Frequent safety assessments will be utilized by the Sponsor/Medical Monitor and Investigators to determine whether dose modification, additional safety measures, or termination of the ongoing studies is required at any time. Serum immunogenicity sampling will be performed to monitor for the emergence of anti-drug antibodies. Thorough evaluation of safety monitoring procedures and of AEs and serious adverse events (SAEs) will be reviewed on an ongoing basis by the Sponsor's Medical Monitor and Global Pharmacovigilance representatives to monitor for any safety signals or trends.

In addition, an independent Data Monitoring Committee (DMC) will also be established for Studies 251PP201 and 251PP301 to monitor the benefit/risk profile of BIIB092.

For information on specific risk mitigation strategies, please refer to Section 10, Section 11.2.2, and Section 15.4.

A need exists for disease-modifying therapies for subjects with AD and those with PSP. The doses of BIIB092 currently being explored have the potential to benefit study subjects. Furthermore, the nonclinical efficacy profile and the evidence for anti-eTau activity, together with the benign safety profile, indicate that the balance of benefit to risk is likely to be favorable for study subjects.

**Rationale:** The additions to text on the topic of the benefits and risks to subjects participating in this clinical study have been extracted from the Investigational Medicinal Product Dossiers (IMPD) and added to the protocol at the request of the Swedish Medical Products Agency and now been have added it to global protocol.

### Section 5, Schedule of Activities

### Change:

The screening period window was increased up to 90 days with Sponsor approval.

The list of assessments to be performed, in case the screening period was increased up to 90 days, was modified.

The timing of clinical assessments at Visit S3 was updated.

The timing window for coagulation tests after randomization was updated.

The timing window for the electrocardiogram (ECG) performed after the end of infusion on Study Day 1 was updated.

The fasting requirement for subjects before blood samples for hematology, clinical chemistry and urinalysis laboratory assessments was removed.

The timing of the postbaseline Clinical Dementia Rating Scale (CDR) assessment was updated.

The timing of the Alzheimer's Disease Assessment Scale-Cognitive (13 item) [ADAS-Cog 13] and Columbia - Suicide Severity Rating Scale (C-SSRS) assessments during the screening period was updated.

The reporting of serious AEs and concomitant medication was updated.

# Now reads:

**Table 1:** Schedule of Activities

| Study Week | Baseline Screening | | | | | | | | | | Place | ebo-con | trolled | Period <sup>4,</sup> | 5,6 | | | | | | | | | FU <sup>7</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Period <sup>1,2</sup> within 65 days <sup>3</sup> of Day 1 | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>8</sup> | 90 |
| Study Day | S1 | S2 | S39 | 1 | 29<br>±7 | 57<br>±7 | 85<br>±7 | 113<br>±7 | 141<br>±7 | 169<br>±7 | 197<br>±7 | 225<br>±7 | 253<br>±7 | 281<br>±7 | 309<br>±7 | 337<br>±7 | 365<br>±7 | 393<br>±7 | 421<br>±7 | 449<br>±7 | 477<br>±7 | 505<br>±7 | 533<br>±7 | 547<br>±7 | 631<br>±7 |
| Study day infusion | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Initial screening consent (optional) 10 | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Full informed consent <sup>11</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Randomization | | | | X | | | | | | | | | | | | | | | | | | | | | |
| Eligibility criteria | X | X | X | X | | | | | | | | | | | | | | | | | | | | | |
| NIA-AA criteria review | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history | X | X | X | X | | | | | | | | | | | | | | | | | | | | | |
| Body weight | X | | | X | X | X | X | | | X | | | | X | | | X | | | X | | | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test <sup>12</sup> | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Follicle-stimulating hormone <sup>13</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Alcohol/drug screen | X | | | | | | | | | | | | | | | | | | | | | | | | |
| HbA <sub>1c</sub> | X | | | | | | | | | | | | | | | | | | | | | | | | |
| HIV <sup>14</sup> /<br>hepatitis tests | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Physical examination | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | X |
| Neurological examination | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | X |

# CONFIDENTIAL

| Study Week | Bas | Baseline Screening Period <sup>1,2</sup> within 65 days <sup>3</sup> of Day 1 | | | | | | | | | | Place | ebo-con | Placebo-controlled Period <sup>4,5,6</sup> | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | wi | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>8</sup> | 90 |
| Study Day | S1 | S2 | S3 <sup>9</sup> | 1 | 29<br>±7 | 57<br>±7 | 85<br>±7 | 113<br>±7 | 141<br>±7 | 169<br>±7 | 197<br>±7 | 225<br>±7 | 253<br>±7 | 281<br>±7 | 309<br>±7 | 337<br>±7 | 365<br>±7 | 393<br>±7 | 421<br>±7 | 449<br>±7 | 477<br>±7 | 505<br>±7 | 533<br>±7 | 547<br>±7 | 631<br>±7 |
| 12-lead paper ECG <sup>16</sup> | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | X |
| Vital signs <sup>17</sup> | X | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology/ clinical chemistry/ urinalysis <sup>-8</sup> | X | | | X | | | X | | | X | | | | | | X | | | | | | X | | X | X |
| Blood sample for anti-<br>BIIB092 Ab <sup>4</sup> | | | | X | X | | | | | X | | | | | | X | | | | | | | X | | X |
| Blood sample for<br>BIIB092 concentration | | | | X | X <sup>1918</sup> | X | X <sup>1918</sup> | X | X | X <sup>1918</sup> | X | | | | | X <sup>1918</sup> | | | X | | | | X <sup>1918</sup> | | X |
| Blood sample for<br>plasma and serum<br>biomarkers <sup>4</sup> | | | | X | | | | X | | | | | | | | X | | | X | | | | X | | |
| Brain MRI <sup>2120</sup> | | X | | | | | | | | | X | | | | | | X | | | | | | | X | |
| CDR <sup>2625</sup> | X | | | | | | | | | X | | | | | | | X | | | | | | | X | |
| NPI-10 | | | X | | | | | | | X | | _ | | | | _ | X | | | | _ | | | X | |
| ISLR | X | | | | | | | | | | | | | | | | | | | | | | | | |
| ISLT | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | |

and procedures

| Study Week | Bas | seline So | creening | | | | | | | | | Place | bo-con | trolled | Period <sup>4</sup> | ,5,6 | | | | | | | | | FU <sup>7</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Period <sup>1,2</sup> within 65 days <sup>3</sup> of Day 1 | | | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 76<br>EOT | 78/<br>EOS<br>or<br>ET <sup>8</sup> | 90 |
| Study Day | S1 | S2 | S3 <sup>9</sup> | 1 | 29<br>±7 | 57<br>±7 | 85<br>±7 | 113<br>±7 | 141<br>±7 | 169<br>±7 | 197<br>±7 | 225<br>±7 | 253<br>±7 | 281<br>±7 | 309<br>±7 | 337<br>±7 | 365<br>±7 | 393<br>±7 | 421<br>±7 | 449<br>±7 | 477<br>±7 | 505<br>±7 | 533<br>±7 | 547<br>±7 | 631<br>±7 |
| DKEFS Category<br>Fluency and Letter<br>Fluency tests | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | |
| DSST | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | |
| Trails A | X | | X | | | | X | | | | X | | | X | | | | X | | | X | | | X | |
| eCog (39-item version) | | | X | | | | | | | | X | | | | | | | X | | | | | | X | |
| ADAS-Cog- 13 <sup>26</sup> | | X | X | | | | | | | X | | | | | | | X | | | | | | | X | |
| FAQ | | | X | | | | | | | X | | | | | | | X | | | | | | | X | |
| ADCS-ADL | | | X | | | | | | | X | | | | | | | X | | | | | | | X | |
| C-SSRS <sup>26</sup> | | X | X | | | | | | | X | | | | | | | | X | | | | | | X | |
| MMSE | X | | | | | | X | | | X | | | | X | | | X | | | | X | | | X | |
| RUD-Lite | | | X | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | |
| ZBI | | | X | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | |
| QoL-AD | | | Х | | | | | | X | | | | | | | X | | | | | X | | | X if<br>ET | |
| AE reporting | | | | | | | | • | I | Monitor | and reco | ord con | tinuous | ly begii | nning o | n Day 1 | at the st | art of c | losing | • | | | • | | |
| SAE reporting | | | | | | | | | Moni | itor and | record | contin | uously | throug | ghout tl | he study | | | | | | | | | |
| Concomitant therapy | Monitor and record continuously throughout the study Monitor and record continuously throughout the study | | | | | | | | | | | | | | | | | | | | | | | | |

| reporting | | |
|---|---|---|
| Ab = antibodies; AD | D = Alzheimer's disease; ADAS-Cog 13 = Alzheime | ner's Disease Assessment Scale-Cognitive (13 item); ADCS-ADL = Alzheimer's Disease |
| Cooperative Study | - Activities of Daily Living; AE = adverse event; | ; CDR = Clinical Dementia Rating Scale; |

# CONFIDENTIAL

| ; C-SSRS = Columbia - Suicide Severity Rating Scale; DBP = diastolic blood pressure; DKEFS = Delis-Kaplan Executive Function System; DSST = Digital Control of the Control |
|---|
| Symbol Substitution Test; ECG = electrocardiogram; eCog = Everyday Cognition; EOS = end of study; EOT = end of treatment; ET = early termination; |
| FAQ = Functional Activities Questionnaire; FU = follow up; HbA1c = glycosylated hemoglobin; HIV = human immunodeficiency virus; ICF = informed |
| consent form; ; ISLR = International Shopping List Test Delayed Recall; ISLT = International Shopping List Test |
| Immediate Recall; ; MMSE = Mini-Mental State Examination; MRI = magnetic resonance imaging; NIA-AA = National Institute on |
| Aging – Alzheimer's Association; NPI-10 = Neuropsychiatric Inventory-10; |
| ; QoL-AD = Quality of Life in Alzheimer's Disease; ; RUD-Lite = Resource Utilization in Dementia-LightLite |
| Version; SAE = serious adverse event; SBP = systolic blood pressure; Trails A = Trail Making Test Part A; ZBI = Zarit Burden Interview |
| The screening process will generally involve up to 3 visits, and most screening procedures will be performed within these designated visits (S1-S3). However |
| additional screening visits may be needed for some procedures, e.g., MRI |
| assessments (e.g., if the MRI scan does not pass the quality control process). Brain MRI (S2) will only be performed after the subject has met the eligibility |
| criteria and has acceptable laboratory tests from Visit S1. |

- The clinical assessments performed during Visit S1 are to be administered in the order specified: 1) MMSE; 2) neuropsychological tests in the following order: ISLT, DSST, Trails A, Category Fluency and Letter Fluency tests from the DKEFS, ISLR; 3) CDR. Note that the Visit S1 results from CDR, ISLT/ISLR, and MMSE will be used to determine subject eligibility; Visit S3 ISLT assessments will provide baseline measures. At Visit S3, the clinical assessments will be administered as follows: 1) neuropsychological tests in the following order: ISLT, DSST, Trails A, Category Fluency and Letter Fluency tests from the DKEFS; 2) ADAS-Cog 13; 3) OoL-AD.
- The nominal It is recommended that all the screening procedures be completed within 65-day days; however, the overall screening period may be increased with the permission of extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate ( ). The following screening assessments should be repeated if the screening period is >65 days: confirmation of eligibility criteria, abbreviated medical history, and physical examination, ECG, hematology, elinical chemistry, and serum pregnancy test (women of childbearing potential). In addition, some cognitive and /or safety assessments may require repeating depending on the duration of the screening window extension, in discussion with the Medical Monitor.
- <sup>4</sup> All assessments and blood collection during dosing days will be performed prior to infusion, unless otherwise specified. Doses should be administered at least 21 days apart.
- <sup>5</sup> The visits at Weeks 32, 36, 44, and 64 may qualify for home visits, if appropriate; see Section 7.1 for details.
- <sup>6</sup> Prior to initiation of and/or a change in AD medication, a subject should have an unscheduled visit for assessment of AEs/serious-SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ.
- <sup>7</sup> Subjects who complete the Treatment Period and do not enter an extension study (separate protocol, to be initiated at the Sponsor's discretion) are to return to the study site for a Follow-up Safety Visit at Week 90. Subjects who discontinue study treatment and withdraw from the study early are to have a Follow-up Safety Visit 14 weeks after the final dose. Subjects who discontinue study treatment prematurely are to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment.
- <sup>8</sup> All subjects who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures. These subjects should be encouraged to attend at least the Week 24, Week 52, and Week 78 visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Subjects who discontinue study treatment prematurely will also be asked to return to


the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment (see Table 1 for the schedule of assessments). Subjects who withdraw from the study prematurely are to return to the study site for an ET visit and ET assessments. If the withdrawn subject has discontinued treatment within 3 months of the previous primary efficacy assessment (CDR) and no significant changes in cognitive status are suspected by the Investigator, the clinical efficacy assessments specified in the ET visit are not required; the study site should notify the Sponsor in such cases. An MRI scan should be performed if withdrawal occurs  $\geq$ 6 months after the previous MRI. Blood for biomarker analysis should be collected if the subject withdraws  $\geq$ 4 weeks after the previous sample was collected.

Visit S3 all clinical assessments must be scheduled within 7 days before Study Day 1 or performed at Study Day 1 before randomization,

Subjects and the subjects' partners/informants or their legally authorized representatives, and the subjects' partners/informants or their legally authorized representatives, and the subjects' partners/informants or countries where applicable laws allow, may sign this optional form for an initial screening which allows administration of the CDR, MMSE, ISLT/ISLR, DKEFS Category Fluency and Letter Fluency tests, DSST, and Trails A to determine eligibility based on cognitive assessments. The order of assessments is as specified in footnote 2.

<sup>11</sup>All subjects **and the subjects' partners/informants** or their legally authorized representatives, and the subjects' partners/informants in countries where **applicable laws allow**, must sign this full informed consent, including those who have previously signed the optional initial screening consent and have met the eligibility criteria based on cognitive assessments.

<sup>12</sup>Pregnancy testing is required for women of childbearing potential only; for these subjects, a serum pregnancy test is to be performed at Screening and EOS (or ET) Visits, and a urine pregnancy test is to be performed at every dosing visit.

<sup>13</sup>Women who report postmenopausal status at Visit S1 must have a follicle-stimulating hormone test at that visit to confirm that they are not of childbearing potential.

<sup>14</sup>To be performed based upon Investigator assessment of HIV risk factors. The requirement for testing during Screening may be omitted if it is not permitted by local regulations.



<sup>16</sup>Triplicate 12-lead (paper) ECGs will be obtained at each specified timepoint. ECGs are to be performed in triplicate, with each ECG performed about 1 minute apart and before blood draws on appropriate days. In addition, triplicate ECGs will also be performed <del>15 minutes</del> 1 hour after the end of infusion on Study Day


1 only. Each ECG must be performed after the subject has been resting (supine) for 10 minutes. ECGs will be read by a central reading facility. Clinical significance of potential ECG abnormalities will be determined by the Investigator.

<sup>&</sup>lt;sup>2120</sup>Brain MRI may include, but will not be limited to, the following sequences: 3D T1 weighted, fluid attenuated inversion recovery, T2\* weighted, diffusion weighted imaging, and proton density/T2 weighted MRI. For further details on MRI sequences, please see the procedural manual for MRI. To occur after cognitive testing has concluded for the sScreening pPeriod. After randomization, the visit date for this MRI can vary by ±10 days from the specified visit day.



<sup>2625</sup> Postbaseline It is recommended that postbaseline CDR assessments should be conducted within ±1 hour of at the same time of day at which the baseline assessment was performed to avoid diurnal violation. The rater who conducts the CDR for a subject/partner informant cannot complete any other rating scales for that same subject/partner or be the study site coordinator and will be blinded to all other study-related data.


<sup>&</sup>lt;sup>17</sup>Vital signs will include SBP, DBP, heart rate, body temperature, and respiratory rate and will be measured with the subject supine and after the subject has been resting for at least 10 minutes. In addition, blood pressure and heart rate will be measured after the subject has been standing for ≥2 minutes at the following timepoints: preinfusion and 1 hour (±15 minutes) after the end of infusion on Days 1, 29, 57, and 85. Three separate SBP/DBP readings at least 15 minutes apart will be made at the Screening Visit to determine eligibility. Single vital sign readings will be obtained at other timepoints.

<sup>&</sup>lt;sup>18</sup>Fasting is required prior to safety laboratory tests.

<sup>&</sup>lt;sup>1918</sup>Two samples must be obtained: 1 sample taken before infusion and 1 sample taken at ≤10 minutes after the end of infusion.

<sup>&</sup>lt;sup>2019</sup>The results are not required for randomization.

During the screening period, ADAS-Cog 13 and C-SSRS are scheduled at Visit S2; however, they may be performed at Visit S1, if more convenient per site and subject's availability. If ADAS-Cog 13 and C-SSRS assessments are performed at Visit S1, all other clinical assessments should be performed before ADAS-Cog 13, followed by C-SSRS.

### **Rationale:**

In footnote #3 and footnote #22 (now footnote #21), text was added to clarify that the screening period may be extended to 90 days, if needed, the Sponsor's approval.

Footnote #3 was modified to clarify the assessments that are to be repeated if the screening period is increased to 90 days.

In footnote #9, the timing of clinical assessments at Screening Visit 3 was updated to provide flexibility to be performed at Study Day 1, in case of site's and/or subject's availability,

In footnote #15, the timing window was increased to reduce burden on subjects and to allow appropriate time for review of the coagulation tests results. Additional text was added to clarify that the repeats test may be performed locally.

Footnote #16 was updated to increase the timing window and facilitate performing the ECG after the end of infusion on Study Day 1, now timed with vital sign assessment.

Footnote #18 (Version 1) was deleted. No safety concerns are expected with removal of the fasting requirement. It would be difficult to confirm compliance with the requirement of fasting across the study and the number of protocol deviations for blood sample collection. Furthermore, cognitive testing and, particularly, the primary efficacy endpoint, the CDR sum of boxes, are often performed on the same visit as the collection of blood samples for hematology and clinical chemistry laboratory assessments. Requiring this elderly subject population to fast before performing cognitive assessment tests may increase the variability in the data collected at these visits.

In footnote #25, the timing of the postbaseline CDR assessments was updated to allow additional flexibility in the schedule of study visits and reduce burden on subjects.

The timing of ADAS-Cog-13 and C-SSRS assessments during the screening period was updated to allow some flexibility and therefore reduce burden on subjects (footnote # 26 was added).

Clarification was made to the serious AE and concomitant medication reporting in the Schedule of Activities table, that it will be collected throughout the study, including during the screening period and made consistent with Section 15.3.3, Serious Adverse Events.

This change also affects Section, 7.1, Study Overview; Section 7.2, Study Duration for Subjects; Section 9.1, Screening; Section 13.1, Clinical Efficacy Assessments; Section 14.2, Laboratory Safety Assessments; and Section 15.3.1, Adverse Events.

# Section 6, Study Objectives and Endpoints

**Change:** An update was made to primary safety endpoints, pharmacokinetic (PK) and pharmacodynnamic objectives and endpoints.

# Now reads:

| Primary Objective | Primary Endpoints |
|---|---|
| To evaluate the safety and tolerability of BIIB092 in subjects with MCI due to AD or with mild AD | Incidence of AEs and /serious AEs (SAEs) from Baseline to the end of the study treatment period.; incidence of abnormalities and changes from Baseline over time in laboratory safety assessments (including elinical chemistry, hematology, and urinalysis), vital signs, and 12 lead electrocardiograms (ECGs); and changes in physical examination findings. |

| <b>Exploratory Objectives</b> | Exploratory Endpoints |
|---|---|
| To assess BIIB092 eoneentrations PK in serum following multiple doses in subjects with MCI due to AD or with mild AD. | Changes from, Baseline over time up to Week 90 in serum BIIB092 concentration Trough serum BIIB092 concentrations and end-of-infusion serum BIIB092 concentrations from the samples collected at the visits indicated in the schedule of activities. |

**Rationale:** The primary endpoint text was updated to facilitate handling of data disclosed to ClinicalTrials.gov and other registries under transparency requirements.

The exploratory PK objectives and endpoints were updated to streamline the generated data and PK evaluation. For the PK evaluation, the actual drug levels are used, not the changes from baseline.



### Section 8.1, Inclusion Criteria

### Change:

The eligibility criteria text related to informed consent was updated.

The International Shopping List Test Immediate Recall (ISLT) or International Shopping List Test Delayed Recall (ISLR) score requirement was modified.

#### Now reads:

To be eligible to participate in this study, candidates must meet the following eligibility criteria at Screening, or at the timepoint specified in the individual eligibility criterion listed:

1. Ability of the subject or his/her informant/study partner and/or legally authorized representative to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations. In countries where applicable laws allow, the participant's informant/study partner and/or legally authorized representative may provide informed consent in lieu of the subject's signature.

. . . . .

- 5. Must meet all of the clinical criteria for MCI due to AD or mild AD according to the NIA-AA [McKhann 2011], and in addition must have the following at Screening Visit 1:
  - ISLT or ISLR score ≤1 SD below of the age-adjusted normative mean
  - CDR global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD
  - MMSE score of 22 to 30 (inclusive)
  - CDR Memory Box score of ≥0.5

. . . . . .

**Rationale:** The text was updated to clarify that applicable laws will be followed in case of subject's loss of capacity of consent.

The ISLT or ISLR score was clarified as per recommendation from the Cogstate Science Team.

This change affects Section 5, Schedule of Activities (Footnote #10 and Footnote #11), Section 9.1, Screening, Section 15, Safety Definitions, Recording, Reporting, and Responsibilities and Section 17.3, Subject Information and Consent.

# Section 8.2, Exclusion Criteria

**Change:** The eligibility criterion regarding vaccination was updated.

#### Now reads:

26.30. Vaccinations within 710 days prior to randomization (Study Day 1).

**Rationale:** Exclusion criterion #26 (now exclusion criterion #30), was modified to exclude vaccinations within 10 days prior to randomization to be consistent with allowed vaccinations during the study as outlined in Section 14.1.1.1, Allowed Concomitant Therapy.

# Section 9.1, Screening

**Change:** Rescreening requirements for subjects were updated.

### Now reads:

Subjects who fail screening may be rescreened once at the Sponsor's discretion,

MMSE, hepatitis B or C criteria, having a CDR global score >1, or abnormal CONFIDENTIAL

Section 9.2 Randomization

MRI findings. Note: Subjects with a CDR global score of 0 but who meet the other entry criteria may repeat the screening after 6 months from the initial evaluation.

**Rationale:** Screening failures due to failed key clinical assessments will not be allowed to rescreen. Rescreening for subjects who meet entry criteria except having a normal CDR global score of 0 is allowed to capture subjects who are at risk of cognitive decline over the following 6 months.

| Section 7.2, Italiaanii Eatlai |
|--------------------------------|
| Change: |
| Now reads: |
| Rationale: |

# Section 11.2.2, Infusion Interruption

**Change:** Additional text related to infusion time, use of premedication, and management of infusion-related reactions was added.

#### Now reads:

The IV administration infusion time for all treatment groups is 1 to 2 hours at approximately 100 mL/hour. No premedications should be used prior to the start of study treatment infusion unless discussed with the Medical Monitor in advance and written documentation is received from Biogen authorizing the use of the premedication.

• If any mild or moderate infusion-related reactions occurs during an infusion, the infusion should be slowed or interrupted, and supportive treatment should be instituted. Upon resolution of symptoms, if the infusion had been slowed, the original infusion rate may be resumed; the infusion may be slowed or interrupted and appropriate treatment per local standards of care may be given at the discretion of the Investigator (or designee). Based on the clinical response, the Investigator or designee will determine if the infusion may be resumed/continued in consultation with the Medical Monitor as needed. If the infusion is


resumed/continuedhad been interrupted, the infusion rate may be restarted at a rate that does should not exceed the original infusion rate -(sSee the DHA for infusion rate information-).

If a severe infusion-related reaction occurs during an infusion, the subject should be
permanently discontinued from treatment. Severity and appropriate supportive care
must be initiated in accordance with local practice.

Criteria for determining the severity of events is are described in Section 15.2.3.

Discussion with the Medical Monitor can occur as needed, and it should not delay management of the medical emergency.

Refer to Section 15.3 for reporting of AEs and Section 10 for discontinuation of study treatment.

**Rationale:** Additional text was added to provide details on administration of BIIB092 and management of infusion reactions, should a subject experience an infusion reaction event during the study. This change is provided at the request of the Swedish Medical Products Agency. Because this change relates to clarification of safety measures, it is also made available to all the participating sites within the global protocol.

### Section 13.2, Pharmacokinetic Assessments

**Change:** The methodology of PK assessments was updated.

#### Now reads:

Serum PK parameters of BIIB092 to will be ealculated using a nonlinear mixed effects approach. These parameters assessed may include, but will not be limited to, the following:

- Maximum observed concentration (C<sub>max</sub>)
- Area under the concentration time curve End of infusion concentration

**Rationale:** The text was updated to make the analysis methodology compatible with the data to be generated in this study. This study will only inform about the peak and trough concentrations, which will not be enough for a nonlinear mixed effects model.

A nonlinear mixed effects model is planned as a meta-analysis, combining data from multiple other studies, and will be conducted and reported separately.


Section 15.2.1, Investigator Assessment of Events



# Section 15.4.3.1, Unblinding for Medical Emergency

**Change:** The text regarding different ways of accessing the interactive response technology (IRT) system was modified.

#### Now reads:

In a medical emergency when knowledge of the subject's treatment assignment may influence the subject's clinical care, the Investigator or appropriate designee may access the subject's treatment assignment byin the IRT system by accessing the internet or using a phone-based interface. Further information about the IRT unblinding function or 24-hour, 7-day-a-week support contact information is available in the IRT manual for the study.

The Investigator must document the reasons for unblinding in the subject's source documents. The Investigator is strongly advised not to divulge the subject's treatment assignment to any individual not directly involved in managing the medical emergency, or to personnel involved with the analysis and conduct of the study.

The Investigator can contact Biogen or its designee to discuss such situations, but such a discussion should not delay management of the medical emergency. The Investigator should inform Biogen or its designee as soon as possible if unblinding occurs.

**Rationale:** This change was made to clarify how to access the IRT system in the case of unblinding for a medical emergency and that unblinding for a medical emergency can be completed at any time. This change is provided at the request of the Swedish Medical Products Agency. Because this change relates to clarification of the process of unblinding for a medical emergency, it is also made available to all the participating sites within the global protocol.

# Section 16.9, Interim Analyses

**Change:** Text regarding review by an independent team of interim analysis data for the purpose of future study planning was added.

Text regarding the interim analyses was modified.

### Now reads:

Interim analyses may be performed after 50% to 70% of, or all, 50% to 100% of subjects have completed the Week 52 visit (or discontinued) for the purpose of future study planning and/or futility analyses. In order to maintain the treatment blind, an independent group external to Biogen that will not be involved in the conduct of the study after unblinding will perform the interim analyses. This independent group will present the unblinded interim analyses to the DMC for review. After the DMC review, a small internal independent team (separate from the study team) may review the unblinded results for the purpose of future study planning under a study integrity charter. No Type I error adjustment will be made. No changes will be made to this study based on the interim analysis results.

**Rationale:** The text was added to clarify how unblinded outputs from interim analysis that may support clinical study design of future studies will be evaluated. A small internal team independent from the study team will be involved in this evaluation to avoid any influence of this assessment on study conduct.

The text regarding interim analyses was modified to clarify that one or more interim analyses may be performed when between 50% and 100% of subjects have completed the Week 52 visits (or discontinued).

### SUMMARY OF MINOR CHANGES TO THE PROTOCOL

The following minor changes were made to the protocol, as appropriate:

- The version number and date were updated throughout the protocol.
- On the Sponsor Signature Page, the signatory for this protocol was changed.
- Resource Utilization in Dementia (RUD)-Light was corrected to RUD-Lite throughout the protocol.
- •
- ADAS-Cog-13 was updated to ADAS-Cog 13, throughout the protocol.
- Section 2, List of Abbreviations was updated.
- In Section 8.2, Exclusion Criteria, eligibility requirement related medical history was clarified (exclusion criterion 6 was updated and exclusion criterion 7 was called out to be a separate criterion.
- In Section 8.2, Exclusion Criteria #9 (now reads #10), eligibility requirement related to brain magnetic resonance imaging (MRI) was updated.
- In Section 8.2, Exclusion Criteria, eligibility requirement related to impaired liver and renal function were separately called out for clarification) now reads as exclusion criteria #20 and #21).
- In Section 8.2, Exclusion Criteria #38 (now reads #45), eligibility requirement related to enrollment any other interventional clinical study was modified.
- In Section 11.5, Continuation of Treatment, text was updated to clarify the planned long-term extension of this study. This changes also affects Section 5, Schedule of Activities (footnote 7), and Section 7.2, Study Duration for Subjects.
- In Section 12.1, BIIB092, the amount per vial and details regarding excipients/components were removed.
- In Section 15, Safety Definitions, Recording, Reporting, and Responsibilities, an
  administrative change was made to notify Biogen instead of Quintiles in case of a
  safety event. This also affects Section, 19.1.1, Contract Research Organization.
- In Section 19.1.3, Electronic Data Capture, text was modified to clarify the Sponsor's definition of source data in the study.


- In Section 17 and Section 19, reference to Quintiles was updated to Contract Research Organization (CRO) to avoid a protocol amendment if there is a change in vendor.
- Typographical errors and formatting were corrected.



Biogen MA Inc. 225 Binney Street Cambridge, MA 02142 United States

Biogen Idec Research Limited Innovation House 70 Norden Road Maidenhead Berkshire SL6 4AY United Kingdom

# **AMENDMENT SUMMARY**

Biogen Protocol 251AD201

Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with Mild Alzheimer's Disease

Version 3

Date: 29 March 2019

EUDRA CT Number: 2017-002901-37

Version 3 of the protocol has been prepared for this amendment, which supersedes Version 2.

# PRIMARY REASON FOR AMENDMENT

The primary reason for this amendment to Protocol 251AD201 is to add a dose-blinded long-term extension (LTE) period of approximately 3 years. The primary purpose of the LTE is to obtain long-term safety and tolerability information on BIIB092 and further explore its effects on immunogenicity, disease progression, and additional clinical and health outcomes.

New text is shown in **bold** type; deleted text is shown with a strikethrough.

Section 7.1, Study Overview

Now reads:

. . .

The study consists of a double-blind, placebo-controlled period and a dose-blinded LTE period. The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. For participants who complete both the placebo-controlled period and the LTE period, the total study duration will be approximately 247 weeks. The placebo-controlled period comprises a Screening Period of up to approximately 9 weeks (65 days), a Treatment Period of 76 weeks, and for participants not entering the LTE period, an End-of-Study (EOS) Visit at Week 78 and a Follow-up Safety Visit at Week 90, or approximately 14 weeks after the last dose of study treatment. However, the overall sScreening Period for the placebo-controlled period may be extended up to 90 days in consultation with the Medical Monitor in advance and provided that written documentation is received from the Sponsor or delegate (e.g., for logistical issues such as PET radioligands). At the end of the placebo-controlled period, participants who meet the LTE entry criteria may enter the dose-blinded LTE period. The LTE period comprises an LTE Screening Period of approximately 4 weeks starting at Week 76, a 144-week Treatment Period, an EOS Visit at Week 226, and a Follow-up Safety Visit at Week 238, or approximately 14 weeks after the last dose of study treatment.

. . .

During the LTE period, participants who were randomized to receive BIIB092 during the placebo-controlled period will continue to receive BIIB092 at the dose they were randomly assigned. Participants receiving placebo during the placebo-controlled period will receive BIIB092 at the high dose (2000 mg) once every 4 weeks during the LTE period. The BIIB092 dose concentration (i.e. low, medium, or high) to which participants are assigned to receive during the LTE period may be changed based on emerging data from the BIIB092 clinical development program.

The visits at Weeks 84, 88, 96, 112, 116, 120, 136, 140, 144, 160, 164, 168, 184, 188, 192, 208, 212, and 216 of the LTE period may be conducted as home visits, if the Investigator is in

agreement and appropriate services are available to perform the required study procedures and adequately monitor for potential safety events. These are study visits that do not require extensive assessments, e.g., administration of clinical scales or the conduct of MRI, MRI, However, if the participant experienced a clinically significant infusion reaction during the first 24 weeks of the LTE period, then the BIIB092 infusion should not be administered in the home unless previously approved by the Investigator.

Throughout the study, all participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient monitoring facility until the Investigator has determined that these event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

Investigators, study staff (except for a designated Pharmacist/Technician), and study subjects participants and their families, caregivers, and legal representatives will be blinded to the subjects' participants' randomized treatment assignments and, during the LTE period, the BIIB092 dose.



The schedule of study assessments is presented in Section 5.

Figure 1: Study Schematic Design

# Deleted Figure:



# **Inserted Figure:**



 $A\beta$  = amyloid beta; AD = Alzheimer's disease; EOS = End of Study; LTE = long-term extension; MCI = Mmild Ccognitive Impairment; N = number of subjects participants; Q4W = once every 4 weeks; Q12W = once every 12 weeks

Note: Overall, participating subjectsparticipants will have a 2:1 chance of being randomized to BIIB092 versus placebo during the placebo-controlled period, and all participants will receive BIIB092 during the dose-blinded LTE period.

Note: The study comprises a double-blind, placebo-controlled period and an LTE period. The total duration for participants who complete the placebo-controlled period and do not enter the LTE period will be approximately 99 weeks. The total study duration for participants who complete both the placebo-controlled period and the LTE period will be approximately 247 weeks. The double-blind placebo-controlled period comprises a Screening Period of up to-approximately 9 weeks (65 days), a Treatment Period of 76 weeks, and for participants not entering the LTE period, an End of Study EOS Visit at Week 78, and a Follow-up Safety Visit at Week 90, or approximately 14 weeks after the last dose of study treatment. The LTE period comprises an LTE Screening Period of approximately 4 weeks starting at Week 76, a 144-week Treatment Period starting at Week 80, an EOS Visit at Week 226, and a Follow-up Safety Visit at Week 238, or approximately 14 weeks after the last dose of study treatment.

**Rationale:** To date, BIIB092 has been generally well tolerated in the clinical study participants. There are no important identified or important potential risks in the program, including in the completed studies CN002001 and CN002003 and in the ongoing studies 251PP201, 251PP301, and 251AD201. The current safety profile supports continued investigation of the proposed doses of 125 to 2000 mg. The LTE will provide additional long-term safety data.

Switching all participants who received placebo during the placebo-controlled period to 1 group (2000 mg every 4 weeks) in the LTE period allows delayed start analysis to be maximized for 1 of the dose groups.

This change also affects Section 5, Schedule of Activities (addition of 3 new tables for the LTE period); Section 6, Study Objectives and Endpoints; Section 7.2, Study Duration for Participants; addition of Section 8.3, Inclusion Criteria for Long-Term Extension Period and Section 8.4, Exclusion Criteria for Long-Term Extension Period; Section 9.1 Screening; Section 9.2, Randomization; Section 9.3, Blinding Procedures; Section 10.1, Discontinuation of Study Treatment; Section 11.1, Regimen; Section 11.5, Continuation of Treatment; Section 13.6, Immunogenicity; and Section 16, Statistical Methods and Determination of Sample Size.
### SUMMARY OF MAJOR CHANGES TO THE PROTOCOL

Changes to the protocol are presented chronologically. New text is shown in **bold** type; deleted text is shown with a strikethrough.

## Section 1, Synopsis

The Synopsis was revised to reflect changes made throughout the protocol.

### Section 4.5, Overall Benefits and Risk Assessment

**Change:** Updated the benefits and risks assessment information.

#### Now reads:

Due to its eTau lowering effects, BIIB092 has the therapeutic potential to prevent transmission of tau pathology in neurodegenerative disorders known as tauopathies, which include PSP and AD. The proposed indications under the current program of research are for use in patients with PSP and AD.

To date, 2 clinical studies have been completed with BIIB092. These include the first in human study, CN002001 (SAD study in healthy adult subjects) and CN002003 (MAD study in subjects with PSP). In addition to this study, 2 studies are ongoing: Study 251PP201 (formerly referred to as CN002004), an open label extension study, and Study 251PP301 (formerly referred to as CN002012), a Phase 2b randomized controlled efficacy and safety study in subjects with PSP. Please refer to Section 4.3.2 for more information.

All available clinical benefit and risk information to date has been derived from studies in healthy volunteers or subjects with PSP. PSP is a rare neurodegenerative disease that results in a rapidly progressing, fatal movement disorder that includes cognitive and behavioral abnormalities. There are currently no approved or effective treatments for PSP. Nonclinical models support the anti-eTau mechanism as potentially efficacious in the treatment of PSP.

Binding to eTau, the murine antibody from which BIIB092 is derived, prevented tau transmission in nonclinical studies. Furthermore, the murine antibody from which BIIB092 was derived prevented tau dependent behavioral and pathologic changes in a mouse model of tauopathy. Finally, BIIB092 reduced free eTau levels in the CSF of cynomolgus monkeys following a single IV administration. For additional details, please refer to Section 4.3.1. By binding eTau, it is expected that BIIB092 will prevent tau transmission in diseases such as AD and PSP and thereby potentially provide therapeutic benefit.

The nonclinical toxicity profile of BIIB092 was used to determine the starting dose and eligibility criteria and to develop appropriate safety monitoring for BIIB092 studies. Clinical data from the completed first in human SAD study in healthy adult subjects (CN002001) demonstrated that single doses of BIIB092 up to 4200 mg in Caucasian subjects and up to 2100 mg in Japanese subjects were generally safe and well tolerated. The completed (MAD) study in subjects with PSP (CN002003) evaluated multiple doses of BIIB092 (150, 700, and 2100 mg) or placebo administered once every 4 weeks for 3 months. The available data suggest that multiple doses of BIIB092 up to 2100 mg are safe and well tolerated in subjects with PSP. Correspondingly, the current ongoing open label, long term extension, safety and tolerability study (251PP201) also suggests that multiple doses of BIIB092 up to 2100 mg are safe and well tolerated in subjects with PSP.

Frequent safety assessments will be utilized by the Sponsor/Medical Monitor and Investigators to determine whether dose modification, additional safety measures, or termination of the ongoing studies is required at any time. Serum immunogenicity sampling will be performed to monitor for the emergence of anti-drug antibodies. Thorough evaluation of safety monitoring procedures and of AEs and serious adverse events (SAEs) will be reviewed on an ongoing basis by the Sponsor's Medical Monitor and Global Pharmacovigilance representatives to monitor for any safety signals or trends.

In addition, an independent Data Monitoring Committee (DMC) was established to monitor the benefit/risk profile of BIIB092.

For information on specific risk mitigation strategies, please refer to Section 10, Section 11.2.2, and Section 15.4.

A need exists for disease modifying therapies for participants with AD and those with PSP. The doses of BHB092 currently being explored have the potential to benefit study subjects. Furthermore, the nonclinical efficacy profile and the evidence for anti eTau activity, together with the benign safety profile, indicate that the balance of benefit to risk is likely to be favorable for study subjects.

### 4.5.1. Overall Benefit

BIIB092 has the potential to slow or stop the spread of tau pathology observed in neurodegenerative diseases such as PSP, AD, and other tauopathies.

In participants with PSP, BIIB092 has been evaluated in 2 completed clinical studies (Studies CN002001 and CN002003) and is currently being evaluated in the ongoing Studies 251PP201 and 251PP301. The first-in-human study of BIIB092 (Study CN002001) was designed as a randomized, double-blind, placebo-controlled, SAD study in healthy participants to characterize the safety, tolerability, PK, PD, and immunogenicity of single doses of BIIB092, ranging from 21 to 4200 mg. Study CN002003, a Phase 1b study, was designed as a randomized, double blind, placebo-controlled MAD study to characterize the safety, tolerability, PK, PD, and immunogenicity of multiple doses of BIIB092, ranging from 150 to 2100 mg, in participants with PSP. In both of these completed studies, BIIB092


was found to be well tolerated at the doses tested in both healthy participants and participants with PSP. The ongoing Phase 1b study, Study 251PP201, is designed as an open-label extension study to evaluate the long term safety and tolerability of multiple doses of BIIB092 in participants with PSP who participated in Study CN002003. Several interim analyses of the data being collected in this study have been performed to date. Study 251PP301 is an ongoing Phase 2b study designed as a randomized, double blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of IV administered BIIB092 in participants with PSP.

In participants with AD, this study (Study 251AD201) will evaluate the safety and efficacy of BIIB092.

Based on the PK and PD data from Studies CN002001 and CN002003, the mean concentrations of BIIB092 in CSF increased in a generally dose-proportional manner. A robust and persistent lowering of unbound N-terminal tau was observed following administration of single and multiple doses of BIIB092 in healthy participants and in participants with PSP, consistent with the observations in cynomolgus monkeys.

#### 4.5.2. Potential Risks

The nonclinical studies conducted to date have demonstrated an acceptable safety profile for BIIB092 to support continued use in clinical studies.

As of 25 November 2018, an estimated 486 healthy participants or participants with PSP or AD have been exposed to BIIB092 in clinical studies. The following summary of the safety profile of BIIB092 is based on safety data from the completed Studies CN002001 and CN002003 and the ongoing Study 251PP201. In the SAD study in healthy participants, there were no safety findings of note, and development continued in patients with PSP. In participants with PSP, to date, the most commonly reported AEs were fall, urinary tract infection (UTI), contusion, and headache. Most AEs have been reported as mild or moderate in intensity. Serious AEs (SAEs) have generally been consistent with disease (UTI, respiratory arrest, aspiration pneumonia, and progressive PSP) or are not unexpected in the patient population enrolled in the trials (cholecystitis, cancer, fractures, and anemia). There have been 3 deaths, all of which were likely related to underlying disease (respiratory arrest, aspiration pneumonia, and progressive disease). None of the SAEs or deaths were considered related to BIIB092 by Investigators. No safety concerns have been identified from laboratory, vital signs, or electrocardiogram (ECG) assessments. Nonserious infusion reactions have been observed and are an identified risk of BIIB092.

BIIB092 is a humanized IgG4 monoclonal antibody. While a low risk of immunogenicity is suggested by preclinical studies, the risk of immunogenicity in humans is unknown. Immunogenicity is an AE of special interest that is under monitoring in all ongoing studies. No safety data regarding this topic have emerged that would change the safety profile of BIIB092.

In general, BIIB092 has been well tolerated in the clinical study participants. There are no important identified or potential risks in the program. The safety profile is acceptable to continue development.

# **4.5.3.** Summary

Currently available treatments for AD offer modest symptomatic relief, but none has the potential to modify the underlying disease pathology or course of the disease. In addition, no medications have been approved for the treatment of PSP. Therefore, there is a significant unmet need for the development of effective disease-modifying therapies in both PSP and AD.

Based on the PK and PD data from Studies CN002001 and CN002003, the mean concentrations of BIIB092 in CSF increased in a generally dose-proportional manner. A robust and persistent lowering of unbound N-terminal tau was observed following administration of single and multiple doses of BIIB092 in healthy participants and in participants with PSP, consistent with the observations in cynomolgus monkeys.

Based on the safety data from the completed Studies CN002001 and CN002003 and the data from an interim analysis of the ongoing Study 251PP201, BIIB092 was generally well tolerated and demonstrated an acceptable safety profile for continued development.

The overall analysis of potential benefits (based on the robust and persistent lowering of unbound N terminal tau in healthy participants and in participants with PSP, consistent with cynomolgus monkeys) and risks (available safety data indicating that BIIB092 is generally well tolerated) supports the continued development of BIIB092 in both PSP and AD.

**Rationale:** Updated the benefit and risk assessment information for BIIB092 to align with the Investigational Medicinal Product Dossier. Note that the overall risk and benefit assessment remains unchanged as a result of this update.

### Section 7.1, Study Overview

**Change:** Require that participants be observed for a minimum of 1 hour after the end of infusion on dosing visits.

| N | $\mathbf{ow}$ | read | ls: |
|---|---------------|------|-----|
|---|---------------|------|-----|

. . .

Throughout the study, all participants should be observed and monitored by study staff for a minimum of 1 hour after the end of an infusion. Participants who experience an AE or SAE related to BIIB092 infusion should remain at the site or be sent to an inpatient

monitoring facility until the Investigator has determined that the event(s) has resolved or do not require further monitoring at the site or in an inpatient setting.

**Rationale:** The requirement to monitor participants for 1 hour after dosing was added to further ensure the safety of the participants.

This change also affects Section 5, Schedule of Activities and Section 7.2, Study Duration of Participants.

# Section 8.1, Inclusion Criteria



### Section 8.2, Exclusion Criteria

**Change:** Exclusion criteria regarding the participants' hepatitis B and C status, medical history, medication use, and study procedure were updated and clarified. Additionally, criterion 2was split into criteria 2 and 3, and as a result, all subsequent exclusion criteria were renumbered.

#### Now reads:

Medical history

- 2. History of, or positive test result at Screening for, Current hepatitis C virus antibody or infection (defined as positive hepatitis C virus [HCV] antibody and detectable HCV ribonucleic acid [RNA]). Participants with positive HCV antibody and undetectable HCV RNA are eligible to participate in the study (United States Centers for Disease Control and Prevention).
- 3. Current hepatitis B virus infection (defined as positive for both-hepatitis B surface antigen [HBsAg] and/or total hepatitis B core antibody [anti-HBc]) unless fully recovered with no active infection indicated by a serology panel. Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study.

. . . . .

10.11. Brain MRI performed at Screening Visit 2 (centrally read) that shows evidence of any of the following:

. . . . .

 Cortical infarct (including cerebellar infarct) [defined as >1.5 cm in diameter] or any infarct in the hippocampus.

. . . . .

- 19.20. History of premalignant or malignant disease. Exceptions to premalignant disease exclusions may be made after discussion with the Sponsor. The following exceptions may be made for malignant disease exclusions after discussion with the Sponsor:
  - SubjectsParticipants with cancers in remission ≥5 years prior to Screening Visit 1.
  - SubjectsParticipants with a history of excised or treated basal cell or squamous carcinoma of the skin
  - SubjectsParticipants with localized prostate cancer with treatment cycles that completed at least 6 months prior to Screening Visit 1.

. . . . .


Medications

2930. Use of the following medications:

. . . . .

Antipsychotics High-dose antipsychotics used on a regular basis, except for low. Low doses of atypical and typical antipsychotics (e.g., risperidone, aripiprazole, or quetiapine) if used on an as-needed basis or if used at a stable dose for 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1. The definition of "low doses" and "high dose" should be judged by the Investigator, and the Medical Monitor can be consulted if needed.

. . . . .

34.35. Participation within the 12 months prior to Screening Visit 1 in a study of any other agent(s) **not included in exclusion criteria 32, 33, and 34** with a purported disease-modifying effect in AD, unless documentation of receipt of placebo is available.

. . . .

Study Procedures

.....



### Section 9.2, Randomization

**Change:** A slight change in the ratio of study participants with mild cognitive impairment (MCI) due to AD versus mild AD was made.


### Now reads:

Enrollment will be monitored, via the interactive response technology (IRT) system, so that the population of subjectsparticipants with mild AD represents aboutapproximately 6050% of the total number of subjectsparticipants enrolled in the study.

**Rationale:** A reassessment of the ratio of study participants with MCI due to AD versus mild AD was completed. The ratio was changed as a result and is not expected to affect the objectives of the study.

# Section 14.2, Laboratory Safety Assessments



### Now reads:



# Rationale:




### Section 15.3.2, Adverse Events of Special Interest

**Change**: Immunogenicity was added as an adverse event (AE) of special interest.

Now reads:

No AEs of special interest have been identified for BIIB092 to date. Immunogenicity is an AE of special interest that is under monitoring in all ongoing studies. Participants will also be monitored for possible infusion-associated AEs and/or hypersensitivity reactions during and after completion of the investigational medicinal product infusion.

**Rationale**: The addition of immunogenicity as an AE of special interest was done to align with updates made to the Investigator's Brochure, Section 6.3.2.5 Adverse Events of Special Interest.

This changes also affects Section 4.5.2, Potential Risks and Section 5, Schedule of Activities.

# Section 17.3, Participant Information and Consent

**Change:** Updated language to state that participants can withdraw at any time from the study and how withdrawal from substudies impacts their participation in the overall study.

Now reads:

. . . .

Participants or their legally authorized representatives, in countries where applicable laws allows, who chose to participate in the LTE period must provide informed consent before any LTE period screening tests are performed.

- - -

The participant's study partner/informant must also provide written informed consent to participate in the study and be reconsented to participate in the LTE period. The original


forms will be managed and archived in the same manner as the participants' ICFs, as described above.

| Participants or the | <u>eir informant/study</u> | y partner ca | n withdraw | consent to | participate in | the |
|---|---|---|---|---|---|---|
| study at any time. | | | | | | |

**Rationale:** Language was added to clarify that participants can withdraw at any time from the study and clarify how withdrawal from substudies during the placebo-controlled period and LTE period impacts their participation in the overall study.

### SUMMARY OF MINOR CHANGES TO THE PROTOCOL

The following minor changes were made to the protocol, as appropriate:

- The version number and date were updated throughout the protocol.
- Sponsor Signature Page was updated.
- Typographical errors (i.e. Section 5, Schedule of Activities Table 1, CSSR-S assessment was moved from Week 56 to Week 52 Visit) and formatting were corrected.
- The term "subject" was replaced with "participant" throughout the document to reflect current standards when referring to participants in a study.
- Section 2, List of Abbreviations, was updated.
- Section 7.1, Study Overview, the number of study sites was increased from 90 to 100.



- Section 8.1, Inclusion Criteria, inclusion criterion 9 was updated to clarify that informant/study partner is required to give informed consent. Informant/study partner consent was previously required per in protocol version 2, Section 9.1, but it is now clarified in criterion 9.
- Section 10.1, Discontinuation of Study Treatment, was updated to clarify that
  participants who experiences an AE or an SAE that does not resolve or requires
  continued treatment that meets exclusionary criteria must be permanently
  discontinued from study treatment.
- Section 13.2, Pharmacokinetic Assessments, was corrected to include both trough and end-of-infusion BIIB092 concentrations.
- Section 16.8.1, Analysis Population, the term "immunogenicity" was replaced with "anti-BIIB092 antibody" as appropriate throughout the document when referring to anti-drug antibody assessment to avoid confusion with the AE of special interest similarly referred to as immunogenicity.



Biogen MA Inc. 225 Binney Street Cambridge, MA 02142 United States

Biogen Idec Research Limited Innovation House 70 Norden Road Maidenhead, Berkshire SL6 4AY United Kingdom

# AMENDMENT SUMMARY

Biogen Protocol 251AD201

Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects with Mild Cognitive Impairment due to Alzheimer's Disease or with Mild Alzheimer's Disease

Version 4

Date: 13 January 2020

EUDRA CT Number: 2017-002901-37

Version 4 of the protocol has been prepared for this amendment, which supersedes Version 3.

## PRIMARY REASON FOR AMENDMENT

The primary reason for this amendment to Protocol 251AD201 is to update the number of randomized participants from 528 to 654.

New text is shown in **bold** type; deleted text is shown with a strikethrough.

### Section 7.1, Study Overview

#### Now reads:

The study will be conducted in a parallel-group design, with 3 BIIB092 dose groups (including 4 BIIB092 doses) and a placebo group. Approximately 528 participants willwere planned to be randomized across approximately 100 study sites globally. As a result of fast recruitment leading to over-enrollment, the final number of randomized subjects is 654.

. . .

Randomized participants will receive 1 of the following study treatments by IV infusion every 4 weeks, starting on Study Day 1 during the placebo-controlled period:

- low-dose BIIB092 125 mg once every 4 weeks or 375 mg once every 12 weeks and placebo at the other 4-week dosing visits to maintain the treatment blind (88 participants planned in total, 44 per regimen)
- medium-dose BIIB092 600 mg once every 4 weeks (88 participants planned)
- high-dose BIIB092 2000 mg once every 4 weeks (176 participants planned)
- placebo (176 participants **planned**)

**Rationale:** The number of study participants was updated to reflect the final number of participants randomized after over-enrollment. The increase from 528 to 654 participants represents a significant change to the study plan. Because the statistical analysis is based on a sample size of 528, language emphasizing the planned sample size was added for clarification.

This change also affects Section 13.3, Pharmacodynamic Assessments.

## SUMMARY OF MAJOR CHANGES TO THE PROTOCOL

Changes to the protocol are presented chronologically. New text is shown in **bold** type; deleted text is shown with a strikethrough.

# Section 1, Synopsis

The synopsis was revised to reflect changes made throughout the protocol.

### Section 5, Schedule of Activities

**Change:** The following changes were made to the timing of scheduled assessments:

Safety Procedures

The frequency of MRIs was adjusted by removing MRI from Week 176 and Week 128 and adding it to Week 156. MRI will now be performed at Week 104 (6 months after start of LTE), Week 156 (18 months after start of LTE), and Week 226 (36 months after start of LTE). A row for body weight was added to Tables 2 through 4. Body weight measurements were added to all clinical visits that include a physical examination. A row for tobacco use status was added to Tables 1 through 4 below concomitant therapy and procedures reporting.

#### Biomarker

The frequency of PK/biomarkers/anti-BIIB092 antibodies collection during the LTE was adjusted for multiple study visits. PK/biomarkers/anti-BIIB092 antibodies will now be assessed at Week 116, Week 156, Week 196, and Week 224.

#### Clinical Assessments

Removal of NPI-10 and FAQ at Week 176 and ISLT, DKEFS, DSST, Trails A, and eCog at Week 180.

**Rationale:** To reduce the burden to participants, the original 4 MRIs planned during the LTE at Weeks 104, 128, 176, and 226 (at 6, 12, 24, and 36 months after starting the LTE, respectively) were reduced to 3 MRIs at Weeks 104, 156, and 226 (at 6, 18, and 36 months after starting the LTE, respectively). The Week 104 MRI represents a critical safety assessment for participants switching from placebo to treatment during the LTE. The Week 226 MRI is key for PD evaluation and for safety assessment at the end of the study. The Week 128 and Week 176 MRIs were condensed into a single Week 156 MRI in order to minimize participant burden. Based on


Amendment Summary for Protocol 251AD201, Version 4

current evaluations, this frequency of MRI monitoring is not expected to significantly affect the participants' benefit-risk. In addition, ad hoc MRI visits are possible as needed.

The frequency of biomarker and clinical assessments was reduced to decrease the burden to participants, particularly towards the end of the study.

A row for body weight was added to Tables 2 through 4 to provide further clarification on the frequency of body weight measurements.

A row for tobacco use status was added to Tables 1 through 4 to provide clarification on frequency and timing of the assessment.

This change also affects Section 11.4.3, Tobacco Use.

# Section 5, Schedule of Activities

**Change:** A footnote was added to Table 1 for the Week 78 MRI.

#### Now reads:

<sup>23</sup>Sites should schedule the Week 78 MRI within 10 days prior to the Week 78 visit where possible to allow for MRI results to be available before participants enter the LTE at Week 80.

**Rationale:** This change was made to improve the efficiency of eligibility assessments by allowing MRI results to be available before entering the LTE at Week 80.

## Section 5, Schedule of Activities

**Change:** The footnote in Table 1 regarding blood samples for assessment of BIIB092 concentration on days of infusion was revised.

### Now reads:

<sup>20</sup>Two samples must be obtained: 1 sample taken before infusion and 1 sample taken at  $\leq$ 1015 minutes after the end of infusion.

**Rationale:** This change was made to increase flexibility by providing a larger time window for sample collection with minimal impact on PK.



# Section 7.1, Study Overview

**Change:** All references to optional home visits were removed.

the home unless previously approved by the Investigator.

#### Now reads:

The visits at Weeks 32, 36, and 64 of the placebo controlled period may be conducted as home visits, if the Investigator is in agreement and appropriate services are available to perform the required study procedures and adequately monitor for potential safety events. These are study visits that do not require extensive assessments, e.g., administration of clinical scales

However, if the participant experienced a elinically significant infusion reaction during the first 24 weeks of the study, then the BIB092 infusion should not be administered in the home unless previously approved by the Investigator.

. . .

The visits at Weeks 84, 88, 96, 112, 116, 120, 136, 140, 144, 160, 164, 168, 184, 188, 192, 208, 212, and 216 of the LTE period may be conducted as home visits, if the Investigator is in agreement and appropriate services are available to perform the required study procedures and adequately monitor for potential safety events. These are study visits that do not require extensive assessments, e.g., administration of clinical scales. However, if the participant experienced a clinically significant infusion reaction during the first 24 weeks of the study or LTE period, then the BIB092 infusion should not be administered in


**Rationale:** These changes were made for logistical reasons and are not expected to affect patient safety.

This change also affects Section 5, Schedule of Activities and Section 7.2, Study Duration for Participants.

### Section 10.1, Discontinuation of Study Treatment

**Change:** Changes were made to recommended visits for participants who discontinue study treatment to reflect changes in the Schedule of Activities.

#### Now reads:

All participants who discontinue study treatment prematurely will be asked to remain in the study and continue all protocol-specified visits and procedures for the period in which they discontinued treatment (i.e., placebo-controlled or LTE). Participants who discontinue treatment during the placebo-controlled period should be encouraged to attend at least the Week 24, Week 52, and Week 78/EOS Visits and who discontinue treatment during the LTE should be encouraged to attend at least the Week 80, 104, 116, 128, 152, 156, 176, 196, 200, 224, and 226/EOS Visits, depending on when treatment was discontinued, and undergo all the scheduled procedures. At a minimum, these visits should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including at least the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. Participants who discontinue study treatment prematurely, regardless of the treatment period, will be asked to return to the study site for a Follow-up Safety Visit 14 weeks after receiving the last dose of study treatment. See Table 1, Table 2, Table 3, and Table 4 for the Schedule of Activities.

**Rationale:** Revision made to account for updates to timing of significant assessments in Table 2, Table 3, and Table 4.

### Section 11.4.1.2, Disallowed Concomitant Therapy

**Change:** Details were added regarding UVs for a change in AD medication.

### Now reads:

Participants should have an unscheduled visit (UV) prior to the initiation of, and/or a change in, dose, or discontinuation of AD medication. That visit should include assessment of AEs/SAEs and concomitant medications and key clinical assessments, including, at a minimum, the CDR, MMSE, ISLT, ADAS-Cog 13, ADCS-ADL, and FAQ. During the UV, these clinical assessments need not be repeated if performed within the previous 30 days. If the visit for a change in AD medication occurs at the same time as another planned visit, all originally scheduled assessments must also take place as required and without repetition (see Table 1, Table 2, Table 3, and Table 4).

**Rationale:** Details were added to minimize participant burden and to optimize the assessments performed during a change in AD medication as well as provide clarification for study sites.

This change also affects Section 5, Schedule of Activities.

# SUMMARY OF MINOR CHANGES TO THE PROTOCOL

The following minor changes were made to the protocol, as appropriate:

- The version number and date were updated throughout the protocol.
- Section 2, List of Abbreviations, was updated.
- Abbreviations were updated throughout the protocol where appropriate.
- The abbreviation list in the Figure 1 footnotes was updated to clarify that N represents the **planned** number of participants.
- All references to free eTau were changed to N-terminal tau or removed.
- Section 16.5.2, Methods of Analysis, was revised to clarify that concentration values below the limit of quantification will be appropriately handled per the Statistical Analysis Plan.
- Internal references were added as hyperlinks where appropriate.
- Typographical errors and formatting were corrected.

# LIST OF ABBREVIATIONS

| AD | Alzheimer's disease |
|---|---|
| ADAS-Cog 13 | Alzheimer's Disease Assessment Scale – Cognitive (13 item) |
| ADCS-ADL | Alzheimer's Disease Cooperative Study – Activities of Daily Living |
| AE | adverse event |
| CDR | Clinical Dementia Rating Scale |
| DKEFS | Delis-Kaplan Executive Function System |
| DSST | Digit Symbol Substitution Test |
| eCog | Everyday Cognition |
| EOS | end of study |
| FAQ | Functional Activities Questionnaire |
| ISLT | International Shopping List Test Immediate Recall |
| _IV | intravenous |
| LTE | long-term extension |
| MCI | mild cognitive impairment |
| MMSE | Mini-Mental State Examination |
| MRI | magnetic resonance imaging |
| NPI-10 | Neuropsychiatric Inventory – 10 |
| PD | pharmacodynamic(s) |
| PK | pharmacokinetic(s) |
| SAE | serious adverse event |
| Trails A | Trail Making Test, Part A |
| UV | unscheduled visit |